#### The GlaxoSmithKline group of companies

Division: Worldwide DevelopmentInformation Type: Reporting and Analysis Plan (RAP)

Title : Reporting and Analysis Plan for the effects of GSK2586881 on the responses to acute hypoxia and exercise

Compound Number : GSK2586881

Effective Date : 25-JUN-2018

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 204987.
- This RAP is intended to describe the safety, pharmacodynamic and pharmacokinetic analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Interim Analysis and Statistical Analysis Complete (SAC) deliverables.

#### **RAP Author(s):**

| Approver | Date | Approval Method |
|---|---|---|
| Principal Statistician (Respiratory, Clinical Statistics) | Not Applicable | Not Applicable |
| Manager (Respiratory, Clinical Pharmacology Modelling and Simulation) | 20-JUN-2018 | Pharma TMF |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

# **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Clinical Development Manager (CPSSO) | 15-JUN-2018 | Pharma TMF |
| Clinical Research Scientist (CPSSO) | 14-JUN-2018 | Pharma TMF |
| Project Physician Leader<br>(Respiratory TAU) | 25-JUN-2018 | Email |
| Principal Data Manager (CPSSO) | 25-JUN-2018 | Pharma TMF |
| SERM Director (GCSP) | 14-JUN-2018 | Pharma TMF |
| Manager (Respiratory, Clinical Programming) | 25-JUN-2018 | Pharma TMF |
| Translational Pharmacology Manager (Respiratory Fibrosis DPU) | 19-JUN-2018 | Pharma TMF |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|---------------------------------------------|-------------|-----------------|
| Director (Respiratory, Clinical Statistics) | 20-JUN-2018 | Pharma TMF |
| Manager (Respiratory, Clinical Programming) | 14-JUN-2018 | Pharma TMF |

# **TABLE OF CONTENTS**

| | | F | PAGE |
|---|---|---|---|
| 1. | REPO | RTING & ANALYSIS PLAN SYNOPSIS | 6 |
| 2. | SLIMIN | MARY OF KEY PROTOCOL INFORMATION | a |
| ۷. | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | Study Objective(s) and Endpoint(s) | |
| | 2.3. | Study Design | |
| | 2.4. | Statistical Hypotheses | |
| 3. | | NED ANALYSES | |
| | 3.1. | Interim Analyses | |
| | | 3.1.1. Part 1 | |
| | 2.0 | 3.1.2. Part 2 | |
| | 3.2. | Final Analyses | 14 |
| 4. | ANAL' | YSIS POPULATIONS | 14 |
| | 4.1. | Protocol Deviations | 15 |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | CONV | 'ENTIONS | 16 |
| 6. | STUD | Y POPULATION ANALYSES | 17 |
| | 6.1. | Overview of Planned Analyses | |
| 7. | DDIM | ARY STATISTICAL ANALYSES | 10 |
| ١. | 7.1. | Overview of Planned Analyses | |
| | 7.2. | Planned Statistical Analyses | |
| | | , | |
| 8. | | NDARY ANALYSES | |
| | 8.1. | Safety Analyses | |
| | | 8.1.1. Overview of Planned Analyses | |
| | 0.0 | 8.1.2. Planned Safety Statistical Analyses | |
| | 8.2. | Pharmacokinetic Analyses | |
| | | 8.2.1. Overview of Planned Pharmacokinetic Analyses | |
| | | 8.2.2. Drug Concentration Measures | |
| | | 8.2.3.1. Deriving Pharmacokinetic Parameters | |
| | | 8.2.4. Population Pharmacokinetic (PopPK) Analyses | |
| | 8.3. | Pharmacodynamic and Biomarker Analyses | |
| | 0.5. | 8.3.1. Overview of Planned Pharmacodynamic and Biomarker | 25 |
| | | Analyses | 25 |
| | | 8.3.2. Planned Pharmacodynamic and Biomarker Statistical | |
| | 8.4. | AnalysesPharmacokinetic / Pharmacodynamic Analyses | |
| | ∪. <del>1</del> . | Thatmacodinetic / Thatmacodynamic Analyses | 21 |
| 9. | REFE | RENCES | 28 |
| 10. | APPEI | NDICES | 29 |
| | 10.1. | Appendix 1: Time & Events | 30 |
| | | 10.1.1. Protocol Defined Time & Events | |

| | | | Screening and Follow up | |
|---|---|---|---|---|
| | | | Treatment Period 1 and 2 | |
| 10.2. | | | ent States | |
| | 10.2.1. | | States for AE Data | |
| | | | Treatment States for AE Dates | |
| | 10.2.2. | | States for Concomitant Medication Data | 35 |
| | | 10.2.2.1. | Treatment States for Concomitant Medication | |
| | | | Dates | |
| 10.3. | Appendix | | splay Standards & Handling Conventions | |
| | 10.3.1. | | atment & Sub-group Display Descriptors | |
| | 10.3.2. | | efinition & Derivations | |
| | | 10.3.2.1. | Baseline Definitions | 37 |
| | | 10.3.2.2. | Derivations and Handling of Missing Baseline | |
| | | | Data | 38 |
| | 10.3.3. | | Process & Standards | |
| 10.4. | Appendix | k 4: Derived | and Transformed Data | 41 |
| | 10.4.1. | General | | 41 |
| | 10.4.2. | Study Pop | ulation | 41 |
| | 10.4.3. | Safety | | 42 |
| | 10.4.4. | | dynamic and Biomarker | |
| 10.5. | Appendix | k 5: Premati | ure Withdrawals & Handling of Missing Data | 43 |
| | 10.5.1. | | Withdrawals | |
| | 10.5.2. | Handling o | f Missing Data | 43 |
| | | | Handling of Missing Dates | |
| | | | Handling of Partial Dates | |
| | | | Handling of Missing Data for Statistical | |
| | | | Analysis | 45 |
| 10.6. | Appendix | k 6: Values | of Potential Clinical Importance | |
| | | | Values' | |
| | 10.6.2. | | | |
| | 10.6.3. | | | |
| 10.7. | | | ker Details | |
| 10.8. | | | Checking and Diagnostics for Statistical | |
| | Analyses | S | | 49 |
| 10.9. | Appendix | k 9: Populat | ion PK and Pharmacokinetic / | |
| | | | Or Biomarker) Analyses | 50 |
| | 10.9.1. | | PK Dataset File Structure | |
| | 10.9.2. | Population | PK/PD Dataset File Structure : ANGII | 52 |
| | 10.9.3. | Population | PK/PD Dataset File Structure : ANG1-5 | 54 |
| | 10.9.4. | Population | PK/PD Dataset File Structure : ANG1-7 | 57 |
| | 10.9.5. | | PK/PD Dataset File Structure : Oxygen | |
| | | | /PASP | 59 |
| 10.10. | Appendix | | viations & Trade Marks | |
| | | | ons | |
| | | | (S | |
| 10 11 | | | Data Displays | |
| | | | ay Numbering | |
| | 10.11.2 | Mock Exar | nple Shell Referencing | 63 |
| | | | e [Priority] | |
| | 10 11 4 | Study Pon | ulation Tables | 64 |
| | | | les | |
| | | | ures | |

# 2017N335133\_00 204987

#### CONFIDENTIAL

| 10.11.7. Pharmacokinetic Tables | 73 |
|-----------------------------------------------------|----|
| 10.11.8. Pharmacokinetic Figures | 74 |
| 10.11.9. Pharmacodynamic and Biomarker Tables | |
| 10.11.10. Pharmacodynamic and Biomarker Figures | |
| 10.11.11. Pharmacokinetic / Pharmacodynamic Figures | 34 |
| 10.11.12.ICH Listings | 35 |
| 10.11.13. Non-ICH Listings | |
| Appendix 12: Example Mock Shells for Data Displays | |

# 1. REPORTING & ANALYSIS PLAN SYNOPSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | <ul> <li>The purpose of this Reporting and Analysis Plan is to describe all planned<br/>analyses and outputs required for the Clinical Study Report (CSR) of study<br/>204987. This amendment covers changes to the study following the interim<br/>analysis review of 11 participants.</li> </ul> |
| Protocol | <ul> <li>This RAP amendment is based on the protocol (Dated 23/SEP/2016, GSK Document No.: 2016N283626_00) and protocol amendments 1 &amp; 2 &amp; 3 (Dated:24/FEB/2017, GSK Document No.: 2016N283626_01 &amp; 07/MAR/2017, GSK Document No.: 2016N283626_02 &amp; 06/MAR/2018 GSK Document No.: 2016N283626_03) of study GSK2586881/204987</li> </ul> |
| Study<br>Design | The study will be a single centre, randomised, placebo-controlled and double blind (sponsor open). Subjects will be randomised to receive a single IV dose of GSK2586881 or saline in a crossover design. Approximately 25 subjects will be enrolled to ensure that a minimum of 20 subjects complete all dosing and critical assessments (the target of 20 may be revised by the sample size reestimation) |
| Primary<br>Objective | To evaluate the effect of a single IV dose of GSK2586881 on the HPV response in healthy volunteers during exercise under hypoxic conditions |
| Primary<br>Endpoint | Change from baseline of Pulmonary Artery Systolic Pressure (PASP) measured via Echocardiography |
| Planned<br>Analyses | • An Interim Analysis was planned after approximately 10 patients had completed periods 1 and 2 of the study, to aid the team in decision making with regards to stopping the study for futility or a re-assessment of sample size. Following the interim (referred to as study Part 1), amendments were made to the study before re-starting Part 2. Further interim reviews are planned when approximately 3 and 6 participants have completed periods 1 and 2 in Part 2 of the study. |
| | <ul> <li>All decisions regarding final analysis, as defined in this RAP document, will be<br/>made prior to Database Freeze.</li> </ul> |
| Analysis<br>Populations | <ul> <li>All Subjects Screened Population will contain all subjects that complete at least<br/>one Visit 1 (Screening) procedure.</li> </ul> |
| | <ul> <li>The Modified Intent-to-Treat (mITT) Population will comprise all randomised<br/>subjects, excluding those who were randomised in error.</li> </ul> |
| | The Modified Intent-to-Treat (mITT1) Part 1 Population will comprise all subjects in the mITT Population, who were randomised into Part 1 of the study. |
| | The Modified Intent-to-Treat (mITT2) Part 2 Population will comprise all subjects in the mITT Population, who were randomised into Part 2 of the study |
| | The Pharmacokinetic (PK) Population will comprise all subjects in the mITT Population, for whom a PK sample was obtained and analysed and on active treatment. |

| Overview | Key Elements of the RAP |
|---|---|
| | The Pharmacokinetic (PK1) Population Part 1 will comprise all subjects in the mITT Population, randomised in Part 1 of the study, for whom a PK sample was obtained and analysed and on active treatment. |
| | The Pharmacokinetic (PK2) Population Part 2 will comprise all subjects in the mITT Population, randomised in Part 2 of the study, for whom a PK sample was obtained and analysed and on active treatment. |
| Hypothesis | No formal statistical hypotheses are being tested. A Bayesian statistical analysis framework with non-informative priors for model parameters (unless otherwise specified) will be used to obtain posterior distributions for effects of interest. These posterior distributions will be used to obtain a number of probability statements about the magnitude of treatment effects (e.g. probability of any treatment related reduction in PASP, or probability that the treatment related reduction in PASP ≥ 5 mmHg). A rule of thumb for "end of study success" is if the probability of any treatment related reduction in PASP (T3-T0) exceeds 0.95 (success is also conditional on the probability of (absolute) treatment related reductions in oxygen saturation exceeding 5% being small). |
| Primary<br>Analyses | The primary endpoint, change from baseline in PASP following exercise under hypoxic conditions (Ti-T0) will be analysed using a Bayesian repeated measures mixed effects regression model, to compare the effects of Placebo vs GSK2586881. Analyses will be performed for Part 1 and Part 2 separately. |
| Secondary | Pharmacodynamic/Biomarker: |
| Analyses | RAS peptide responses: Ang II, Ang(1-7), Ang(1-5) will be analysed in a manner similar to the primary endpoint using Bayesian repeated measures mixed modelling to compare the effects of Placebo vs GSK2586881, for Part 2, if data permit. Part 1 data may also be analysed. Data from Part 1 and Part 2 will also be presented descriptively. |
| | Safety: |
| | Oxygen saturation will be analysed in a manner similar to the primary efficacy endpoint using Bayesian repeated measures mixed modelling to compare the effects of Placebo vs GSK2586881. Analyses will be performed for Part 1 and Part 2 separately. Vital signs, 12-Lead ECG, AEs and Labs will be tabulated and/or listed by treatment group, study part (Part 1 and 2) and timepoint as appropriate. |
| | Immunogenicity: |
| | Data will be tabulated and/or listed. |
| | Pharmacokinetic: |
| | Plasma concentrations of GSK2586881 and derived PK parameters will be summarised descriptively/graphically and listed for Part 1 and Part 2 of the study. |
| Exploratory | Pharmacodynamic/Biomarker: |
| Analyses | The disease biomarker Surfactant Protein D will be analysed in a manner similar to the primary efficacy endpoint using Bayesian repeated measures mixed modelling to |

| Overview | Key Elements of the RAP |
|---|---|
| | compare the effects of Placebo vs GSK2586881, for Part 2, if data permit. Part 1 data may also be analysed. Data from Part 1 and Part 2 will also be presented descriptively. |
| | Ventilatory parameters (Oxygen consumption (VO2), Carbon dioxide production (CO2), Total Tidal Volume, Inspiratory Tidal Volume, Expiratory Tidal Volume, Total Respiratory Time, Inspiratory Time, Expiratory Time, Duty Cycle, Mean Respiratory Flow and Respiratory rate) will be summarised descriptively and listed, by treatment group, timepoint and study part (Part 1 and 2). |
| | Pulmonary vascular resistance (PVR) will be summarised descriptively and listed, by treatment and timepoint, for Part 2. A statistical analysis similar to that described for PASP will also be performed. |
| | Pharmacogenetics |
| | Analysis of pharmacogenetic data will be carried out separately by the GSK Genetics team and a separate RAP will be produced. As this is an exploratory endpoint, the results will be available separately to the CSR (or to be included as an appendix). |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no major changes or deviations to the originally planned statistical analysis specified in the protocol (Dated: 23/SEP/2016) and protocol amendments 1, 2 and 3 (dated 24/FEB/2017, 07/MAR/2017 and 06MAR2018).

This amendment details changes to the display of outputs in relation to separate summaries of Part 1 and 2 data (as detailed in protocol amendment 3).

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objective | Primary Endpoint |
| To evaluate the effect of a single<br>IV dose of GSK2586881 on the<br>HPV response in healthy<br>volunteers during exercise under<br>hypoxic conditions | Change from baseline of Pulmonary Artery Systolic<br>Pressure (PASP) measured via Echocardiography |
| Secondary Objectives | Secondary Endpoints |
| To evaluate the effect of a single IV dose GSK2586881 on RAS peptide responses To evaluate the safety of a single IV dose of GSK2586881 in healthy volunteers | <ul> <li>Effect of GSK2586881 on baseline levels and changes in response to hypoxia and exercise of RAS peptides (e.g. Ang II, Ang(1-7), Ang(1-5))</li> <li>Vital signs (heart rate, systolic and diastolic blood pressure)</li> <li>Oxygen saturation</li> <li>12-lead ECGs</li> <li>Adverse Events (AEs)</li> <li>Immunogenicity</li> <li>Clinical laboratory assessments</li> <li>Continuous pulse oximetry (assessed by the site)</li> </ul> |
| To evaluate the pharmacokinetics | Plasma concentrations of GSK2586881 |
| of a single IV dose of GSK2586881 | Derived pharmacokinetic parameters |
| Exploratory Objectives | Exploratory Endpoints |
| To evaluate the effect of a single<br>IV dose of GSK2586881 on<br>ventilatory parameters in healthy<br>volunteers during exercise in<br>hypoxic conditions | <ul> <li>Change from baseline of:</li> <li>Oxygen consumption (VO2)</li> <li>Carbon dioxide production (CO2)</li> <li>And other parameters as data permit</li> </ul> |
| To evaluate the pharmacodynamic<br>activity of a single IV dose of<br>GSK2586881 in healthy volunteers<br>during exercise in hypoxic<br>conditions | Change from baseline in Surfactant Protein D and/or additional analytes to be determined |
| To evaluate the effect of a single<br>IV dose of GSK2586881 on the<br>HPV response in healthy<br>volunteers under hypoxic | Estimation of pulmonary vascular resistance (PVR) measured via Echocardiography |

| Objectives | Endpoints |
|---|---|
| conditions (and during exercise under hypoxic conditions). | |
| To evaluate Pharmacogenetics | Evaluate I/D polymorphisms in the Angiotensin<br>Converting Enzyme (ACE) gene and analyse the<br>impact on Ang II (and possibly other RAS peptides),<br>hypoxic pulmonary vasoconstriction and responses<br>to GSK2586881 administration |

# 2.3. Study Design



| Overview of S | Study Design and Key Features |
|---|---|
| Treatment | Treatment A: Placebo |
| Assignment | <ul> <li>Treatment B: GSK2586881 0.8 mg/kg</li> </ul> |
| | <ul> <li>Subjects will be randomised to one of two treatment sequences AB or BA</li> </ul> |
| Interim<br>Analysis | <ul> <li>Planned after approximately 10 subjects had completed treatment periods 1 and 2 (Part 1). The study may have been stopped if a reasonable change in PASP was not observed or if a review of safety data suggested a change in the benefit-risk profile. Following the interim, the decision was taken to continue the study with modifications to the protocol (Part 2).</li> <li>In Part 2 an interim review is planned when approximately 3 subjects have completed treatment periods 1 and 2. A further review may take place when approximately 6 subjects have completed treatment periods 1 and 2, dependent on data observed in the earlier review. Subsequent interim reviews may take place, if deemed appropriate.</li> </ul> |

# 2.4. Statistical Hypotheses

There are no formal statistical hypotheses. This is an exploratory study and will be analysed, utilising a Bayesian framework.

# 3. PLANNED ANALYSES

# 3.1. Interim Analyses

#### 3.1.1. Part 1

An interim analysis was planned after approximately 10 subjects had completed the following critical assessments:

| Interim Analysis | Definition / Criteria / Purpose |
|---|---|
| PASP at T0 and T3 for both study periods | <ul> <li>Assess treatment differences between GSK2586881 and Placebo in change from pre-dose PASP to hypoxic/exercised PASP [T3-T0].</li> <li>To decide whether to continue the study or stop based on futility.</li> <li>To conduct an advisory sample-size re-estimation with the view to potentially reduce the number of subjects participating in the study below 20. Precision estimates will be updated based on the variability observed from the interim analyses to aid the team in decision making.</li> <li>PASP data will be summarised and listed. Statistical analysis will be completed as described in Section 7.2 including a graphic of treatment estimates over time.</li> </ul> |
| Oxygen saturation<br>at T0 and T3 for<br>both study periods | <ul> <li>To estimate treatment differences between GSK2586881 and Placebo in change from pre-dose oxygen saturation to hypoxic/exercised oxygen saturation [T3-T0], with a view to stopping the study if there is evidence that GSK2586881 causes a reduction in oxygen saturation in healthy volunteers. As a non-binding guide high posterior probability of observing ≥5% absolute differences in mean oxygenation saturation values between placebo and active arms would be of concern; but clinical judgement would override any statistical methods if, for example, the majority of subjects displayed consistent patterns of reductions e.g. between 2-3%.</li> <li>Oxygen saturation data will be summarised and listed. Statistical analysis</li> </ul> |

| Interim Analysis | Definition / Criteria / Purpose |
|---|---|
| _ | will be completed as described in Section 8.1.2 including a graphic of treatment estimates over time. |
| Adverse Events | <ul> <li>To compare adverse events within the two treatment groups and explore any potential safety signals that may emerge.</li> <li>AEs will be tabulated by treatment group (if there are a sufficient number of events) and listed.</li> </ul> |
| Angiotensin biomarker concentrations (Ang II, Ang(1-5), Ang(1-7)) | <ul> <li>For the first 5 subjects only to allow time for the samples to be analysed by the lab.</li> <li>Data will be listed only due to expected small sample size. Individual subject plots may be produced.</li> <li>If Angiotensin data (Ang II, Ang(1-5), Ang(1-7)) is not available at the time of the interim, analysis of the specified eCRF data will still go ahead as planned. A positive outcome in relation to PASP, Oxygen Saturation and AEs would lead to the study continuing without the need to review Angiotensin data.</li> <li>Should a negative outcome be observed with PASP or Oxygen Saturation, then confirmation of the decision to stop the study for futility would not occur until the Angiotension data from the initial transfer were available and reviewed.</li> <li>Any negative results with regards to AEs (as agreed by the study team), regardless of other endpoint results, would result in the study stopping.</li> </ul> |

The interim analysis was to use a data snapshot that had been cleaned to the best extent allowed by the timeframes (i.e. the interim data would not be fully cleaned or fully QC'd data and there would not be a locked database). The date of the source data cut was to be indicated on each interim related output (implemented in HARP via the *d\_datadate* macro input parameter in the *ts\_setup* macro call). Results were to be restricted to selected members of the study team. Results or discussions were not to be circulated to blinded staff involved in the conduct of the study at the sites.

The following table represents a guide to the outputs to be produced for the interim analysis. All outputs were to be produced in HARP.

| Endpoint / Parameter/<br>Display Type | | Absolute | | | | | | | | Change from Baseline | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | s Ana | lysis | Sum | Summary | | Individual | | Stats Analysis | | | Summary | | Individual |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| PASP | | | | Υ | Υ | Υ | Υ | <b>Y</b> 3 | Υ | | Υ | | | |
| Oxygen Saturation | | | | Υ | Υ | Υ | Υ | <b>Y</b> 3 | Υ | | Υ | | | |
| All AEs | | | | Y1 | | | Y <sup>2</sup> | | | | | | | |
| RAS Peptides (AngII,<br>Ang(1-5), Ang(1-7)) | | | | | | Y | Y | | | | | | | |

#### NOTES:

- Y = Yes display generated.
- 1. Produced if sufficient data
- 2. SAEs will be flagged within this listing

• 3. One table to include statistical analysis medians (95% Crl) and posterior probabilities. Also include within subject correlation as a footnote to support sample size re-estimation.

The sample size re-estimation was to be performed once the primary analysis for the interim had been completed and assuming that no overwhelming data supporting the need to stop for futility was observed. Estimates of standard deviations and within subject correlation were to be obtained from the PASP outputs produced during the interim and/or from SAS outputs from the statistical modelling. The sample size re-estimation was to be performed by re-running programs (using R) used to obtain pre-study precision estimates. The sample size re-estimation program and associated excel outputs of precision estimates were to be archived.

The interim analysis was performed when 11 subjects had been randomised. One subject did not complete both periods 1 and 2 due to withdrawal due to AE, therefore 10 subjects were analysed for the primary endpoint. Following a review of the data, the decision was made to make modifications to the protocol and continue the study (Part 2). Major modifications are a change in the hypoxia chamber altitude from 4000m to 5000m and echo recordings at the T3 timepoint being taken 2 minutes into exercise (due to use of semi-recumbent cycle), rather than at the end of a 10 minute exercise period. Part 1 and 2 of the study will be analysed separately.

#### 3.1.2. Part 2

For Part 2 of the study, up to 14 subjects are planned to be randomised. Two interim analysis reviews are planned as follows:

- Review of PASP, oxygen saturation and AE data when approximately 3 subjects have completed Treatment Periods 1 and 2.
- Review of PASP, oxygen saturation and AE data when approximately 6 subjects have completed Treatment Periods 1 and 2. This second review may not be required and will be dependent on data observed during the first interim review. The timing of this review may be altered, as necessary, dependent on subject recruitment. Further interim reviews may take place, if appropriate.

At each review, the study may be stopped for futility if PASP results are highly variable, or if the PASP profile for the placebo group is not as expected (indicative of the model not working given the alterations to the study) or if review of the safety data suggests a change in the benefit-risk profile. If clear criteria for stopping the study are not met, the study will continue to the next interim analysis review, or on to the planned maximum number of evaluable subjects. Further interim reviews may be performed if deemed appropriate by the study team.

The following table represents a guide to the outputs to be produced for the interim analysis reviews. All outputs were to be produced in HARP. Adverse events (AEs) will be assessed via Inform or a listing produce via HARP.

| Endpoint / Parameter/ Display Type | | | Þ | Absolu | te | | | Change from Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | s Ana | lysis | Summary | | Individual | | Stat | Stats Analysis | | Summary | | Individua | |
| | Т | F | L | Т | F | F | L | Τ | F | L | Τ | F | F | L |
| PASP | | | | | | Υ | Υ | | | | | | | |
| Oxygen Saturation | | | | | | Υ | Υ | | | | | | | |
| All AEs | | | | | | | <b>Y</b> 1 | | | | | | | |

**NOTES**: Y = Yes display generated, 1. Produced if sufficient data available

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol (and subject to decisions made from the interim analyses).
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.
- 3. All criteria for unblinding the randomisation codes have been met (note that the study is being run as sponsor-unblinded, however, only a partial randomisation schedule will be made available to the GSK programming team for the interim analysis).
- 4. Randomisation codes have been distributed according to RandAll NG procedures.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Subjects<br>Screened | Comprising of all subjects who complete at least one Visit 1 (Screening) procedure. | <ul> <li>Subject disposition<br/>(including reasons for<br/>screening failures)</li> <li>Listing of any<br/>AEs/SAEs for non-<br/>randomised subjects</li> </ul> |
| Modified Intent-<br>To-Treat (mITT) | Comprising of all randomised subjects, excluding those who were randomised in error. A subject who is recorded as a screen failure, but is randomised and does not receive a dose of study treatment is considered to have been randomised in error. Any other subject who receives a randomisation number will be considered to have been randomised. | Study Population,<br>Safety & PD/Biomarker<br>listings and selected<br>tables/figures |
| Modified Intent-<br>To-Treat Part 1<br>(mITT1) | This will comprise all subjects in the mITT population, who were randomised into Part 1 of the study (planned 4000m altitude) | Safety & PD/Biomarkers tables and figures (Part 1) |
| Modified Intent-<br>To-Treat Part 2<br>(mITT2) | This will comprise all subjects in the mITT population, who were randomised into Part 2 of the study (planned 5000m altitude) | Safety & PD/Biomarkers tables and figures (Part 2) |
| Pharmacokinetic (PK) | Subjects in the 'mITT' population, for whom a pharmacokinetic sample was obtained and analysed and on active treatment. | PK Listings |
| Pharmacokinetic<br>Part 1 (PK1) | Subjects in the 'mITT' population, randomised in Part 1 of the study, for whom a pharmacokinetic sample was obtained and analysed and on active treatment. | PK Part 1 tables and figures |
| Pharmacokinetic | Subjects in the 'mITT' population, randomised | PK Part 2 tables and |

| Population | Definition / Criteria | Analyses Evaluated |
|--------------|-----------------------------------------|--------------------|
| Part 2 (PK2) | in Part 2 of the study, for whom a | figures |
| | pharmacokinetic sample was obtained and | |
| | analysed and on active treatment. | |

#### NOTES:

 Please refer to Appendix 11: List of Data Displays which details the population to be used for each display being generated.

#### 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, subject management or subject assessment) will be summarised and listed.
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.
- A listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 10.1 | Appendix 1: Time & Events |
| 10.2 | Appendix 2: Treatment States |
| 10.3 | Appendix 3: Data Display Standards & Handling Conventions |
| 10.4 | Appendix 4: Derived and Transformed Data |
| 10.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| 10.6 | Appendix 6: Values of Potential Clinical Importance |
| 10.7 | Appendix 7: Biomarker Details |
| 10.8 | Appendix 8: Model Checking and Diagnostics for Statistical Analyses |
| 10.9 | Appendix 9: Population PK and Pharmacokinetic / Pharmacodynamic (or Biomarker) Analyses |
| 10.10 | Appendix 10: Abbreviations & Trade Marks |
| 10.11 | Appendix 11: List of Data Displays |
| 10.12 | Appendix 12: Example Mock Shells for Data Displays |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Analyses

The study population analyses will be based on the Modified Intent-To-Treat populations (mITT, mITT1 and mITT2, as appropriate), unless otherwise specified.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 11: List of Data Displays.

 Table 2
 Overview of Planned Study Population Analyses

| Endpoint / Parameter / Display Type | Data D | isplays G | enerated | |
|---|---|---|---|---|
| | Table | Figure | Listing | Population for displays |
| Subject Disposition | | | | |
| Subject Disposition | Υ | | | mITT |
| Screening Status and Reasons for Screen Failure | Y | | Υ | All Subjects Screened |
| Reasons for Subject Withdrawal | | | Υ | mITT |
| Important Protocol Deviations | Υ | | Υ | mITT |
| Subjects with Inclusion/Exclusion Criteria Deviations | | | Υ | mITT |
| Randomised and Actual Treatments | | | Υ | mlTT |
| Subjects for Whom the Treatment Blind was Broken | | | Υ | mITT |
| Populations Analysed | | | | |
| Study Populations | Υ | | | All Subjects Screened |
| Subjects Excluded from Any Population | | | Υ | All Subjects Screened |
| <b>Demographic and Baseline Characteristics</b> | | | | |
| Demographic Characteristics | Υ | | Υ | mITT1 and mITT2 |
| Race and Racial Combinations | Υ | | Υ | mITT1 and mITT2 |
| Prior and Concomitant Medications | | | | |
| Medical Conditions <sup>1</sup> | Υ | | | mITT |
| Concomitant Medications | | | Υ | mITT |
| <b>Exposure and Treatment Compliance</b> | | | | |
| Exposure to Study Treatment | | | Υ | mITT |

#### NOTES:

- Y = Yes display generated.
- 1. Separate summaries for past and current conditions

#### 7. PRIMARY STATISTICAL ANALYSES

### 7.1. Overview of Planned Analyses

The primary analyses will be based on the Modified Intent-To-Treat populations (mITT, mITT1 and mITT2).

Table 3 provides an overview of the planned analyses, with full details of data displays being presented in Appendix 11: List of Data Displays.

Table 3 Overview of Planned Analyses

| Endpoint / | | | A | bsolu | te | | | Change from Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter/ Display | Stat | Stats Analysis S | | Summary | | Individual | | Stats Analysis | | | Summary | | Individual | |
| Туре | T | F | L | T | F | F | L | T | F | L | T | F | F | L |
| Primary | | | | | | | | | | | | | | |
| Pulmonary Artery | | | | Υ | Υ | Υ | Υ | Y1 | Υ | | Υ | | | |
| Systolic Pressure | | | | | | | | | | | | | | |
| (PASP) | | | | | | | | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. One table to include statistical analysis medians (95% CrI) and posterior probabilities.

# 7.2. Planned Statistical Analyses

# Primary Statistical Analyses

## **Endpoint**

Pulmonary Artery Systolic Pressure (PASP)

#### **Model Specification**

- The description below describes the current thinking of how to analyse this endpoint. The
  proposed model will be assessed, and if not appropriate alternative models could be used.
  Reasons for and a full description of alternative modeling methods used would be fully
  documented in the CPSR.
- The data will be inspected prior to analysis to determine whether a data transformation is required. Any data transformations (e.g. natural logarithm) will be applied to observed individual data prior to any modeling or derivations (e.g. prior to deriving subject baseline)
- Separate analyses will be performed for Part 1 and Part 2 of the study.
- A Bayesian repeated measures mixed effects model (fitted using SAS PROC MCMC), will be
  used to model the change from baseline (Ti-T0) in PASP. Based on the study design there are
  4 post-dose timepoints (T1, T2, T3 and T4). The timepoint of primary interest is T3; in Part 1
  this is immediately after exercise at an altitude of 4000m and in Part 2, this is 2 minutes into a
  reduced exercise challenge at an altitude of 5000m.
- Covariates for period, treatment and timepoint (i.e., T1 to T4) will be included as fixed effects.
   Adjusted period-specific baseline and subject-level baseline will be included as continuous parameters (see Section 10.3.2.1). Subject will be included as a random effect and timepoint will be included as a repeated effect. Treatment by timepoint and adjusted period-specific baseline by timepoint interactions will be included. An unstructured variance-covariance matrix

#### **Primary Statistical Analyses**

will be fitted. Non-informative priors will be used for the model parameters, (see Section 10.8).

- Examination of covariates (for example Age, Weight, Height) may take place, if data permit. In
  this case, the equivalent model may be fitted in PROC MIXED and the covariate assessed at a
  10% alpha level. The final Bayesian model would then be fit based upon the final model (after
  covariate examination) obtained using PROC MIXED. Alternatively, changes in deviance
  information criteria (DIC) may be assessed as part of the PROC MCMC modelling to examine
  covariates.
- Appropriate combinations of the model parameters would be used to obtain posterior distributions for the GSK2586881 vs placebo comparisons at each of the post dosing timepoints (T1 to T4).
- The change from baseline across the different post-dose timepoints will be represented via
  adjusted posterior medians for GSK2586881 and placebo, as well as associated 95% equitailed credible intervals. These results will be presented within tabular and graphical form after
  data has been back transformed (if applicable).
- The difference between GSK2586881 and placebo, for the change from baseline across postdose timepoints will be represented via adjusted medians, as well as their associated 95% equi-tailed credible intervals. These results will be presented within tabular form after data has been back transformed (if applicable).
- The posterior distributions will also be used to produce several posterior probability statements, presented in tabular format; the most important being the probability that the change from baseline in PASP is reduced by GSK2586881 at time T3.
- Posterior probabilities of interest include (looking for <u>high probabilities</u> to favour increases to a lesser extent in PASP on GSK2586881):
  - Probability that change from baseline in PASP is reduced by GSK2586881

     (i.e., probability that a treatment difference is negative, or if a log transformation is applied then the probability that the ratio is less than 1).
  - Probability that change from baseline in PASP is reduced by >=2.5mmHg and
     >=5mmHg by GSK2586881

(i.e., probability that a treatment difference is <=-2.5 mmHg and <=-5mmHg. In the case of a log-transformation, ratios of interest would be <0.95 and <0.90, representing 5% and 10%difference between groups)

Probability cut-offs may be re-assessed at the time of analysis

# **Model Checking & Diagnostics**

Refer to Appendix 8: Model Checking and Diagnostics for Statistical Analyses

#### **Model Results Presentation**

- Summary tables for absolute and change from baseline by treatment and timepoint (T0 to T4) (for Part 1 and Part 2)
- Listing of absolute data
- Individual subject profiles by treatment group and timepoint (for Part 1 and Part 2)
- Summary table of statistical analysis, adjusted change from baseline posterior medians and 95% credible intervals by treatment and timepoint, together with estimated posterior median treatment differences (GSK2586881 – Placebo) and 95% credible intervals for the change from baseline at times T1 to T4 along with posterior probabilities of interest (for Part 1 and Part 2)
- Figure of absolute PASP by timepoint (for Part 1 and Part 2)
- Figure of statistical analysis adjusted change from baseline medians and 95% credible intervals by treatment group and timepoint (for Part 1 and Part 2)

# 8. SECONDARY ANALYSES

# 8.1. Safety Analyses

# 8.1.1. Overview of Planned Analyses

The safety analyses will be based on the Modified Intent-To-Treat populations (mITT, mITT1 and mITT2), unless otherwise specified.

Table 4 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 11: List of Data Displays.

Table 4 Overview of Planned Safety Analyses

| Endpoint / Parameter/<br>Display Type | Absolute | | | | | | Change from Baseline | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | | | Sum | Summary Ind | | ridual | Stat | ts Ana | lysis | Summary | | Indiv | ridual |
| | Т | F | L | T | F | F | L | Т | F | L | Т | F | F | L |
| Oxygen Saturation | | | | | | | | | | | | | | |
| Oxygen Saturation,<br>measured by continuous<br>pulse oximetry | | | | Υ | Y | Υ | Y | <b>Y</b> 1 | Y | | Υ | | | |
| Oxygen Saturation vs PASP <sup>2</sup> | | | | | Y | | | | | | | | | |
| Pulmonary Vascular Res | istand | ce | | | | | | | | | | | | |
| PVR collected via ECHO | | | | Υ | Υ | Υ | Υ | <b>Y</b> 1 | Υ | | Υ | | | |
| Adverse Events | | | | | | | | | | | | | | |
| All AEs for Non- | | | | | | | Υ | | | | | | | |
| randomised Subjects | | | | | | | | | | | | | | |
| All AEs by SOC and PT <sup>3</sup> | | | | Υ | | | Υ | | | | | | | |
| AEs Leading to Study Discontinuation | | | | | | | Υ | | | | | | | |
| Drug-Related AEs by SOC and PT | | | | Υ | | | | | | | | | | |
| All Serious AEs | | | | Υ | | | Υ | | | | | | | |
| All Laboratory <sup>4</sup> | | | • | | • | • | | • | • | • | • | | | |
| Laboratory Values of PCI | | | | | | | Υ | | | | | | | |
| All Laboratory Data for Subjects with any Value of PCI | | | | | | | Y | | | | | | | |
| ECG | | | | | | | | | | | | | | |
| ECG Findings | | | | Υ | | | Υ | | | | | | | |
| ECG Values by Visit | | | | Υ | | | | | | | Υ | | | |
| ECG Values of PCI | | | | Υ | | | Υ | | | | Υ | | | |
| All ECG Values for Subjects with any Value | | | | | | | Y | | | | | | | |

| Endpoint / Parameter/<br>Display Type | | | Α | bsolu | te | | | Change from Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sta | Stats Analysis S | | Sum | Summary | | Individual | | Stats Analysis | | | mary | Individual | |
| | T | F | L | T | F | F | L | Т | F | L | Т | F | F | L |
| of PCI | | | | | | | | | | | | | | |
| Vital Signs | | | | | | | | | | | | | | |
| Vital Signs by Visit | | | | Υ | | | | | | | Υ | | | |
| Vital Signs of PCI | | | | | | | Υ | | | | | | | |
| All Vital Signs for<br>Subjects with any Value<br>of PCI | | | | | | | Y | | | | | | | |
| Immunogenicity | | | | | | | | | | | | | | |
| Immunogenicity | | | | Υ | | | Υ | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated, PCI = Potential Clinical Importance
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. One table to include statistical analysis medians (95% Crl) and posterior probabilities.
- 2. Scatter plot of x vs y (OS vs PASP) by treatment group, timepoint indicated by panel. To be produced for the mITT2 population only.
- 3. Listing will include subject's numbers for individual AE's and AE system organ classes, preferred terms and verbatim term.
- 4. Chemistry and haematology data will be assessed for PCI values.
- Chemistry collected: BUN, Creatinine, Glucose, Potassium, Sodium, Calcium, AST (SGOT), ALT (SGPT), Alkaline phosphatase, Total and direct bilirubin, Total protein, Albumin.
- Haematology collected: Platelet count, RBC count, haemoglobin, hematocrit, MCV, MCH, neutrophils, lymphocytes, monocytes, eosinophils, basophils.
- Urinalysis collected: Specific gravity, pH, glucose, protein, blood and ketones by dipstick, microscopic examination (if blood or protein is abnormal).
- With the exception of Immunogenicity table (mITT) and OS vs PASP scatter plot (mITT2), all tables and figures
  will be produced separately for the mITT1 and mITT2 populations. Listings will be produced based on the overall
  mITT population.

# 8.1.2. Planned Safety Statistical Analyses

# Planned Statistical Analyses

#### Endpoint(s)

Oxygen Saturation

#### **Model Specification**

- Refer to Section 7.2. Oxygen Saturation will be analysed in the same manner as for the primary endpoint PASP.
- Posterior probabilities of interest include (looking for <u>very low probabilities</u> to remove any concerns with regards to Oxygen Saturation reduction on GSK2586881):
  - Probability that the change from baseline on Oxygen Saturation is reduced by GSK
     (i.e., probability that a treatment difference is <0% or if a log transformation is
     applied then the probability that the ratio < 1).</li>

#### **Planned Statistical Analyses**

Probability that the change from baseline in Oxygen Saturation is reduced by GSK by
 3% and >=5% (absolute difference) compared to placebo.

(i.e., probability that a treatment difference (absolute) is <-3% and <=-5%. In the case of a log-transformation, ratios of interest would be <0.94 and <0.92 representing 6% and 8% difference between groups)

Probability cut-offs may be re-assessed at the time of analysis

#### **Model Checking**

Refer to Appendix 8: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- Summary tables for absolute and change from baseline by treatment and timepoint (T0 to T4) (for Part 1 and Part 2)
- Listing of absolute data
- Individual subject profiles by treatment group and timepoint (for Part 1 and Part 2)
- Summary table of statistical analysis, adjusted change from baseline posterior medians and 95% credible intervals by treatment and timepoint, together with estimated posterior median treatment differences (GSK2586881 – Placebo) and 95% credible intervals for the change from baseline at times T1 to T4 along with posterior probabilities of interest (for Part 1 and Part 2)
- Figure of absolute Oxygen Saturation by timepoint (for Part 1 and Part 2)
- Figure of statistical analysis adjusted change from baseline medians and 95% credible intervals by treatment group and timepoint (for Part 1 and Part 2)

### **Planned Statistical Analyses**

#### Endpoint(s)

Pulmonary Vascular Resistance (PVR)

#### **Model Specification**

- Refer to Section 7.2. PVR will be analysed in the same manner as for the primary endpoint PASP.
- Posterior probabilities of interest to include (looking for <u>high probabilities</u> to favour increases to a lesser extent in PVR on GSK2586881):
  - Probability that change from baseline in PVR is reduced by GSK2586881 (i.e., probability that a treatment difference is negative, or if a log transformation is applied then the probability that the ratio is less than 1).
  - Probability that change from baseline in PVR is reduced by >=0.1 wood units and >=0.3 wood units

(i.e., probability that a treatment difference is <=-0.1 wood units and <=-0.3 wood units. In the case of a log-transformation, ratios of interest would be <0.95 and 0.90, representing 5% and 10% difference between groups)

• Probability cut-offs may be re-assessed at the time of analysis

#### **Model Checking**

Refer to: Appendix 8: Model Checking and Diagnostics for Statistical Analyses

#### Model Results Presentation (Part 2 only)

- Summary tables for absolute and change from baseline by treatment and timepoint (T0 to T4)
- Listing of absolute data
- Individual subject profiles by treatment group and timepoint

#### **Planned Statistical Analyses**

- Summary table of statistical analysis, adjusted change from baseline posterior medians and 95% credible intervals by treatment and timepoint, together with estimated posterior median treatment differences (GSK2586881 – Placebo) and 95% credible intervals for the change from baseline at times T1 to T4 along with posterior probabilities of interest
- Figure of absolute PVR by timepoint
- Figure of statistical analysis adjusted change from baseline medians and 95% credible intervals by treatment group and timepoint

# 8.2. Pharmacokinetic Analyses

#### 8.2.1. Overview of Planned Pharmacokinetic Analyses

The pharmacokinetic (PK) analyses will be based on the Pharmacokinetic populations for Part 1 and Part 2, unless otherwise specified.

Table 5 provides an overview of the planned analyses, with full details being presented in Appendix 11: List of Data Displays.

Table 5 Overview of Planned Pharmacokinetic Analyses

| Endpoints | | Untrans | formed | | Log-Transformed | | | |
|---|---|---|---|---|---|---|---|---|
| | Sum | mary | Indiv | idual | Sum | mary | Individual | |
| | F | T | F | L | F | T | F | L |
| Plasma GSK2586881 concentrations | <b>Y</b> 1, 3 | Y | Y1,2 | Y | | | | |
| Pharmacokinetic Parameters | | Υ | | Υ | | Υ | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- Linear and Semi-Log plots will be created on the same display.
- 2. One output for one graph per subject and a further output with all subject profiles on the same graphic
- 3. Separate Mean (± SD) and Median plots will be generated.
- All tables and figures will be produced separately for the PK1 and PK2 populations. Listings will be produced for the overall PK population.

#### 8.2.2. Drug Concentration Measures

Refer to Appendix 3: Data Display Standards & Handling Conventions (Section 10.3.3 Reporting Process & Standards).

#### 8.2.3. Pharmacokinetic Parameters

#### 8.2.3.1. Deriving Pharmacokinetic Parameters

- Refer to Appendix 3: Data Display Standards & Handling Conventions (Section 10.3.3 Reporting Process & Standards).
- The pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using Win Nonlin Pro V6.3 or greater.
- All calculations of non-compartmental parameters will be based on actual sampling times.
- Pharmacokinetic parameters described in Table 6 will be determined from the plasma concentration-time data, as data permits.

Table 6 Derived Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| AUC(0-2.5h)<br>post-dose | Area under the concentration-time curve over the study period (pre-dose to 30 mins rest post chamber exit). |
| AUC(0.5-2.0h)<br>post-dose | Area under the concentration-time curve over the time period for the hypoxia challenge (immediately prior to chamber entry to chamber exit). |
| AUC(0-∞) | Area under the concentration-time curve extrapolated to infinity. |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| t½ | Apparent terminal half-life will be calculated as: |
| | t½ = ln2 / lambda_z |
| CL | Clearance |
| V | Volume of distribution |
| Lambda_z | The first order rate constant associated with the terminal (log-linear) portion of the concentration-time curve. |
| Lambda_z_lower | First time point used in computing Lambda_z. |
| Lambda_z_upper | Last time point used in computing Lambda_z. |
| #pts | Number of points used in computing Lambda_z. |
| r-squared | R-squared of Lambda_z computation. |

#### NOTES:

- Additional parameters may be included as required.
- Lambda z is the terminal phase rate constant.

#### 8.2.4. Population Pharmacokinetic (PopPK) Analyses

A population PK analysis may be conducted. The plasma concentration-time data may be merged with historical data and analysed as part of a population PK meta-analysis. The timeline for these analyses will be independent of the analysis described in this RAP. To support this analysis a NONMEM-specific data file will be generated, the specifications of which are provided in Appendix 9: Population PK and Pharmacokinetic / Pharmacodynamic (or Biomarker) Analyses.

# 8.3. Pharmacodynamic and Biomarker Analyses

### 8.3.1. Overview of Planned Pharmacodynamic and Biomarker Analyses

The pharmacodynamic and biomarker analyses will be based on the Modified Intent-To-Treat populations (mITT, mITT1 and mITT2), unless otherwise specified. Biomarker data will be analysed for those subjects in the Modified Intent-To-Treat populations for whom a sample was obtained and analysed.

Table 7 provides an overview of the planned pharmacodynamic and Biomarker analyses, with full details of data displays being presented in Appendix 11: List of Data Displays.

Table 7 Overview of Planned Pharmacodynamic and Biomarker Analyses

| Endpoint | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | bsolu | | ı | | Change from Baseline | | | | | | |
| | | Stats Analysis Summ | | | | | <u>idual</u> | | | | | mary | Individua | |
| | T | F | L | T | F | F | L | Т | F | L | T | F | F | L |
| RAS Peptide Response | <u>s<sup>1</sup></u> | | | | | | | | | | | | | |
| Ang II | | | | Υ | Υ | Υ | Υ | <b>Y</b> 1 | <b>Y</b> 1 | | | | | |
| Ang(1-7) | | | | Υ | Υ | Υ | Υ | <b>Y</b> 1 | <b>Y</b> 1 | | | | | |
| Ang(1-5) | | | | Υ | Υ | Υ | Υ | <b>Y</b> 1 | <b>Y</b> 1 | | | | | |
| Other Biomarkers (Dise | ease E | Bioma | rkers | | | | | | | | | | | |
| Surfactant Protein D | | | | Υ | Υ | Υ | Υ | <b>Y</b> 1 | <b>Y</b> 1 | | | | | |
| <b>Ventilatory Parameters</b> | 2 | | | | | | | | | | | | | |
| Oxygen consumption (VO2) | | | | Υ | | | Υ | | | | | | | |
| Carbon Dioxide Production (CO2) | | | | Υ | | | Υ | | | | | | | |
| Total Tidal Volume | | | | Υ | | | Υ | | | | | | | |
| Inspiratory Tidal<br>Volume | | | | Υ | | | Υ | | | | | | | |
| Expiratory Tidal<br>Volume | | | | Υ | | | Υ | | | | | | | |
| Total Respiratory Time | | | | Υ | | | Υ | | | | | | | |
| Inspiratory Time | | | | Υ | | | Υ | | | | | | | |
| Expiratory Time | | | | Υ | | | Υ | | | | | | | |
| Duty Cycle | | | | Υ | | | Υ | | | | | | | |
| Mean Respiratory Flow | | | | Υ | | | Υ | | | | | | | |
| Respiratory Rate | | | | Υ | | | Υ | | | | | | | |
| RAS Peptides vs PASP | & Ox | ygen | Satur | ation <sup>3</sup> | 3 | | | | | | | | | |
| Ang II vs PASP | | | | | Υ | | | | | | | | | |
| Ang(1-7) vs PASP | | | | | Υ | | | | | | | | | |
| Ang(1-5) vs PASP | | | | | Υ | | | | | | | | | |
| Ang II vs Oxygen<br>Saturation | | | | | Υ | | | | | | | | | |
| Ang(1-7) vs Oxygen<br>Saturation | | | | | Υ | | | | | | | | | |
| Ang(1-5) vs Oxygen<br>Saturation | | | | | Υ | | | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Statistical analysis of RAS peptides and SPD to be performed for Part 2. Part 1 may also be analysed.
- 2. Parameters will be included in the same summary/figure/listing paging by RAS peptide where applicable
- 3. Scatter plots of x vs y for mITT population, panel by timepoint, include study part in a legend, one plot for PASP, one plot for Oxygen Saturation (page by RAS peptide).
- Unless otherwise stated as in #3, all tables and figures will be produced separately for the mITT1 and mITT2 populations. Listings will be produced based on the mITT population

# 8.3.2. Planned Pharmacodynamic and Biomarker Statistical Analyses

#### **Planned Statistical Analyses**

#### Endpoint(s)

- RAS Peptide Responses: Ang II, Ang(1-7), Ang(1-5)
- Disease Biomarker: Surfactant Protein D

#### **Model Specification**

- Refer to Section 7.2. Change from baseline in PD/Biomarker endpoints will be analysed in a
  manner similar to the primary endpoint PASP. Data will be assessed prior to analysis to
  confirm the need for any data transformations. Log transformation highly likely to be required.
- Analyses will be performed for Part 2. Part 1 may also be analysed.
- Repeated measures timepoints of interest will be:
- Pre-dose (T0)
- End of Infusion
- 15 min Post-dose (T1)
- 15-45 min Post-dose
- 60 min post chamber entry (T2)
- Immediately post exercise (T3)
- Immediately post chamber exit
- 30 mins post chamber exit (T4)
  - Posterior probabilities of interest may include:
  - AngII: probability that the ratio <1, <0.50 and <0.25, representing any, 50% and 75% greater reduction in AngII levels on GSK2586881 compared to placebo</li>
  - Ang(1-5) & Ang(1-7): probability that the ratio >1, >1.50 and >1.75, representing any, 50% and 75% greater increase in Ang(1-5) and Ang(1-7) levels on GSK2586881 compared to placebo
  - SPD: probability that the ratio <1, >1 and >1.5, representing any decrease, any increase and a 50% increase in SPD levels on GSK2586881 compared to placebo
  - Probability cut-offs may be re-assessed at the time of analysis

#### **Model Checking**

• Refer to Appendix 8: Model Checking and Diagnostics for Statistical Analyses

#### **Model Results Presentation**

• Summary tables for absolute by treatment and timepoint (as detailed above) (for Part 1 and

### **Planned Statistical Analyses**

Part 2)

- Listing of absolute data
- Individual subject profiles by treatment group and timepoint (for Part 1 and 2)
- Summary table of statistical analysis, adjusted change from baseline posterior medians and 95% credible intervals by treatment and timepoint, together with estimated posterior median treatment differences (GSK2586881 – Placebo) and 95% credible intervals for the change from baseline at ALL timepoints (not just T1 to T4), along with posterior probabilities of interest. (Part 2 and Part 1(as required))
- Figure of absolute data by timepoint (for Part 1 and 2)
- Figure of statistical analysis adjusted change from baseline medians and 95% credible intervals by treatment group and timepoint (Part 2 and Part 1(as required))

# 8.4. Pharmacokinetic / Pharmacodynamic Analyses

The pharmacokinetic/pharmacodynamic (PK/PD) analyses will be based on the mITT and mITT2 population, unless otherwise specified. For the RAS peptides, PASP and Oxygen Saturation endpoints, exploratory plots vs pharmacokinetic concentrations will initially be reviewed to identify endpoints where there is a potential trend. If there is evidence for a trend, further PK/PD analyses may be conducted. The timeline for these analyses will be independent of the analysis described in this RAP. To support this analysis a NONMEM-specific data file will be generated, the specifications of which are provided in Appendix 9: Population PK and Pharmacokinetic / Pharmacodynamic (or Biomarker) Analyses.

Table 8 provides an overview of the planned PK/PD analyses with further details of data displays being presented in Appendix 11: List of Data Displays. Details of missing data imputation specific to PK/PD graphics are provided in Section 10.5.2.

| Endpoint | | Absolute | | |
|---|---|---|---|---|
| | Sun | nmary | Indiv | ridual |
| | Т | F | F | L |
| RAS Peptide Ang II vs PK concentration | | Υ1 | | |
| RAS Peptide Ang(1-7) vs PK concentration | | Υ1 | | |
| RAS Peptide Ang(1-5) vs PK concentration | | <b>Y</b> 1 | | |
| PASP vs PK concentration | | Υ2 | | |
| PASP (T2 & T3) vs AUC(0.5-2.0) | | Y2 | | |

#### NOTES:

- Scatter plots, timepoints indicated by panel.
- 1. RAS peptides vs PK will form one graphic, page by RAS peptide. Study part will be identified by a different colour/symbol combination. To be produced for the mITT population.
- 2. Produced for Part 2 only (mITT2 population).
- T = Table, F = Figure, L = Listing, Y = Yes display generated.

## 9. REFERENCES

GlaxoSmithKline Document Number: 2016N283626\_00, The effects of GSK2586881 on the responses to acute hypoxia and exercise: Effective date: 23-Sep-2016

GlaxoSmithKline Document Number: 2016N283626\_01, The effects of GSK2586881 on the responses to acute hypoxia and exercise: Effective date: 24-Feb-2017

GlaxoSmithKline Document Number: 2016N283626 02, The effects of GSK2586881 on the

responses to acute hypoxia and exercise: Effective date: 07-Mar-2017

GlaxoSmithKline Document Number: 2016N283626\_03, The effects of GSK2586881 on the

responses to acute hypoxia and exercise: Effective date: 06-Mar-2018

# 10. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 5 | : General Considerations for Data Analyses & Data Handling Conventions |
| Section 10.1 | Appendix 1: Time and Events |
| Section 10.2 | Appendix 2: Treatment States |
| Section 10.3 | Appendix 3: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 10.4 | Appendix 4: Derived and Transformed Data |
| | General, Study Population & Safety |
| | Pharmacodynamic and or Biomarkers |
| Section 10.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Section 10.6 | Appendix 6: Values of Potential Clinical Importance |
| Section 10.7 | Appendix 7: Biomarker Details |
| Section 10.8 | Appendix 8: Model Checking and Diagnostics for Statistical Analyses |
| Section 10.9 | Appendix 9: Population PK and Pharmacokinetic / Pharmacodynamic (or |
| | Biomarker) Analyses |
| Other RAP App | endices |
| Section 10.10 | Appendix 10: Abbreviations & Trade Marks |
| Section 10.11 | Appendix 11: List of Data Displays |
| Section 10.12 | Appendix 12: Example Mock Shells for Data Displays |

# 10.1. Appendix 1: Time & Events

# 10.1.1. Protocol Defined Time & Events

# 10.1.1.1. Screening and Follow up

| Procedure | Screening <sup>1</sup><br>(up to 28 days prior to<br>Treatment Period 1, Day 1) | Follow up<br>(7-10 days post<br>last dose) | Notes |
|---|---|---|---|
| Informed consent | X | | |
| Inclusion and exclusion criteria | X | | |
| Demography | X | | |
| Full physical exam, including height and weight | X | Х | Height and weight to be measured at screening only. Weight at screening will be used for dosing calculation. |
| Alcohol, Drugs of Abuse, Smoking test | X | | |
| Medical history (includes substance usage | X | | Substances: Drugs, Alcohol, tobacco |
| [and family history of premature CV disease]) | | | |
| Past and current medical conditions [including | X | | |
| cardiovascular medical history] | | | |
| Serum OR urine pregnancy test (WCBP) | X | | |
| HIV, Hep B and Hep C screen | X | | |
| Laboratory assessments (include liver | X | Χ | Non Fasting |
| chemistries) | | | |
| Immunogenicity | | Χ | |
| 12-lead ECG | X | Χ | Triplicate ECG required at screening. |
| Vital signs | X | Х | Triplicate vital signs required at screening. |
| Spirometry | X | | |
| Echocardiogram | X | | |
| Concomitant Medication review | X | Х | |
| Hypoxia chamber plus exercise | X | | Part 1: Tolerance to 4000m for 10 mins followed by incremental exercise testing to determine maximum oxygen uptake (VO2max) and calculate 70% of VO2max (to be used for the exercise challenge during the Treatment Periods). Part 2: Tolerance to 5000m for 10 mins followed by incremental exercise testing to determine maximum oxygen uptake (VO2max) and calculate 50% of |

| Procedure | Screening <sup>1</sup> (up to 28 days prior to Treatment Period 1, Day 1) | Follow up<br>(7-10 days post<br>last dose) | Notes |
|---|---|---|---|
| | | idot docoj | VO2max (to be used for the exercise challenge during the Treatment Periods) |
| Pharmacogenetic sample (PGx) | X | | Can be taken any time after consent has been signed. Only required once and is optional. |
| AE/SAE review | X | Х | As per timings detailed in protocol Section 7.2.1.1 |

<sup>1.</sup> Screening assessments are allowed to be conducted on more than one day

## 10.1.1.2. Treatment Period 1 and 2

| | | | | Tre | atmei | nt Perio | d 1 and | l 2 (Washou | ut 3-14 c | days) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Times relative to start of dosing | | | | Нур | oxic Cl<br>mes rel | hallenge | e ~80 min<br>entry to | | , | | Notes |
| Procedure | Pre-dose | 40 | 15 min | 15-45 min | 0-60 min | 60 min | 60-70 min | Immediately after<br>exercise | On exit from chamber | After 30 min rest | 60 min after exit<br>from Chamber | |
| Randomisation | Х | | | | | | | | | | | Treatment Period 1 only. Randomisation can occur up to the day before the first treatment period |
| Brief physical exam | Χ | | | | | | | | | | | |
| Vital signs | Χ | | | Χ | | | | χ5 | | | Х | |
| Immunogenicity | Χ | | | | | | | | | | | |
| 12-lead ECG | Χ | | | Χ | | | | | | | Х | |
| Echocardiogram | Χ | | Χ | | | Χ | | X6 below | | Х | | |
| Subject enters chamber | | | | | Х | | | | | | | Subject enters chamber approximately 30 min after study treatment |
| Study Treatment (Dosing) | | Χ | | | | | | | | | | |
| Subject leaves chamber | | | | | | | | Х | | | | Subject leaves chamber after the fourth echocardiogram, blood samples and vital signs have been taken. |
| Exercise challenge | | | | | | | X | | | | | Part 1: exercise at 70% VO2 max for ~5-10 min. Echo conducted immediately after. Part 2: exercise at 50% VO2 max for 2 min. Echo started at 2 min into the challenge, and the subject continues exercising. |
| Ventilatory parameters | Χ | | Х | | | Х | | | | Х | | Measurements to be taken 2 min before echocardiograms. |

| | Treatment Period 1 and 2 (Washout 3-14 days) | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | mes rel<br>tart of | | | | mes rel | | e ~80 min<br>entry to<br>) | | | | Notes |
| Procedure | Pre-dose | 0h | 15 min | 15-45 min | 0-60 min | 60 min | 60-70 min | Immediately after<br>exercise | On exit from chamber | After 30 min rest | 60 min after exit<br>from Chamber | |
| Pulse Oximetry<br>(O2 saturation) | <b>←</b> = | ===== | :=== | ==== | :===: | ===== | ===== | ====== | ===== | | =====> | Will be continuously monitored for safety. A measurement should be recorded at time of each echocardiogram and databased. Part 2: when the echo is recorded during the exercise challenge, pulse oximetry will be recorded immediately prior to initiation of the echo at 2 minutes into exercise. |
| Telemetry | <b>←</b> = | | ==== | | ==== | | ===== | ======= | ===== | | =====> | Will be continuously monitored for safety. |
| RAS Biomarkers | Χ | X <sup>1</sup> | X <sup>2</sup> | X <sup>3</sup> | | X <sup>2</sup> | | X <sup>2</sup> | X <sup>4</sup> | X <sup>2</sup> | | |
| SP-D | Χ | X <sup>1</sup> | X <sup>2</sup> | X <sup>3</sup> | | X <sup>2</sup> | | X <sup>2</sup> | X <sup>4</sup> | X <sup>2</sup> | | |
| PK sampling | Χ | X <sup>1</sup> | X <sup>2</sup> | X <sup>3</sup> | | X <sup>2</sup> | | X <sup>2</sup> | X <sup>4</sup> | X <sup>2</sup> | | |
| AE/SAE review | | <b>←==</b> | | ==== | ==== | ===== | | | ===== | | =====> | |
| Concomitant medication review | Χ | | | | | | | | | | | |

- 1. Take at the end of the infusion

- Taken immediately after echocardiogram
   Immediately before entering the chamber
   To be taken as soon as possible after leaving chamber
   On this occasion ONLY, vital signs to be taken after the blood draw.
   In Part 2, echo at this time-point taken 2 minutes into the exercise challenge (not immediately after exercise).

# 10.2. Appendix 2: Treatment States

#### 10.2.1. Treatment States for AE Data

This study is a single dose two period crossover study. As such, AEs will be attributed to the treatment received within the relevant study period based on the dates and times of the AEs in relation to dosing date and time. This is as per IDSL dataset standards. This is detailed in the table below.

#### 10.2.1.1. Treatment States for AE Dates

| Treatment State | Definition |
|---|---|
| | AE Start Date / Time < Study Treatment Start Date / Time (Period 1) |
| Pre-Treatment | This will apply to all subjects enrolled into the study, including those not randomised. We may have non-randomised and randomised subjects who have pre-treatment AEs/SAEs. For non-randomised subjects these events will be captured in the 'non-randomised' listing. For randomised subjects these events will be captured in summary listings with treatment group='Pre-Treatment'. |
| On-Treatment (Period 1) | If AE Start Date / Time is on or after Study Treatment Start Date / Time (Period 1) & before Study Treatment Start Date / Time (Period 2). Study Treatment Start Date / Time (Period 1) ≤ AE Start Date / Time < Study Treatment Start Date / Time (Period 2) |
| | For randomised subjects, this derivation ensures that AEs starting on or after the Period 1 dose up until the Period 2 dose will be captured and assigned to the Period 1 treatment. |
| On-Treatment (Period 2) | If AE Start Date / Time is on or after Study Treatment Start Date / Time (Period 2) & before Follow-Up. Study Treatment Start Date / Time (Period 2) ≤ AE Start Date / Time ≤ Follow-Up Date |
| | For randomised subjects, this derivation ensures that AEs starting on or after the Period 2 dose up until the Follow-up Visit will be captured and assigned to the Period 2 treatment. |
| Post-Treatment | If AE Start Date is on or after Follow-Up. AE Start Date > Follow-Up Date |
| | There shouldn't be any instances of this. Subjects will return for a follow-up and visit and any AEs would be documented at that point (and hence included in Period 2 treatment group). No further follow-up of patients is required. |
| Onset Time Since 1st<br>Dose (Days/Hours/Mins) | If Study Treatment Start Date / Time (Period 1) ≤ AE Start Date / Time = AE Start Date / Time – Study Treatment Start Date / Time (Period 1) + 1 (min) Missing otherwise. |
| | A calculation to assess the time since the Period 1 dose up until the start time of |

| | nition |
|---|---|
| the A Example If Pe start 1h 1 If Pe occu | AE. This will be calculated for all AEs, regardless of which period/treatment AE was assigned to. mple: eriod 1 Dose was administered at 08:00am 01OCT2016 and Period 1 AE red at 09:10am 01OCT2016, then onset time since <b>first</b> dose would be 0d 1m. eriod 2 Dose was administered at 08:30am 08OCT2016 and a Period 2 AE urred on 08OCT2016 at 10:00am, then onset time since <b>first</b> dose would be 1h 1m. |
| Dose (Days/Hours/Mins) If AE 1) & = AE [PEI If AE 2) & = AE Miss A ca to w Exan [PEI If Pei start 0d 1 [PEI If Pei occurrence | EStart Date / Time is on or after Study Treatment Start Date / Time (Period before Study Treatment Start Date / Time (Period 2). EStart Date / Time – Study Treatment Start Date / Time (Period 1) +1 (min) RIOD 2] EStart Date / Time is on or after Study Treatment Start Date / Time (Period on or before Follow-Up. EStart Date / Time – Study Treatment Start Date / Time (Period 2) + 1 (min) Sing otherwise. Ilculation to assess the time since the dose in the relevant Period/treatment hich the AE is attributable to. Imple: RIOD 1] Period 1 Dose was administered at 08:00am 01OCT2016 and Period 1 AE and at 09:10am 01OCT2016, then onset time since period dose would be the 11m (i.e. identical to value in previous row example in this case) RIOD 2] Period 2 Dose was administered at 08:30am 08OCT2016 and a Period 2 AE arred on 08OCT2016 at 10:00am, then onset time since period dose would be 11m (11m) |
| (Days/Hours/Mins) Example AEs | Resolution Date / Time – AE Start Date / Time + 1 (min) mple: started at 08:00am and resolved at 08:30am on the same day, then duration ld be 0d 0h 31m |
| | ationship is marked 'YES' on eCRF OR value is missing |

#### 10.2.2. Treatment States for Concomitant Medication Data

This study is a single dose two period crossover study. As such, Concomitant Medications will be attributed to the treatment received within the relevant study period based on the dates and times of the Concomitant Medications in relation to dosing date and time. This is as per IDSL dataset standards. This is detailed in the table below.

# 10.2.2.1. Treatment States for Concomitant Medication Dates

| Treatment State | Definition |
|---|---|
| Pre-Treatment | CM Start Date / Time < Study Treatment Start Date / Time (Period 1) |
| On-Treatment (Period 1) | If CM Start Date / Time is on or after Study Treatment Start Date / Time (Period 1) & before Study Treatment Start Date / Time (Period 2). Study Treatment Start Date / Time (Period 1) ≤ CM Start Date / Time < Study Treatment Start Date / Time (Period 2) |
| | For randomised subjects, this derivation ensures that CMs starting on or after the Period 1 dose up until the Period 2 dose will be captured and assigned to the Period 1 treatment group. |
| On-Treatment (Period 2) | If CM Start Date / Time is on or after Study Treatment Start Date / Time (Period 2) & before Follow-Up. Study Treatment Start Date / Time (Period 2) ≤ CM Start Date / Time ≤ Follow-Up Date |
| | For randomised subjects, this derivation ensures that CMs starting on or after the Period 2 dose up until the Follow-up Visit will be captured and assigned to the Period 2 treatment. |
| Study Day | Should relate to day since first dose i.e the day of the dose administered during Period 1 should be 'Day 1'. |
| Period Day | Day within the treatment period, for example, Period 1 Day 1 or Period 2 Day 1 |
# 10.3. Appendix 3: Data Display Standards & Handling Conventions

### 10.3.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| RandAll NG Data Displays for Reporting | | ng | |
| Code | Description | Description | Order [1] |
| Α | Placebo | Placebo | 1 |
| В | GSK2586881 0.8 mg/kg | GSK2586881 0.8 mg/kg | 2 |

<sup>1.</sup> Order represents treatments being presented in TFL, as appropriate.

### 10.3.2. Baseline Definition & Derivations

### 10.3.2.1. Baseline Definitions

For all endpoints (expect as noted in baseline definitions) the baseline value will be the latest predose assessment. Baseline definitions are applicable to <u>each period</u>.

| Parameter | Study Assessments Considered As Baseline | | Baseline Used in |
|---|---|---|---|
| | Screening | Day 1 (Pre-Dose) Time T0 | Data Display |
| Safety | Safety | | |
| PASP | X | X | T0 |
| Oxygen Saturation | | X | T0 |
| Labs | X | | Screening |
| ECGs | X <sup>1</sup> | X | T0 |
| Vital Signs | <b>X</b> <sup>1</sup> | X | T0 |
| Biomarkers/Pharmacodynamic | | | |
| RAS peptides | | X | T0 |
| Other biomarkers | | X | T0 |
| Ventilatory parameters | | X | T0 |

<sup>&</sup>lt;sup>1</sup>Unless otherwise stated, the mean of replicate assessments at any given time point will be used as the value for that time point.

For statistical analyses (for example, Bayesian mixed model for PASP):

- Baseline is defined as the measurement taken pre-dose during each treatment period (i.e., time T0). This can also be referred to as 'period-specific baseline'.
- **Subject-level baseline** is defined as the mean of the two period-specific baseline readings (the pre-dose T0 reading from each of the two treatment periods) for each subject.

 Period-level baseline (or 'adjusted period-specific baseline') is defined as the difference between the baseline ('period-specific baseline') and 'subject-level baseline' for each period and each subject (i.e., the 'period-specific baseline' minus 'subject-level baseline' in each period).

The statistical modelling will include terms for 'subject-level baseline' and 'adjusted period-specific baseline'.

### 10.3.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|----------------------|----------------------------------------------|
| Change from Baseline | = Post-Dose Visit Value – Baseline [Ti – T0] |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 10.3.2.1 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

### 10.3.3. Reporting Process & Standards

| Reporting Process | Reporting Process |
|---|---|
| Software | |
| Generate tables, | The currently supported versions of SAS software will be used to perform all data analyses. Generate tables, figures and listings. |
| | n of R (or alternative supported available packages) will be used in sample n for the interim analysis |
| Reporting Area | |
| HARP Server | : UK1SALX00175.corpnet2.com |
| HARP Area | : \ARPROD\GSK2586881\204987\Internal_01 |
| | : \ARPROD\GSK2586881\204987\Internal_02 |
| | : \ARPROD\GSK2586881\204987\Final_01 |
| QC Spreadsheet | : \ARWORK\GSK2586881\204987\Internal_01\documents |
| | : \ARWORK\GSK2586881\204987\Internal_02\documents |
| | : \ARWORK\GSK2586881\204987\Final_01\documents |
| Analysis Datasets | |
| <ul> <li>Analysis datasets will be created according to Legacy GSK A&amp;R dataset standards (Integrated<br/>Data Standards Library)</li> </ul> | |
| • RAS Peptide data samples for Ang II, Ang(1-5) and Ang(1-7) will be processed by Q2 and data | |

- RAS Peptide data samples for Ang II, Ang(1-5) and Ang(1-7) will be processed by Q2 and data provided to GSK Data Management.
- Surfactant Protein D samples and Immunogenicity samples will be processed by GSK and data will be provided to GSK Data Management
- Pharmacokinetic samples will be processed by Covance and data will be provided to GSK Data Management

### **Generation of RTF Files**

RTF files will be generated for the interim and final reporting efforts

### **Reporting Standards**

### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - o 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses :
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

### **Unscheduled Visits**

Descriptive

- Unscheduled visits will not be included in summary tables or figures, unless otherwise stated.
- All unscheduled visits will be included in listings

| 7 th disorication visits will be included in listings. | |
|---|---|
| Descriptive Summary Statistics | |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Descriptive Summary Statistics (Log Transformed Data) | N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data and between geometric coefficient of variation (CV <sub>b/w</sub> (%)): $CV_b$ (%) = $\sqrt{\exp(SD^2) - 1}$ * 100 (NOTE: SD is the SD of log transformed data) |
| Reporting of Pharmacokinetic Concentration Data | |
| Descriptive | Refer to IDSL Statistical Principle 6.06.1 |
| Summary Statistics | Assign zero to NQ values (Refer to GUI_51487 for further details) |
| Reporting of Pharmacokinetic Parameters | |

N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD)

| Reporting Standards | |
|---|---|
| Summary Statistics | of logged data and [between and or within] geometric coefficient of variation |
| (Log Transformed) | (CVb/w (%)) will be reported. |
| | [1] $CV_b$ (%) = $\sqrt{(exp(SD^2) - 1) * 100}$ |
| | (SD = SD of log transformed data) |
| | [2] $CV_w$ (%) = $\sqrt{(exp(MSE) - 1) * 100}$ |
| | (MSE = mean square error from mixed effect model of loge-transformed data). |
| Parameters Not | Tmax, first point, last point and number of points used in the determination of |
| Being Log | lambda_z for listings |
| Transformed | |
| Listings | Include the first point, last point and number of points used in the |
| | determination of lambda_z for listings and R squared |
| Graphical Displays | |
| Refer to IDSL Statistical Principles 7.01 to 7.13. | |

### 10.4. Appendix 4: Derived and Transformed Data

### 10.4.1. **General**

### **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target then the mean will be taken.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

### **Study Day**

- Calculated as the number of days from randomisation date :
  - Ref Date = Missing
     → Study Day = Missing
  - Ref Date < Randomisation Date → Study Day = Ref Date Randomisation Date
  - Ref Data ≥ Randomisation Date → Study Day = Ref Date (Randomisation Date) + 1

### 10.4.2. Study Population

### **Demographics**

### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)]<sup>2</sup>

### **Extent of Exposure**

- Number of days of exposure to study drug will be calculated based on the formula:
   Duration of Exposure in Days = Treatment Stop Date (Treatment Start Date) + 1
- Subjects who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.

### 10.4.3. Safety

### **ECG Parameters**

### **RR Interval**

• IF RR interval (msec) is not provided directly, then RR can be derived as :

[1] If QTcB is machine read & QTcF is not provided, then:

$$RR = \left[ \left( \frac{QT}{OTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

 If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.

#### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fridericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as :

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01</li>
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1</li>

# 10.4.4. Pharmacodynamic and Biomarker

### **Biomarkers**

### **RAS Peptides**

Ang II, Ang(1-5), Ang(1-7)

### **Disease Biomarker**

Surfactant Protein D

Variance stabilising transformations (e.g. taking natural logarithms of the observed responses) may be implemented on a per endpoint basis, if deemed necessary by the study statistician. If transformations are used the results will be reported on the back-transformed response scales.

# 10.5. Appendix 5: Premature Withdrawals & Handling of Missing Data

# 10.5.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as any subject who completes all phases in the study including the follow-up visit.</li> <li>Withdrawn subjects will not be replaced in the study.</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 10.5.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument : |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing<br/>displays. Unless all data for a specific visit are missing in which case the<br/>data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to<br/>be missing data and should be displayed as such.</li> </ul> |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |
| PK | If dosing and/or sampling times are missing, the relevant concentrations will be deleted from the population PK and PK/PD analysis dataset and summarized in a deletion record listing. Samples listed as having no sample (NS), no result (NR) or insufficient sample (IS) will be excluded from the PK data set and also included in the deletion record listing. GSK2586881 concentrations below the lower limit of quantification (LLQ) for the assay will be reported as NQ (Below Quantification Limit). All NQ values will be set to "." (missing) in the population PK and PK/PD dataset. Individuals with all plasma concentrations reported as NQ will be included in the data set. |
| | For PK/PD graphics only which are generated by S&P, ½ LLQ can be used for NQ PK data to coincide with methods used for Biomarker data as below. Variables relating to different imputation methods for PK data will be available within the derived A&R PKCNC dataset (e.g. differentiating between setting NQ values to missing or ½ LLQ). |
| Biomarkers | Any values below the Lower Limit of Quantification (LLQ) will be assigned a value of ½ LLQ for display purposes in Figures and for computation of summary statistics. Any values above the Upper Limit of Quantification (ULQ) will be assigned to the ULQ for display purposes in Figures and for computation of summary statistics. If multiple LLQ and /or ULQ values are available per assay |

| Element | Reporting Detail |
|---|---|
| | (for example if multiple runs with different standard curves are utilised) then the LLQ and/or ULQ value used for the above imputation shall be the minimum of the available LLQs and/or the maximum of the ULQs. |
| | If the number of LLQ (and/or ULQ) values is large for an individual biomarker then alternative analysis strategies may be required. "Large" is hard to define prospectively and may depend upon the dataset in question but a general rule of thumb is if >30% of values are LLQ and/or ULQ. If "large" numbers of LLQ and/or ULQ values are observed methodologies to summarise and analyse the responses similar to those detailed in "Standards for the Handling of NQ impacted PK Parameters" (Respiratory DB and CPMS - 14th December 2009) may be employed. Any such methodology will be documented in the statistical contributions to the clinical study report. |

# 10.5.2.1. Handling of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Treatment States and Phases.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> <li>Start or end dates which are completely missing (i.e. no year specified) will remain missing, with no imputation applied.</li> </ul> |

# 10.5.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant Medications | Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: |
| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will<br/>be used for the month</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day<br/>(dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | The recorded partial date will be displayed in listings. |

| Element | Reporting Detail |
|---|---|
| Adverse<br>Events | Any partial dates for adverse events will be raised to data management. If the full date cannot be ascertained, the following assumptions will be made: • If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month. |
| | <ul> <li>However, if these results in a date prior to Week 1 Day 1 and the event could possibly have occurred during treatment from the partial information, then the Week 1 Day 1 date will be assumed to be the start date.</li> <li>The AE will then be considered to start on-treatment (worst case).</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day<br/>(dependent on the month and year) and 'Dec' will be used for the month.</li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 10.5.2.3. Handling of Missing Data for Statistical Analysis

No missing data imputation methods will be used.

# 10.6. Appendix 6: Values of Potential Clinical Importance

# 10.6.1. Laboratory Values

Laboratory parameters have been reviewed against those specified in the protocol and any parameters not specified here have been assigned as not essential for assessment.

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Llomotoprit | Ratio of | Male | | 0.54 |
| Hematocrit | 1 | Female | | 0.54 |
| Homoglobin | g/L | Male | | 180 |
| Hemoglobin | | Female | | 180 |
| Lymphocytes | x109/ L | | 0.8 | |
| Neutrophil Count | x109/ L | | 1.5 | |
| Platelet Count | x109/ L | | 100 | 550 |
| While Blood Cell Count (WBC) | x109/ L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | 30 | |
| BUN | mmol/L | | | ≥ 2x ULN |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | mmol/L | | | ≥ 1.3x ULN |
| Glucose | mmol/L | | 3 | 9 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | μmol/L | High | ≥ 1.5xULN |
| | μmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

# 10.6.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|----------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | ≥ 500 | |
| Absolute PR Interval | msec | < 110 | > 220 |
| Absolute QRS Interval | msec | < 75 | > 110 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | > 60 | |

# 10.6.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

| Vital Sign Parameter | Units | Clinical Concern Range | | | | |
|---|---|---|---|---|---|---|
| (Change from Baseline) | | Decrease Increas | | Decrease Increase | | ease |
| | | Lower | Upper | Lower | Upper | |
| Systolic Blood Pressure | mmHg | ≥ 20 | ≥ 40 | ≥ 20 | ≥ 40 | |
| Diastolic Blood Pressure | mmHg | ≥ 10 | ≥ 20 | ≥ 10 | ≥ 20 | |
| Heart Rate | bpm | ≥ 15 | ≥ 30 | ≥ 15 | ≥ 30 | |

# 10.7. Appendix 7: Biomarker Details

| Biomarker<br>Category | Analyte | Method | Lab | Matrix | Total samples expected per subject |
|---|---|---|---|---|---|
| RAS Peptides <sup>1</sup> | Ang II | LCMS | Q2 | Blood | 8 |
| (key | Ang (1-5) | LCMS | Q2 | Blood | 8 |
| endpoints) | Ang (1-7) | LCMS | Q2 | Blood | 8 |
| Disease<br>Biomarkers | Surfactant Protein D | Elisa | GSK | Serum | 8 |

### NOTES:

- 1. These peptides will be included in the interim analysis.
- Sampling times for each period: Pre-dose (T0), End of Infusion, 15 min Post-dose (T1), 15-45 min Post-dose, 60 min post chamber entry (T2), immediately post exercise (T3), immediately post chamber exit, 30 mins post chamber exit (T4).

# 10.8. Appendix 8: Model Checking and Diagnostics for Statistical Analyses

# Endpoint(s) PASP Oxygen Saturation RAS Peptides (AngII, Ang(1-5), Ang(1-7)) Surfactant Protein D Analysis SAS PROC MCMC: Bayesian repeated measures mixed model

- Fixed effects will be assigned a non-informative prior of N(0, Var=1E6) and may be entered as separate univariate priors or as part of a multivariate distribution (variance covariance structure with zeros for off diagonals) in model hyperpriors.
- The non-informative UN priors should be an inverse Wishart distribution. If the equivalent of an unstructured variance covariance matrix does not fit then an AR(1) w/Random Effect structure may be considered, with non-informative priors φ~U[-1,1] for the off diagonal elements and σ² ~ invGamma(0.0001, scale=0.0001). Example, for N=3:

$$UN = \begin{pmatrix} \sigma_{1}^{2} & \sigma_{21} & \sigma_{31} \\ \sigma_{21} & \sigma_{2}^{2} & \sigma_{32} \\ \sigma_{31} & \sigma_{32} & \sigma_{3}^{2} \end{pmatrix}$$
$$AR(1) = \begin{pmatrix} 1 & \phi & \phi^{2} \\ \phi & 1 & \phi \\ \phi^{2} & \phi & 1 \end{pmatrix} * \sigma^{2}$$

- Appropriate SAS helper procedures (e.g. PROC TRANSREG) may be used to convert typical "long and thin" PROC MIXED input datasets into a format appropriate for repeated measures modelling in PROC MCMC (e.g. constructing sets of factors for each class level and fixing the final level to zero)
- Centring of continuous covariates will take place at the input dataset stage: (valuei average) for each subject i.
- Examination of trace plots of samples versus the simulation number and Geweke diagnostics to assess convergence. Autocorrelation plots and lag summary table to assess the degree of autocorrelation. Monte Carlo standard errors compared to posterior standard deviations (a rule of thumb but not binding target would be <0.05). If further diagnostics required a scatterplot matrix plot of the posterior samples of each parameter.
- Number of burn ins, thinning, starting points, number of posterior draws to take (10,000 as a starting default) will be customised to each model and may not be possible to specify in advance but will be modified to ensure satisfactory diagnostics are produced.
- For robustness, where non-informative priors are used the equivalent PROC MIXED model
  may be fitted (no output from this would be reported) and LS Means and estimates of
  treatment differences compared to the results obtained from the PROC MCMC analysis. SAS
  code for the random and repeated statements would be:

random int / subject=subjid s vcorr;

repeated visit / subject=subjid\*ptrtgrp type=un r rcorr;

 Model assumptions will be applied, but appropriate adjustments may be made based on the data.

# 10.9. Appendix 9: Population PK and Pharmacokinetic / Pharmacodynamic (Or Biomarker) Analyses

### 10.9.1. Population PK Dataset File Structure

The PME compliant file structure is a space-delimited file with each row containing the following columns of information. Data from all active treatments will be included (i.e. exclude placebo).

Decision as to whether this will be required will be made following the planned interim analysis (for study Part 2 at approximately N=3 or approximately N=6).

Note that subject numbers up to and including PP were enrolled into Part 1 of the study. Subject numbers from PP onwards will be enrolled into Part 2 of the study.

| Variable<br>short<br>name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| С | Data Identifier | Integer | - | 0 |
| STUD | Protocol Number | Integer | - | 204987 |
| DRUG | Name of Drug | Integer | - | Maximum 10 characters (numeric or text). 2586881 |
| SUBJ | Subject identifier in study | Integer | - | Maximum 10 characters (numeric or text). Different identifier for each subject |
| CENT | Study centre identifier | Integer | - | |
| LABL | Indicator field describing the type of assessment in that record | Integer | See<br>footnotes | See footnotes |
| AMT | Dose of<br>GSK2586881 | Decimal | Mg | Amount of drug given = Total GSK2586881 dose (mg/kg)* WT For dosing events: total dose of GSK2586881 taken For concentration events: 0 |
| INF | Infusion Time | Decimal | h | Time during which total dose infused. (Time at end of infusion – Time of start infusion) |
| RATE | Rate of Infusion | Decimal | Mg/h | Rate of infusion (AMT/INF) |
| DGRP | Treatment Identifier | Decimal | - | DGRP=0.8 for 0.8 mg/kg treatment<br>Dose of GSK2586881 (for all events) |
| PART | Study Part | Integer | - | 1=Part 1 or 2=Part 2 |
| PERIOD | Study Period | Integer | - | 1=Period 1 or 2=Period 2 |
| DAY | Study day | Integer | - | Maximum 10 characters (numeric or text) N= Day N, Actual Study Day |
| CTIM | Clock Time of<br>Event | HH:MM:SS | - | Clock Time of Event |
| DATE | Date of Record | (DD/MM/YYYY) | - | Date of Record |

| Variable | Assessment | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| short<br>name | description | | | |
| TRFD | Actual time relative | Decimal | Hours | When LABL = 4, TIME = 0 |
| | to FIRST dose | | | Hours since start of first active infusion |
| | | | | (on Day 1). For pre-dose sample, TRFD |
| | | | | is relative to FIRST dose/infusion |
| TRLD | Actual time relative | Decimal | Hours | When LABL = 4, TIME = 0 |
| | to LAST dose | | | Hours since start of LAST infusion. For |
| | | | | pre-dose sample, TRLD is relative to |
| | | | | previous dose prior to sample |
| | | | | For single dose studies TRFD and TRLD are the same |
| TFLAG | Time Flag | Integer | _ | At T0 and LABL=6, TFLAG=0 |
| 11 27 (0 | Timo Tiag | intogo. | | At T1 and LABL=6, TFLAG=1 |
| | | | | At T2 and LABL=6, TFLAG=2 |
| | | | | At T3 and LABL=6, TFLAG=3 |
| | | | | At T4 and LABL=6, TFLAG=4 |
| | | | | Otherwise if LABL=6, TFLAG=5 |
| | | | | If LABL="0" or "4", TFLAG=6 |
| DV | Dependent Variable | Decimal | pg/mL | When LABL=6, observed GSK2586881 |
| | | | | concentration at time specified by TRLD. |
| MDV | NA: : D ( | 1.6 | | When LABL=4 (dosing record), DV=0 |
| MDV | Missing Data | Integer | - | Either '0' if DV value present or 1 if DV |
| | Variable | | | value is non-quantifiable (NQ) or LABL=4 |
| MDV1 | Missing data | Integer | | Either '0' if LABL=6 or '1' if LABL=4 |
| | variable | intogor | | |
| TYPE | F-Flag | Integer | - | If MDV1='1' then TYPE ='0', |
| | | | | If DV value present (but not NQ) TYPE= |
| | | | | '1'<br>If DV value NQTYPE = '2' |
| LLQ | Lower Limit of | Integer | pg/mL | Lower limit of quantification for specific |
| | quantification | | рулпс | analyte SMS dataset (PCLLQ) |
| CMT | Compartment data | Integer | - | DOSE event: CMT=1, specifies the |
| | item | | | compartment into which DOSE is |
| | | | | introduced. OBSERVATION event: |
| | | | | CMT =1, specifies compartment from |
| AGE | Λαο | Decimal | Yrs | which observation is obtained. Integer. Age in years at time of |
| AGE | Age | Decimal | 115 | screening rounded down to give age at |
| | | | | last birthday. |
| WT | Weight | Decimal | Kg | Weight in kilograms at time of screening. |
| HT | Height | Decimal | Cm | Height in centimetres at time of |
| | | | | screening. |
| SEX | Subject gender | Integer | - | Integer. One of the following - |
| | | | | 1 = male |
| CTI IN | Outsiant attended | lata | | 2 = female |
| ETHN | Subject ethnicity | Integer | - | Integer. Code as CRF |
| RACE | Subject race | Integer | - | Integer. Code as CRF |

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| BMI | Body mass index | Decimal | kg/m^2 | body mass index calculated as weight divided by height squared |
| EVID | Event Identification data item | Integer | - | Flag indicating whether LABL contains dosing admin info or drug concentration data. Valid values are - 1 – each dosing record for subject 0 - for all other records |

### Assessments captured in the LABL variable

| Label | Description | Units |
|---|---|---|
| 4 | Dosing records for 0.8 mg/Kg GSK2586881 | |
| 6 | Observed concentration record for GSK2586881 at time specified by TRLD; excludes NA, IS and NR, includes non-quantifiable (NQ) data | pg/mL |

### 10.9.2. Population PK/PD Dataset File Structure : ANGII

The PME compliant file structure is a space-delimited file with each row containing the following columns of information. Data from all treatments will be included.

Decision as to whether this will be required will be made following the planned interim analysis (for study Part 2 at approximately N=3 or approximately N=6).

| Variable | Assessment | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| short name | description | | | |
| С | Data Identifier | Integer | - | 0 |
| STUD | Protocol Number | Integer | - | 204987 |
| DRUG | Name of Drug | Integer | - | Maximum 10 characters (numeric or text). 2586881 |
| SUBJ | Subject identifier in study | Integer | - | Maximum 10 characters (numeric or text). Different identifier for each subject |
| CENT | Study centre identifier | Integer | - | |
| LABL | Indicator field describing the type of assessment in that record | Integer | See<br>footnotes | See footnotes |
| AMT | Dose of<br>GSK2586881 | Decimal | Mg | Amount of drug given = Total<br>GSK2586881 dose (mg/kg) * WT.<br>AMT=0 when LABL=0 |

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| | | | | For dosing events: total dose of GSK2586881 taken For concentration events: 0 |
| INF | Infusion Time | Decimal | h | Time during which total dose infused. (Time at end of infusion – Time of start infusion) |
| RATE | Rate of Infusion | Decimal | Mg/h | Rate of infusion (AMT/INF) |
| DGRP | Treatment Identifier | Decimal | - | DGRP=0 for placebo treatment DGRP=0.8 for 0.8 mg/kg treatment Dose of GSK2586881 (for all events) |
| PART | Study Part | Integer | - | 1=Part 1 or 2=Part 2 |
| PERIOD | Study Period | Integer | - | 1=Period 1 or 2=Period 2 |
| DAY | Study day | Integer | - | Maximum 10 characters (numeric or text) N= Day N, Actual Study Day |
| CTIM | Clock time of Dose or measurement | HH:MM:SS | - | |
| DATE | Date of record | DD/MM/YYY | | |
| TRFD | Actual time relative to FIRST dose | Decimal | Hours | When LABL=0 or 4, TIME =0 Hours since start of FIRST infusion (on Day 1). For pre-dose sample, TRFD is relative to FIRST dose |
| TRLD | Actual time relative to LAST dose | Decimal | Hours | When LABL=0 or 4, TIME=0 Hours since start of LAST dose/infusion. For pre-dose sample,TRLD is relative to previous dose For single dose studies TRLD = TRFD |
| TFLAG | Time Flag | Integer | - | At T0 and LABL=6, TFLAG=0 At T1 and LABL=6, TFLAG=1 At T2 and LABL=6, TFLAG=2 At T3 and LABL=6, TFLAG=3 At T4 and LABL=6, TFLAG=4 Otherwise if LABL=6, TFLAG=5 If LABL="0" or "4", TFLAG=6 |
| BLII | AnglI concentration record | Decimal | | Baseline value (pre-dose value) |
| DV | Angll concentration record | Decimal | | When LABL=6, observed AngII concentration at time specified by TRLD. When LABL=0 or 4, AngII=0 |
| MDV | Missing data variable | Integer | - | Either '0' if DV value present or 1 if DV is non-quantifiable (NQ) value or LABL=0 or 4 |
| MDV1 | Missing data variable | Integer | - | '1' if LABL=0 or 4 "0" when LABL=6 |
| TYPE | F-Flag | Integer | - | If MDV1='1' then TYPE ='0', If DV value present (but not NQ) TYPE= '1' If DV value NQTYPE = '2' |
| CMT | Compartment data | Integer | - | DOSE event: CMT=1, specifies the |

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| | item | | | compartment into which DOSE is introduced. OBSERVATION event: CMT=3 for DV (ANGII) observation event. |
| AGE | Age | Decimal | Yrs | Integer. Age in years at time of screening rounded down to give age at last birthday. |
| WT | Weight | Decimal | Kg | Weight in kilograms at time of screening. |
| HT | Height | Decimal | Cm | Height in centimetres at time of screening. |
| SEX | Subject gender | Integer | - | Integer. One of the following - 1 = male 2 = female |
| ETHN | Subject ethnicity | Integer | - | Integer. Code as CRF |
| RACE | Subject race | Integer | - | Integer. Code as CRF |
| BMI | Body mass index | Decimal | kg/m^2 | body mass index calculated as weight divided by height squared |
| EVID | Event Identification data item | Integer | - | Flag indicating whether LABL contains dosing admin info or drug concentration data. Valid values are - 1 – each dosing record for subject 0 - for all other records |

### Assessments captured in the LABL variable

| Label | Description | Units |
|---|---|---|
| 0 | Dosing record for placebo | |
| 4 | Dosing records for 0.8 mg/Kg GSK2586881 | |
| 6 | Observed record (concentration or ratio) at time specified by TRLD; | |
| | excludes NA, IS and NR, includes non-quantifiable (NQ) data | |

### 10.9.3. Population PK/PD Dataset File Structure : ANG1-5

The PME compliant file structure is a space-delimited file with each row containing the following columns of information. Data from all treatments will be included.

Decision as to whether this will be required will be made following the planned interim analysis (for study Part 2 at approximately N=3 or approximately N=6).

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| С | Data Identifier | Integer | - | 0 |
| STUD | Protocol Number | Integer | - | 204987 |

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| DRUG | Name of Drug | Integer | - | Maximum 10 characters (numeric or text). 2586881 |
| SUBJ | Subject identifier in study | Integer | - | Maximum 10 characters (numeric or text). Different identifier for each subject |
| CENT | Study centre identifier | Integer | - | |
| LABL | Indicator field describing the type of assessment in that record | Integer | See<br>footnotes | See footnotes |
| AMT | Dose of<br>GSK2586881 | Decimal | Mg | Amount of drug given = Total GSK2586881 dose (mg/kg) * WT. AMT=0 when LABL=0 For dosing events: total dose of GSK2586881 taken For concentration events: 0 |
| INF | Infusion Time | Decimal | h | Time during which total dose infused. (Time at end of infusion – Time of start infusion) |
| RATE | Rate of Infusion | Decimal | Mg/h | Rate of infusion (AMT/INF) |
| DGRP | Treatment Identifier | Decimal | - | DGRP=0 for placebo treatment<br>treatment<br>DGRP=0.8 for 0.8 mg/kg treatment<br>Dose of GSK2586881 (for all events) |
| PART | Study Part | Integer | - | 1=Part 1 or 2=Part 2 |
| PERIOD | Study Period | Integer | - | 1=Period 1 or 2=Period 2 |
| DAY | Study day | Integer | - | Maximum 10 characters (numeric or text) N= Day N, Actual Study Day |
| CTIM | Clock time of Dose or measurement | HH:MM:SS | - | |
| DATE | Date of record | DD/MM/YYY | | |
| TRFD | Actual time relative to FIRST dose | Decimal | Hours | When LABL=0 or 4, TIME =0 Hours since start of FIRST infusion (on Day 1). For pre-dose sample, TRFD is relative to FIRST dose |
| TRLD | Actual time relative to LAST dose | Decimal | Hours | When LABL=0 or 4, TIME=0 Hours since start of LAST dose/infusion. For pre-dose sample,TRLD is relative to previous dose For single dose studies TRLD = TRFD |
| TFLAG | Time Flag | Integer | - | At T0 and LABL=6, TFLAG=0 At T1 and LABL=6, TFLAG=1 At T2 and LABL=6, TFLAG=2 At T3 and LABL=6, TFLAG=3 At T4 and LABL=6, TFLAG=4 Otherwise if LABL=6, TFLAG=5 |

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| | • | | | If LABL="0" or "4", TFLAG=6 |
| BL15 | Ang1-5 concentration record | Decimal | | Baseline value |
| DV | Angl1-5 concentration record | Decimal | | When LABL=6, observed Ang1-5 concentration at time specified by TRLD. When LABL=0or 4, Ang1-5=0 |
| MDV | Missing data variable | Integer | - | Either '0' if DV value present or 1 if DV is non-quantifiable (NQ) value or LABL=0 or,4 |
| MDV1 | Missing data variable | Integer | - | '1' if LABL=0 or 4 "0" when LABL=6 |
| TYPE | F-Flag | Integer | - | If MDV1='1' then TYPE ='0', If DV value present (but not NQ) TYPE= '1' If DV value NQTYPE = '2' |
| CMT | Compartment data item | Integer | - | DOSE event: CMT=1, specifies the compartment into which DOSE is introduced. OBSERVATION event CMT=5 for ANG1-5 observation event. |
| AGE | Age | Decimal | Yrs | Integer. Age in years at time of screening rounded down to give age at last birthday. |
| WT | Weight | Decimal | Kg | Weight in kilograms at time of screening. |
| HT | Height | Decimal | Cm | Height in centimetres at time of screening. |
| SEX | Subject gender | Integer | - | Integer. One of the following - 1 = male 2 = female |
| ETHN | Subject ethnicity | Integer | - | Integer. Code as CRF |
| RACE | Subject race | Integer | - | Integer. Code as CRF |
| BMI | Body mass index | Decimal | kg/m^2 | body mass index calculated as weight divided by height squared |
| EVID | Event Identification data item | Integer | - | Flag indicating whether LABL contains dosing admin info or drug concentration data. Valid values are - 1 – each dosing record for subject 0 - for all other records |

# Assessments captured in the LABL variable

| Label | Description | Units |
|---|---|---|
| 0 | Dosing record for placebo | |
| 4 | Dosing records for 0.8 mg/Kg GSK2586881 | |
| 6 | Observed record (concentration or ratio) at time specified by TRLD; excludes NA, IS and NR, includes non-quantifiable (NQ) data | |

# 10.9.4. Population PK/PD Dataset File Structure : ANG1-7

The PME compliant file structure is a space-delimited file with each row containing the following columns of information. Data from all treatments will be included.

Decision as to whether this will be required will be made following the planned interim analysis (for study Part 2 at approximately N=3 or approximately N=6).

| Variable | Assessment | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| short name | description | | | |
| С | Data Identifier | Integer | - | 0 |
| STUD | Protocol Number | Integer | - | 204987 |
| DRUG | Name of Drug | Integer | - | Maximum 10 characters (numeric or text). 2586881 |
| SUBJ | Subject identifier in study | Integer | - | Maximum 10 characters (numeric or text). Different identifier for each subject |
| CENT | Study centre identifier | Integer | - | |
| LABL | Indicator field describing the type of assessment in that record | Integer | See<br>footnotes | See footnotes |
| AMT | Dose of<br>GSK2586881 | Decimal | Mg | Amount of drug given = Total GSK2586881 dose (mg/kg) * WT. AMT=0 when LABL=0 For dosing events: total dose of GSK2586881 taken For concentration events: 0 |
| INF | Infusion Time | Decimal | h | Time during which total dose infused. (Time at end of infusion – Time of start infusion) |
| RATE | Rate of Infusion | Decimal | Mg/h | Rate of infusion (AMT/INF) |
| DGRP | Treatment Identifier | Decimal | - | DGRP=0 for placebo treatment<br>treatment<br>DGRP=0.8 for 0.8 mg/kg treatment<br>Dose of GSK2586881 (for all events) |
| PART | Study Part | Integer | - | 1=Part 1 or 2=Part 2 |
| PERIOD | Study Period | Integer | - | 1=Period 1 or 2=Period 2 |
| DAY | Study day | Integer | - | Maximum 10 characters (numeric or text) N= Day N, Actual Study Day |
| CTIM | Clock time of Dose or measurement | HH:MM:SS | - | |
| DATE | Date of record | DD/MM/YYY | | |
| TRFD | Actual time relative to FIRST dose | Decimal | Hours | When LABL=0 or 4, TIME =0 Hours since start of FIRST infusion (on Day 1). For pre-dose sample, TRFD is relative to FIRST dose |
| TRLD | Actual time relative to LAST dose | Decimal | Hours | When LABL=0 or 4, TIME=0<br>Hours since start of LAST<br>dose/infusion. For pre-dose |

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| | | | | sample,TRLD is relative to previous dose For single dose studies TRLD = |
| | | | | TRFD |
| TFLAG | Time Flag | Integer | - | At T0 and LABL=6, TFLAG=0 At T1 and LABL=6, TFLAG=1 At T2 and LABL=6, TFLAG=2 At T3 and LABL=6, TFLAG=3 At T4 and LABL=6, TFLAG=4 Otherwise if LABL=6, TFLAG=5 If LABL="0" or "4", TFLAG=6 |
| BL17 | Ang1-7 concentration record | Decimal | | Baseline value |
| ANG1-7 | Ang1-7 concentration record | Decimal | | When LABL=6, observed Ang1-7 concentration at time specified by TRLD. When LABL=0or ,4, DV=0 |
| MDV | Missing data variable | Integer | - | Either '0' if DV value present or 1 if DV is non-quantifiable (NQ) value or LABL=0 or 4 |
| MDV1 | Missing data variable | Integer | - | '1' if LABL=0 or 4<br>"0" when LABL=6 |
| TYPE | F-Flag | Integer | - | If MDV1='1' then TYPE ='0', If ANG1-7 value present (but not NQ) TYPE= '1' If ANG1-7 value NQTYPE = '2' |
| CMT | Compartment data item | Integer | - | DOSE event: CMT=1, specifies the compartment into which DOSE is introduced. OBSERVATION event: CMT=4 for ANG1-7 observation event. |
| AGE | Age | Decimal | Yrs | Integer. Age in years at time of screening rounded down to give age at last birthday. |
| WT | Weight | Decimal | Kg | Weight in kilograms at time of screening. |
| HT | Height | Decimal | Cm | Height in centimetres at time of screening. |
| SEX | Subject gender | Integer | - | Integer. One of the following - 1 = male 2 = female |
| ETHN | Subject ethnicity | Integer | - | Integer. Code as CRF |
| RACE | Subject race | Integer | - | Integer. Code as CRF |
| BMI | Body mass index | Decimal | kg/m^2 | body mass index calculated as weight divided by height squared |
| EVID | Event Identification data item | Integer | - | Flag indicating whether LABL contains dosing admin info or drug concentration data. |

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| | | | | Valid values are - 1 – each dosing record for subject 0 - for all other records |

### Assessments captured in the LABL variable

| Label | Description | Units |
|---|---|---|
| 0 | Dosing record for placebo | |
| 4 | Dosing records for 0.8 mg/Kg GSK2586881 | |
| 6 | Observed record (concentration or ratio) at time specified by TRLD; | |
| | excludes NA, IS and NR, includes non-quantifiable (NQ) data | |

# 10.9.5. Population PK/PD Dataset File Structure : Oxygen Saturation/PASP

The PME compliant file structure is a space-delimited file with each row containing the following columns of information. Data from all treatments will be included.

Decision as to whether this will be required will be made following the planned interim analysis (for study Part 2 at approximately N=3 or approximately N=6).

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| С | Data Identifier | Integer | - | 0 |
| STUD | Protocol Number | Integer | - | 204987 |
| DRUG | Name of Drug | Integer | - | Maximum 10 characters (numeric or text). 2586881 |
| SUBJ | Subject identifier in study | Integer | - | Maximum 10 characters (numeric or text). Different identifier for each subject |
| CENT | Study centre identifier | Integer | - | |
| LABL | Indicator field describing the type of assessment in that record | Integer | See<br>footnotes | See footnotes |
| AMT | Dose of<br>GSK2586881 | Decimal | Mg | Amount of drug given = Total GSK2586881 dose (mg/kg) * WT. AMT=0 when LABL=0 For dosing events: total dose of GSK2586881 taken For concentration events: 0 |
| INF | Infusion Time | Decimal | h | Time during which total dose infused. (Time at end of infusion – Time of start infusion) |
| RATE | Rate of Infusion | Decimal | Mg/h | Rate of infusion (AMT/INF) |

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| DGRP | Treatment Identifier | Decimal | - | DGRP=0 for placebo treatment<br>treatment<br>DGRP=0.8 for 0.8 mg/kg treatment<br>Dose of GSK2586881 (for all events) |
| PART | Study Part | Integer | - | 1=Part 1 or 2=Part 2 |
| PERIOD | Study Period | Integer | - | 1=Period 1 or 2=Period 2 |
| DAY | Study day | Integer | - | Maximum 10 characters (numeric or text) N= Day N, Actual Study Day |
| СТІМ | Clock time of Dose or measurement | HH:MM:SS | - | |
| DATE | Date of record | DD/MM/YYY | | |
| TRFD | Actual time relative to FIRST dose | Decimal | Hours | When LABL=1 or 4, TIME =0 Hours since start of FIRST infusion (on Day 1). For pre-dose sample, TRFD is relative to FIRST dose |
| TRLD | Actual time relative to LAST dose | Decimal | Hours | When LABL=0 or 4, TIME=0 Hours since start of LAST dose/infusion. For pre-dose sample, TRLD is relative to previous dose For single dose studies TRLD = TRFD |
| TFLAG | Time Flag | Integer | - | At T0 and LABL=6, TFLAG=0 At T1 and LABL=6, TFLAG=1 At T2 and LABL=6, TFLAG=2 At T3 and LABL=6, TFLAG=3 At T4 and LABL=6, TFLAG=4 Otherwise if LABL=6, TFLAG=5 If LABL="0" or "4", TFLAG=6 |
| BLPASP | PASP | Decimal | mmHg | Baseline Value |
| PASP | PASP | Decimal | mmHg | When LABL=6, PASP at time specified by TRLD. When LABL=1, or 4, PASP=0 |
| BLOS | Oxygen Saturation | Decimal | % | Baseline Value |
| OS | Oxygen Saturation | Decimal | % | When LABL=6, Oxygen Saturation at time specified by TRLD. When LABL=1 or 4, Oxygen Saturation=0 |
| EVID | Event Identification data item | Integer | - | Flag indicating whether LABL contains dosing admin info or drug concentration data. Valid values are - 1 – each dosing record for subject 0 - for all other records |

# Assessments captured in the LABL variable

| Label | Description | Units |
|---|---|---|
| 0 | Dosing record for placebo | |
| 4 | Dosing records for 0.8 mg/Kg GSK2586881 | |
| 6 | Observed record (concentration or ratio) at time specified by TRLD; | |
| | excludes NA, IS and NR | |

# 10.10. Appendix 10: Abbreviations & Trade Marks

# 10.10.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ACE2 | Angiotensin converting enzyme type 2 |
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| ALT | Alanine aminotransferase (SGPT) |
| Ang II | Angiotensin II |
| AST | Aspartate aminotransferase (SGOT) |
| AUC(0-2.5h) | Area under the concentration-time curve over the study period |
| AUC(0.5-2.0h) | Area under the concentration-time curve over the hypoxia challenge |
| A&R | Analysis and Reporting |
| BUN | Blood urea nitrogen |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CL | Clearance |
| Cmax | Maximum observed plasma concentration |
| CO2 | Carbon Dioxide |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> /CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DOB | Date of Birth |
| DP | Decimal Places |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Record Form |
| GSK | GlaxoSmithKline |
| GUI | Guidance |
| HPV | Hypoxic Pulmonary Vasoconstriction |
| IA | Interim Analysis |
| ICH | International Conference on Harmonisation |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| mITT | Modified Intent-To-Treat |
| IV | Intravenous |
| LOC | Last Observation Carries Forward |
| MMRM | Mixed Model Repeated Measures |
| O2 | Oxygen |
| PASP | Pulmonary Artery Systolic Pressure |

| Abbreviation | Description |
|--------------|---------------------------------------------------|
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PVR | Pulmonary Vascular Resistance |
| QC | Quality Control |
| QTcF | Fridericia's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| RAS | Renin-Angiotensin System |
| SAC | Statistical Analysis Complete |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| Tmax | Time to maximum observed concentration |
| T1/2 | Apparent terminal phase half-life |
| V | Volume of Distribution |
| VO2 | Oxygen Consumption |

# 10.10.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| HARP |
| RANDALL NG |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| R (Statistical programming |
| package/language) |
| SAS |
| WinNonLin |

# 10.11. Appendix 11: List of Data Displays

### 10.11.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------------------|------------|------------|
| Study Population | 1.1 to 1.n | 1.1 to 1.n |
| Efficacy | 2.1 to 2.n | 2.1 to 2.n |
| Safety | 3.1 to 3.n | 3.1 to 3.n |
| Pharmacokinetic | 4.1 to 4.n | 4.1 to 4.n |
| Pharmacodynamic and / or Biomarker | 5.1 to 5.n | 5.1 to 5.n |
| Pharmacokinetic / Pharmacodynamic | 6.1 to 6.n | 6.1 to 6.n |
| Section | List | ings |
| ICH Listings | 1 t | 0 X |
| Other Listings | y t | 0 Z |

### 10.11.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix 12: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------------------------|---------|---------|----------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Pharmacodynamic and / or Biomarker | PD_Fn | PD_Tn | PD_Ln |
| Pharmacokinetic / Pharmacodynamic | PKPD_Fn | PKPD_Tn | PK/PD_Ln |

### NOTES:

• Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

### 10.11.3. Deliverable [Priority]

| Delivery | Description |
|---|---|
| IA[1] Interim Analysis (Planned to be completed by GSK) – Study Part 1 | |
| IA[2], IA[3] | Interim Analyses (Planned to be completed by GSK) – Study Part 2 |
| SAC* | Final Statistical Analysis Complete (Planned to be completed by FSP) |

<sup>\*</sup>Please note that where IA and SAC are noted together next to an output, GSK internal stats and programming team will take responsibility for this output, unless otherwise stated.

# 10.11.4. Study Population Tables

| Study | Population Tabl | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Subjec | t Disposition | | | | |
| 1.1. | mITT | ES1A | Summary of Subject Disposition for the Subject Conclusion Record | | SAC |
| 1.2. | All Subjects<br>Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | | SAC |
| Protoc | ol Deviation | | | | |
| 1.3. | mITT | DV1 | Summary of Important Protocol Deviations | | SAC |
| Popula | tions Analysed | | | | |
| 1.4. | All Subjects<br>Screened | SP1A | Summary of Study Populations | Include All Screened, mITT, mITT1, mITT2, PK1 and PK2 populations. Footnote that percentages based on those in the mITT population, so mITT1, mITT2, PK1 and PK2 pops will have a percentage. | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 1.5. | mITT1 | DM3 | Summary of Demographic Characteristics (Part 1) | Age groupings <18, 18-40 and >40 to be used. Due to study entry criteria, only 18-40 will be displayed. Only total column needs to be included for a crossover study. | SAC |
| 1.6. | mITT2 | DM3 | Summary of Demographic Characteristics (Part 2) | As above (Part 2 population) | SAC |
| 1.7. | mITT1 | DM5 | Summary of Race and Racial Combinations (Part 1) | Only total column needs to be included for a crossover study. | SAC |

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 1.8. | mITT2 | DM5 | Summary of Race and Racial Combinations (Part 2) | As above (Part 2 population) | SAC |
| Medica | Medical Conditions | | | | |
| 1.9. | 1.9. mITT MH1 Summary of Past Medical Conditions Total column only. To be kept as overall mITT. SAC | | | | SAC |
| 1.10. | mITT | MH1 | Summary of Current Medical Conditions | Total column only. To be kept as overall mITT. | SAC |

# 10.11.5. Safety Tables

| Safety : | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PASP | | | | | |
| 3.1. | mITT1 | PFT1 | Summary of PASP (Part 1) | IDSL example PFT1 can be followed ('Day' won't be needed). If a log-transformation is required for analysis please include log-transformed summary as a second page using PFT2 example. | IA[1], SAC<br>(GSK) |
| 3.2. | mITT2 | PFT1 | Summary of PASP (Part 2) | As above (Part 2 population) | SAC (GSK) |
| 3.3. | mITT1 | PFT3 | Summary of PASP Change from Baseline (Part 1) | IDSL example PFT3 can be followed ('Day' won't be needed). If a log-transformation is required for analysis please include log-transformed summary as a second page using PFT2 example. | IA[1], SAC<br>(GSK) |

| Safety : | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.4. | mITT2 | PFT3 | Summary of PASP Change from Baseline (Part 2) | As above (Part 2 population) | SAC (GSK) |
| 3.5. | mITT1 | SAFE_T1<br>(non-standard) | Summary of Repeated Measures Bayesian<br>Statistical Analysis of Change from Baseline in<br>PASP (Part 1) | As per non-standard example SAFE_T1 but parameter column could be removed. Note that adjusted treatment differences and posterior probabilities (<0, <-2.5, <-5) are included on page 2 of mock example. Please note details regarding treatment differences in Section 7.2 and update output accordingly if a log-transformation is required (SAFE_T2 applies in this case with addition of posterior probabilities to be added). | IA[1], SAC<br>(GSK) |
| 3.6. | mITT2 | SAFE_T1<br>(non-standard) | Summary of Repeated Measures Bayesian<br>Statistical Analysis of Change from Baseline in<br>PASP (Part 2) | As above (Part 2 population) | SAC (GSK) |
| Oxygen | Saturation | | | | |
| 3.7. | mITT1 | PFT1 | Summary of Oxygen Saturation (Part 1) | IDSL example PFT1 can be followed ('Day' won't be needed). If a log-transformation is required for analysis please include log-transformed summary as a second page using PFT2 example. | IA[1], SAC<br>(GSK) |
| 3.8. | mITT2 | PFT1 | Summary of Oxygen Saturation (Part 2) | As above (Part 2 population) | SAC<br>(GSK) |
| 3.9. | mITT1 | PFT3 | Summary of Oxygen Saturation Change from Baseline (Part 1) | IDSL example PFT1 can be followed ('Day' won't be needed). If a log-transformation is required for analysis please include log-transformed summary as a second page using PFT2 example. | IA[1], SAC<br>(GSK) |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.10. | mITT2 | PFT3 | Summary of Oxygen Saturation Change from Baseline (Part 2) | As above (Part 2 population) | SAC<br>(GSK) |
| 3.11. | mITT1 | SAFE_T1<br>(non-standard) | Summary of Repeated Measures Bayesian<br>Statistical Analysis of Change from Baseline in<br>Oxygen Saturation (Part 1) | As per SAFE_T1 but parameter column could be removed. Note that adjusted treatment differences are included on page 2 of mock example. For OS expecting that we'll need to update the Posterior Probability labels, to <0%, <-3%, <-5%, where 5% is the clinical concern level for a treatment difference where GSK reduces OS to a greater extent. Please see Section 8.1.2 with regards to changes required should a log transformation be needed (SAFE_T2 applies in this case with addition of posterior probabilities to be added). | IA[1], SAC<br>(GSK) |
| 3.12. | mITT2 | SAFE_T1<br>(non-standard) | Summary of Repeated Measures Bayesian<br>Statistical Analysis of Change from Baseline in<br>Oxygen Saturation (Part 2) | As above (Part 2 population) | SAC (GSK) |
| Pulmor | nary Vascular R | Resistance (PVR) | | | |
| 3.13. | mITT2 | PFT1 | Summary of Pulmonary Vascular Resistance (PVR) (Part 2) | See comments for PASP | SAC (GSK) |
| 3.14. | mITT2 | PFT3 | Summary of Pulmonary Vascular Resistance<br>Change from Baseline (PVR) (Part 2) | See comments for PASP | SAC (GSK) |
| 3.15. | mITT2 | SAFE_T1<br>(non-standard) | Summary of Repeated Measures Bayesian<br>Statistical Analysis of Change from Baseline in<br>Pulmonary Vascular Resistance (PVR) (Part 2) | See comments for PASP. Note that adjusted treatment differences and posterior probabilities would initially be (<0, <0.1, <0.3) | SAC (GSK) |

| Safety | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | Adverse Events (AEs) | | | | |
| 3.16. | mITT1 | AE1CP (same as CP_AE1x) | Summary of All Adverse Events by System Organ<br>Class and Preferred Term (Part 1) | Summarise by treatment group. Any pretreatment AEs to be included in the listing only. Will only be created for interim if sufficient number of AEs are observed. | IA[1] (GSK),<br>SAC (FSP) |
| 3.17. | mITT2 | AE1CP (same as CP_AE1x) | Summary of All Adverse Events by System Organ Class and Preferred Term (Part 2) | As above (Part 2 population) | SAC (FSP) |
| 3.18. | mITT1 | AE1CP (same as CP_AE1x) | Summary All Drug-Related Adverse Events by<br>System Organ Class and Preferred Term (Part 1) | Summarise by treatment group. | SAC |
| 3.19. | mITT2 | AE1CP (same as CP_AE1x) | Summary All Drug-Related Adverse Events by<br>System Organ Class and Preferred Term (Part 2) | As above (Part 2 population) | SAC |
| 3.20. | mlTT1 | AE1CP (same as CP_AE1x) | Summary of All Serious Adverse Events by System Organ Class and Preferred Term (Part 1) | Production of this will be dependent on the number of SAEs, listing may suffice (based on clin pharm IDSL standards advice, this is a conditional summary). Summarise by treatment group. Any pre-treatment SAEs to be included only in listing. | SAC |
| 3.21. | mITT2 | AE1CP (same as CP_AE1x) | Summary of All Serious Adverse Events by System Organ Class and Preferred Term (Part 2) | As above (Part 2 population) | SAC |
| ECG | | | | | |
| 3.22. | mITT1 | EG1 | Summary of ECG Findings (Part 1) | | SAC |
| 3.23. | mITT2 | EG1 | Summary of ECG Findings (Part 2) | | SAC |
| 3.24. | mITT1 | EG2 | Summary of ECG Values (Part 1) | | SAC |
| 3.25. | mITT2 | EG2 | Summary of ECG Values (Part 2) | | SAC |
| 3.26. | mITT1 | CP_EG11 | Frequency of ECG Values by Pre-Specified PCI Categories (Part 1) | Categories as per PCI details in Section 10.6.2. | SAC |

| Safety : | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.27. | mITT2 | CP_EG11 | Frequency of ECG Values by Pre-Specified PCI Categories (Part 2) | As above (Part 2 population) | SAC |
| 3.28. | mITT1 | EG2 | Summary of Change from Baseline in ECG Values (Part 1) | | SAC |
| 3.29. | mITT2 | EG2 | Summary of Change from Baseline in ECG Values (Part 2) | | SAC |
| 3.30. | mITT1 | CP_EG12 | Frequency of Change from Baseline ECG Values by Pre-Specified PCI Categories (Part 1) | Categories as per PCI details in Section 10.6.2. | SAC |
| 3.31. | mITT2 | CP_EG12 | Frequency of Change from Baseline ECG Values by Pre-Specified PCI Categories (Part 2) | As above (Part 2 population) | SAC |
| Vital Si | gns | | | | |
| 3.32. | mITT1 | VS1 | Summary of Vital Signs (Part 1) | | SAC |
| 3.33. | mITT2 | VS1 | Summary of Vital Signs (Part 2) | | SAC |
| 3.34. | mITT1 | VS1 | Summary of Change from Baseline in Vital Signs (Part 1) | | SAC |
| 3.35. | mITT2 | VS1 | Summary of Change from Baseline in Vital Signs (Part 2) | | SAC |
| Immun | mmunogenicity | | | | |
| 3.36. | mITT | IMM1 | Summary of Positive Immunogenicity Results | Can be kept as mITT overall | SAC |

# 10.11.6. Safety Figures

| Safety : | Safety : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PASP | PASP CONTRACTOR CONTRA | | | | |
| 3.1. | mITT1 | (non-standard) | Summary of PASP (Absolute) (Part 1) | x-axis will be timepoints T0 to T4, see other mock examples, y-axis will be mean PASP including 95% CI, by treatment groups (add to legend). If data is log-transformed for the analysis then this graphic will need to show geometric means and 95% CIs. | IA1, SAC (GSK) |
| 3.2. | mITT2 | (non-standard) | Summary of PASP (Absolute) (Part 2) | As above (Part 2 population) | SAC (GSK) |
| 3.3. | mlTT1 | SAFE_F1<br>(non-standard) | Adjusted Median Responses and 95% Credible Interval vs Time Profiles of Change from Baseline in PASP (Part 1) | If possible please also add a horizontal line within the graph to indicate the 'hypoxia' in chamber period (approx 30 mins post dose to 120 mins post-dose). Add major tick marks for labels indicated in example graphic. Major tick marks to be PTM labels (or shortened version of). If data is log-transformed for analysis then this graphic will be presenting median ratios. | IA[1], SAC<br>(GSK) |
| 3.4. | mITT2 | SAFE_F1 (non-standard) | Adjusted Median Responses and 95% Credible Interval vs Time Profiles of Change from Baseline in PASP (Part 2) | As above (Part 2 population) | SAC (GSK) |

| Safety | : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.5. | mlTT1 | SAFE_F2<br>(non-standard) | Individual Subject Profiles of PASP (Part 1) | Adjust as space permits, with fewer subjects per page if needed. X-axis and footnote for illustration, can be amended/improved. Vertical reference lines represent start and stop of hypoxia/chamber period. | IA[1], SAC<br>(GSK) |
| 3.6. | mITT2 | SAFE_F2<br>(non-standard) | Individual Subject Profiles of PASP (Part 2) | As above (Part 2 population) | IA[2], IA[3],<br>SAC (GSK) |
| Oxyger | n Saturation | | | | |
| 3.7. | mlTT1 | (non-standard) | Summary of Oxygen Saturation (Absolute) (Part 1) | x-axis will be timepoints T0 to T4, see other mock examples, y-axis will be mean Oxygen Saturation including 95% CI, by treatment groups (add to legend) If data is log-transformed for the analysis then this graphic will need to show geometric means and 95% CIs. | IA[1], SAC<br>(GSK) |
| 3.8. | mITT2 | (non-standard) | Summary of Oxygen Saturation (Absolute) (Part 2) | As above (Part 2 population) | SAC (GSK) |
| 3.9. | mITT1 | SAFE_F1<br>(non-standard) | Adjusted Median Responses and 95% Credible Interval vs Time Profiles of Change from Baseline in Oxygen Saturation (Part 1) | As above for PASP figure | IA[1], SAC<br>(GSK) |
| 3.10. | mITT2 | SAFE_F1 (non-standard) | Adjusted Median Responses and 95% Credible Interval vs Time Profiles of Change from Baseline in Oxygen Saturation (Part 2) | As above (Part 2 population) | SAC (GSK) |
| 3.11. | mITT1 | SAFE_F2<br>(non-standard) | Individual Subject Profiles of Oxygen Saturation (Part 1) | As above for PASP figure | IA[1], SAC<br>(GSK) |

| Safety : | : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.12. | mITT2 | SAFE_F2<br>(non-standard) | Individual Subject Profiles of Oxygen Saturation (Part 2) | As above (Part 2 population) | IA[2], IA[3],<br>SAC (GSK) |
| 3.13. | mlTT2 | PD_F1<br>(non-standard) | Scatter Plot of Oxygen Saturation vs PASP (Part 2) | mITT2 population only Scatter plot: PASP on y axis, treatment groups side by side, timepoint (T0 to T4) split into panels. | SAC |
| Pulmor | nary Vascular R | Resistance (PVR) | | | |
| 3.14. | mITT2 | (non-standard) | Summary of Pulmonary Vascular Resistance (Absolute) (Part 2) | x-axis will be timepoints T0 to T4, see other mock examples, y-axis will be mean PVR including 95% CI, by treatment groups (add to legend) If data is log-transformed for the analysis then this graphic will need to show geometric means and 95% CIs. | SAC (GSK) |
| 3.15. | mITT2 | SAFE_F1 (non-standard) | Adjusted Median Responses and 95% Credible Interval vs Time Profiles of Change from Baseline in Pulmonary Vascular Resistance (Part 2) | See PASP comments | SAC (GSK) |
| 3.16. | mITT2 | SAFE_F2<br>(non-standard) | Individual Subject Profiles of Pulmonary Vascular Resistance (PVR) (Part 2) | See PASP comments | SAC (GSK) |
# 10.11.7. Pharmacokinetic Tables

| Pharma | Pharmacokinetic : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Con | centration Data | a | | | |
| 4.1. | PK1 | PKCT1 (PK01) | Summary of GSK2586881 Pharmacokinetic Concentration-Time Data (ng/mL) (Part 1) | | SAC |
| 4.2. | PK2 | PKCT1 (PK01) | Summary of GSK2586881 Pharmacokinetic Concentration-Time Data (ng/mL) (Part 2) | | SAC |
| PK Para | ameter Data | | | | |
| 4.3. | PK1 | PKPT1 (PK03) | Summary Statistics of Derived Plasma GSK2586881 Pharmacokinetic Parameters (Part 1) | See Section 8.2.3.1 for list of parameters to be expected | SAC |
| 4.4. | PK2 | PKPT1 (PK03) | Summary Statistics of Derived Plasma GSK2586881<br>Pharmacokinetic Parameters (Part 2) | As above (Part 2 population) | SAC |
| 4.5. | PK1 | PKPT3 (PK05) | Summary Statistics of Log-Transformed Derived Plasma GSK2586881 Pharmacokinetic Parameters (Part 1) | See Section 8.2.3.1 for list of parameters to be expected and Section 10.3.3 for details of those NOT to be log transformed | SAC |
| 4.6. | PK2 | PKPT3 (PK05) | Summary Statistics of Log-Transformed Derived Plasma GSK2586881 Pharmacokinetic Parameters (Part 2) | As above (Part 2 population) | SAC |

# 10.11.8. Pharmacokinetic Figures

| Pharma | Pharmacokinetic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Cor | centration Dat | a | | | |
| 4.1. | PK1 | PKCF1X<br>(PK16b) | Individual GSK2586881 Plasma Concentration–Time Plots (Linear and Semi-log) (Part 1) | By Subject plots | SAC |
| 4.2. | PK2 | PKCF1X<br>(PK16b) | Individual GSK2586881 Plasma Concentration–Time Plots (Linear and Semi-log) (Part 2) | By Subject plots – Part 2 | SAC |
| 4.3. | PK1 | PKCF6 (PK24) | Individual GSK2586881 Plasma Concentration–Time Plot (Linear and Semi-log) (Part 1) | All individual subject profiles on the same graphic. | SAC |
| 4.4. | PK2 | PKCF6 (PK24) | Individual GSK2586881 Plasma Concentration–Time Plot (Linear and Semi-log) (Part 2) | As above (Part 2 population) | SAC |
| 4.5. | PK1 | PKCF2 (PK17) | Mean Plasma GSK2586881 Concentration-Time Plot (Linear and Semi-Log) (Part 1) | | SAC |
| 4.6. | PK2 | PKCF2 (PK17) | Mean Plasma GSK2586881 Concentration-Time Plot (Linear and Semi-Log) (Part 2) | | SAC |
| 4.7. | PK1 | PKCF3 (PK18) | Median Plasma GSK2586881 Concentration-Time Plot (Linear and Semi-Log) (Part 1) | | SAC |
| 4.8. | PK2 | PKCF3 (PK18) | Median Plasma GSK2586881 Concentration-Time Plot (Linear and Semi-Log) (Part 2) | | SAC |

# 10.11.9. Pharmacodynamic and Biomarker Tables

| Pharma | Pharmacodynamic and Biomarker : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| RAS Pe | ptides – Key | | | | |
| 5.1. | mlTT1 | PD_T1 (or<br>modify PFT1 &<br>PFT2 | Summary of Key RAS Peptides (Absolute Data) (Part 1) | Log-transformed summary to be included as a second page for each parameter if data is log-transformed for analysis. Ang II, Ang(1-5), Ang(1-7) | SAC |
| 5.2. | mITT2 | PD_T1 (or<br>modify PFT1 &<br>PFT2 | Summary of Key RAS Peptides (Absolute Data) (Part 2) | As above (Part 2 population) | SAC |
| 5.3. | mITT2 | SAFE_T2<br>(non-standard) | Summary of Repeated Measures Bayesian<br>Statistical Analysis of Change from Baseline in<br>Key RAS Peptides (Part 2) | mITT2 only Log transformation likely to be required so output as per SAFE_T2. RAS Peptides are collected at timepoints other than T1 to T4 so these will need to be included. Note that adjusted treatment differences are included on page 2 of mock example. Posterior probabilities see Section 8.3.2. Ang II, Ang(1-5), Ang(1-7) If there is insufficient data to run a statistical analysis from data in Part 2, an analysis of Part 1 may be performed in place – to be discussed at DBF | SAC |
| Disease | Disease Biomarkers | | | | |
| 5.4. | mITT1 | PD_T1 (or<br>modify PFT1 &<br>PFT2 | Summary of Surfactant Protein D (Absolute Data) (Part 1) | Log-transformed summary to be included as a second page if data is log-transformed for analysis. Surfactant Protein D | SAC |

| Pharma | Pharmacodynamic and Biomarker : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.5. | mITT2 | PD_T1 (or<br>modify PFT1 &<br>PFT2 | Summary of Surfactant Protein D (Absolute Data) (Part 2) | As above (Part 2 population) | SAC |
| 5.6. | mlTT2 | SAFE_T2<br>(non-standard) | Summary of Repeated Measures Bayesian<br>Statistical Analysis of Change from Baseline in<br>Surfactant Protein D (Part 2) | mITT2 only Log transformation likely to be required so output as per SAFE_T2, otherwise SAFE_T1. SPD is collected at timepoints other than T1 to T4 so these will need to be included. Note that adjusted treatment differences are included on page 2 of mock example. Posterior probabilities see Section 8.3.2. If there is insufficient data to run a statistical analysis from data in Part 2, an analysis of Part 1 may be performed in place – to be discussed at DBF | SAC |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] | |
|---|---|---|---|---|---|---|
| Ventila | tory Parameter | S | | | | |
| | | III I PEII I | | Ventilatory parameters are collected at the same timepoints as PASP, with the exception of the post exercise timepoint where ventilatory parameters are not collected. Order parameters as follows: | | |
| 5.7. | mITT1 | | Summary of Ventilatory Parameters (Absolum Data) (Part 1) | Summary of Ventilatory Parameters (Absolute Data) (Part 1) | Oxygen consumption (VO2), Carbon dioxide production (CO2), Total Tidal Volume, | SAC |
| | | | | Inspiratory Tidal Volume, Expiratory Tidal Volume, Total Respiratory Time, Inspiratory Time, Expiratory Time, Duty Cycle, Mean Respiratory Flow,Respiratory rate | | |
| 5.8. | mITT2 | PFT1 | Summary of Ventilatory Parameters (Absolute Data) (Part 2) | As above (Part 2 population) | SAC | |

| Pharma | Pharmacodynamic and Biomarker : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Outputs | s to be confirm | ed post DBF | | | |
| 5.9. | mITT1 | SAFE_T2<br>(non-standard) | Summary of Repeated Measures Bayesian<br>Statistical Analysis of Change from Baseline in<br>Key RAS Peptides (Part 1) | mITT1 only Log transformation likely to be required so output as per SAFE_T2. RAS Peptides are collected at timepoints other than T1 to T4 so these will need to be included. Note that adjusted treatment differences are included on page 2 of mock example. Posterior probabilities see Section 8.3.2. Ang II, Ang(1-5), Ang(1-7) | Post SAC (to be confirmed post DBF) |
| 5.10. | mITT1 | SAFE_T2<br>(non-standard) | Summary of Repeated Measures Bayesian<br>Statistical Analysis of Change from Baseline in<br>Surfactant Protein D (Part 1) | mITT1 only Log transformation likely to be required so output as per SAFE_T2, otherwise SAFE_T1. SPD is collected at timepoints other than T1 to T4 so these will need to be included. Note that adjusted treatment differences are included on page 2 of mock example. Posterior probabilities see Section 8.3.2. | Post SAC (to be confirmed post DBF) |

# 10.11.10. Pharmacodynamic and Biomarker Figures

| Pharma | Pharmacodynamic and Biomarker : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| RAS Pe | ptides – Key | | | | |
| 5.1. | mITT1 | (non-standard) | Summary of Key RAS Peptides<br>(Absolute) (Part 1) | x-axis will be timepoints T0 to T4 (plus additional timepoints - see other mock examples), y-axis will be mean RAS including 95% CI, by treatment groups (add to legend). One page per endpoint (3 x RAS endpoints) A log-transformation is likely to be required for analysis so please present geometric means and 95% CIs on a second page. | SAC |
| 5.2. | mITT2 | (non-standard) | Summary of Key RAS Peptides (Absolute) (Part 2) | As above (Part 2 population) | SAC |
| 5.3. | mITT2 | SAFE_F1<br>(non-standard) | Adjusted Median Responses and 95%<br>Credible Interval vs Time Profiles of<br>Change from Baseline in Key RAS<br>Peptides (Part 2) | mITT2 only See example mock SAFE_F1 but page by endpoint (3 RAS endpoints). If log-transformed then median ratios will be plotted. If possible please also add a horizontal line within the graphic to indicate the 'hypoxia' in chamber period (approx 30 mins post dose to 120 mins post-dose). Add major tick marks for labels indicated in example graphic. Major tick marks to be PTM labels (or shortened version of). Note more timepoints for biomarkers other than T1 to T4. If there is insufficient data to run a statistical analysis from data in Part 2, an analysis of Part 1 may be performed in place – to be discussed at DBF | SAC |

| Pharma | acodynamic an | d Biomarker : Fig | ures | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.4. | mlTT1 | SAFE_F2<br>(non-standard) | Individual Subject Profiles of Key RAS<br>Peptides (Part 1) | All subjects on one page, one page per RAS endpoint. X-axis and footnote for illustration and can be amended/improved. Vertical reference lines represent start and stop of hypoxia/chamber period. Note more timepoints for biomarkers other than T1 to T4. Please note, mock shows raw data scales, but data is very likely to need to be log-transformed so please provide a second page per RAS endpoint with y-axis to accommodate log-transformed data. | IA[1], SAC |
| 5.5. | mlTT2 | SAFE_F2 (non-standard) | Individual Subject Profiles of Key RAS Peptides (Part 2) | As above (Part 2 population) | SAC |
| Disease | e Biomarkers | | | , | |
| 5.6. | mlTT1 | (non-standard) | Summary of Surfactant Protein D (Absolute) (Part 1) | x-axis will be timepoints T0 to T4 (plus additional timepoints - see other mock examples), y-axis will be mean SPD including 95% CI, by treatment groups (add to legend). A log-transformation is likely to be required for analysis so please present geometric means and 95% CIs on a second page. | SAC |
| 5.7. | mlTT2 | (non-standard) | Summary of Surfactant Protein D (Absolute) (Part 2) | As above (Part 2 population) | SAC |

| Pharmacodynamic and Biomarker : Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 5.8. | mlTT2 | SAFE_F1<br>(non-standard) | Adjusted Median Responses and 95%<br>Credible Interval vs Time Profiles of<br>Change from Baseline in SPD (Part 2) | mITT2 only See example mock SAFE_F1. If log-transformed then median ratios will be plotted. If possible please also add a horizontal line within the graphic to indicate the 'hypoxia' in chamber period (approx 30 mins post dose to 120 mins post-dose). Add major tick marks for labels indicated in example graphic. Major tick marks to be PTM labels (or shortened version of). Note more timepoints for biomarkers other than T1 to T4. If there is insufficient data to run a statistical analysis from data in Part 2, an analysis of Part 1 may be performed in place – to be discussed at DBF | SAC |
| 5.9. | mlTT1 | SAFE_F2<br>(non-standard) | Individual Subject Profiles of Surfactant<br>Protein D by Treatment Group and<br>Timepoint (Part 1) | Adjust as space permits, with fewer subjects per page if needed. X-axis and footnote for illustration and can be amended/improved. Vertical reference lines represent start and stop of hypoxia/chamber period. Note more timepoints for biomarkers other than T1 to T4. Please note, mock shows raw data scales, but data will most likely need to be log-transformed so in this case please provide a second page with y-axis to accommodate log-transformed data. | SAC |
| 5.10. | mITT2 | SAFE_F2<br>(non-standard) | Individual Subject Profiles of Surfactant Protein D by Treatment Group and Timepoint (Part 2) | As above (Part 2 population) | SAC |

| Pharmacodynamic and Biomarker : Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Key RA | Key RAS Peptides vs PASP & Oxygen Saturation | | | | |
| 5.11. | mITT | PD_F1<br>(non-standard) | Scatter Plot of RAS Peptides (Ang II,<br>Ang(1-7) and Ang(1-5)) vs PASP (Part<br>1 and 2 combined) | Scatter plot: PASP on y axis. Page by RAS endpoint, treatment groups side by side, timepoints T0 to T4 within panels (2 columns, 5 rows per page, 3 pages). Plot T0 to T4 timepoints (timepoints that match for the two endpoints of interest). Identify study part by different colour/symbol. As RAS data is log-transformed, please include a second page y-axis to accommodate log-transformed data. | SAC |
| 5.12. | mITT2 | PD_F1<br>(non-standard) | Scatter Plot of RAS Peptides (Ang II,<br>Ang(1-7) and Ang(1-5)) vs Oxygen<br>Saturation (Part 1 and 2 combined) | Scatter plot: Oxygen Saturation on y axis. Page by RAS endpoint, treatment groups side by side, timepoints T0 to T4 within panels (2 columns, 5 rows per page, 3 pages). Plot T0 to T4 timepoints (timepoints that match for the two endpoints of interest). Identify study part by different colour/symbol. | SAC |
| | | | | | As RAS data is log-transformed, please include a second page y-axis to accommodate log-transformed data. |
| Output | s to be confirm | ed post DBF | | | |
| 5.13. | mlTT1 | SAFE_F1<br>(non-standard) | Adjusted Median Responses and 95%<br>Credible Interval vs Time Profiles of<br>Change from Baseline in Key RAS<br>Peptides (Part 1) | mITT1 only See example mock SAFE_F1 but page by endpoint (3 RAS endpoints). If log-transformed then median ratios will be plotted. If possible please also add a horizontal line within the graphic to indicate the 'hypoxia' in chamber period (approx 30 mins post dose to 120 mins post-dose). Add major tick marks for labels indicated in example graphic. Major tick marks to be PTM labels (or shortened version of). Note more timepoints for biomarkers other than T1 to T4. | Post SAC (to be confirmed post DBF) |

| Pharma | Pharmacodynamic and Biomarker : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.14. | mITT1 | SAFE_F1<br>(non-standard) | Adjusted Median Responses and 95%<br>Credible Interval vs Time Profiles of<br>Change from Baseline in Surfactant<br>Protein D (Part 1) | mITT1 only If log-transformed then median ratios will be plotted. If possible please also add a horizontal line within the graphic to indicate the 'hypoxia' in chamber period (approx 30 mins post dose to 120 mins post-dose). Add major tick marks for labels indicated in example graphic. Major tick marks to be PTM labels (or shortened version of). Note more timepoints for biomarkers other than T1 to T4. | Post SAC (to be confirmed post DBF) |

# 10.11.11. Pharmacokinetic / Pharmacodynamic Figures

| Pharma | Pharmacokinetic / Pharmacodynamic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.1. | mITT2 | PK_F1 | Scatter Plot of Plasma GSK2586881 Concentration vs PASP (Part 2) | mITT2 only Timepoint split into panels (matching timepoints are T0 to T4) Placebo PASP data included at concentration of zero for comparison, see mock example. | SAC |
| 6.2. | mITT | PK_F2 | Scatter Plot of Plasma GSK2586881 Concentration vs RAS Peptides (Ang II, Ang(1-5) and Ang(1-7)) (Part 1 and 2 combined) | mITT (Part 1 and 2 identified by colour/symbol) One page per RAS endpoint. Placebo RAS data included at concentration of zero for comparison, see mock example. Please note, if RAS data is log-transformed then also include a second page per RAS endpoint displaying log-transformed RAS vs concentrations. | SAC |
| 6.3. | mITT2 | PK_F1 | Scatter Plot of AUC(0.5-2h) vs PASP (Part 2) | mITT2 only Timepoint T2 and T3 only, to be included as two separate panels Please include log-transformed AUC graphic on a second page. | SAC |

# 10.11.12. ICH Listings

| ICH : L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1. | All Screened<br>Subjects | ES7 | Listing of Reasons for Screen Failure | Include footnote: Study Part 1 (subject numbers P to PPD Study Part 2 (subject numbers PPD Study Part 2 ) | SAC |
| 2. | mITT | ES2 | Listing of Reasons for Study Withdrawal | Include footnote: Study Part 1 (subject numbers P to PPD Study Part 2 (subject numbers PPD | SAC |
| 3. | mITT | BL2 | Listing of Subjects for Whom the Treatment Blind was Broken | Include footnote: Study Part 1 (subject numbers P to PPD Study Part 2 (subject numbers 20+). | SAC |
| 4. | mITT | CP_TA2 | Listing of Randomised and Actual Treatments | Include footnote: Study Part 1 (subject numbers P to PPD Study Part 2 (subject numbers PPD Study PPD | SAC |
| Protoc | ol Deviations | | | | |
| 5. | mITT | DV2 | Listing of Important Protocol Deviations | Include footnote: Study Part 1 (subject numbers P to PPD Study Part 2 (subject numbers PPD Study Part 2 PPD P | SAC |
| 6. | mITT | IE4 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | Include footnote: Study Part 1 (subject numbers P to PPD Study Part 2 (subject numbers PPD Study Part 2 PPD P | SAC |
| Popula | tions Analysed | | | | |
| 7. | All Screened<br>Subjects | SP3a | Listing of Subjects Excluded from Any Population | Include footnote: Study Part 1 (subject numbers P to PPD Study Part 2 (subject numbers PPD Study Part 2 PPD P | SAC |

| ICH : Li | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 8. | mITT | DM4 | Listing of Demographic Characteristics | Include footnote: Study Part 1 (subject numbers P to PPD Study Part 2 (subject numbers PPD Study PPD PPD Study PPD PP | SAC |
| 9. | mITT | DM10 | Listing of Race | Include footnote: Study Part 1 (subject numbers P to PPD Study Part 2 (subject numbers PPD Study P | SAC |
| Prior a | nd Concomitan | t Medications | | | |
| 10. | mITT | CP_CM4 | Listing of Concomitant Medications | For small studies / limited conmed data, a listing can be used in place of summary table, hence no summary table requested for this study. Include footnote: Study Part 1 (subject numbers to PPD Study Part 2 (subject numbers PPD) | SAC |
| Exposu | ire and Treatmo | ent Compliance | | | |
| 11. | mITT | EX4 | Listing of Exposure Data | Include footnote: Study Part 1 (subject numbers P to PPD Study Part 2 (subject numbers PPD Study PPD Stu | SAC |

| ICH : L | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | | | | |
| 12. | All Screened<br>Subjects | AE9CP | Listing of All Adverse Events for Non-randomised subjects | Only output AEs that occurred for non-randomised subjects only. These should be assigned as pre-treatment. If no AEs then list 'No data to report'. Any SAEs will be noted on this listing. Include footnote: Study Part 1 (subject numbers to PPD Study Part 2 (subject numbers PPD) | SAC |
| 13. | mITT | AE9CP | Listing of All Adverse Events | Will include AEs for mITT patients, including those that occurred pretreatment. Include footnote: Study Part 1 (subject numbers Pto PPD Study Part 2 (subject numbers PPD) | IA[1] (GSK),<br>SAC (FSP) |
| Serious | and Other Sig | nificant Adverse | Events | | |
| 14. | mITT | AE9CPA (same as CP_AE9a) | Listing of Serious Adverse Events | As above Include footnote: Study Part 1 (subject numbers P to PPD Study Part 2 (subject numbers PPD Study Part 2) | SAC |
| 15. | mITT | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | Include footnote: Study Part 1 (subject numbers Pto PPD Study Part 2 (subject numbers PPD | SAC |

| ICH : Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| All Lab | oratory | | | | |
| 16. | mITT | LB6 | Listing of All Laboratory Data for Subjects with Any Value of Potential Clinical Concern/Potential Clinical Importance | Group by chemistry and haematology Include footnote: Study Part 1 (subject numbers to PPD Study Part 2 (subject numbers PPD | SAC |
| 17. | mITT | LB6 | Listing of Laboratory Values of Potential Clinical Importance | Group by chemistry and haematology Include footnote: Study Part 1 (subject numbers to PPD Study Part 2 (subject numbers PPD) | SAC |
| ECG | | | | | |
| 18. | mITT | CP_EG4 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | Include footnote: Study Part 1 (subject numbers P to PPD Study Part 2 (subject numbers PPD) | SAC |
| 19. | mITT | CP_EG4 | Listing of ECG Values of Potential Clinical Importance | Include footnote: Study Part 1 (subject numbers P to PPD Study Part 2 (subject numbers PPD) | SAC |
| 20. | mITT | CP_EG6 | Listing of Abnormal ECG Findings | Include footnote: Study Part 1 (subject numbers P to PPD Study Part 2 (subject numbers PPD | SAC |

| ICH : Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Vital Sig | Vital Signs | | | | |
| 21. | mITT | CP_VS5 | Listing of All Vital Signs Data for Subjects with Any Value of Potential Clinical Importance | Include footnote: Study Part 1 (subject numbers P to PPD Study Part 2 (subject numbers PPD | SAC |
| 22. | mITT | CP_VS5 | Listing of All Vital Signs Data of Potential Clinical Importance | Include footnote: Study Part 1 (subject numbers P to PPD Study Part 2 (subject numbers PPD Study Part 2 PPD P | SAC |

# 10.11.13. Non-ICH Listings

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Safety | | | | | |
| 23. | mITT | PFT9 | Listing of PASP | Follow PFT9 IDSL format, replacing the last four FEV columns on the example with one PASP column. Include footnote: Study Part 1 (subject numbers Pto PPD Study Part 2 (subject numbers PPD) | IA[1], IA[2],<br>IA[3], SAC<br>(GSK) |
| 24. | mITT | PFT9 | Listing of Oxygen Saturation | As above Include footnote: Study Part 1 (subject numbers P to Study Part 2 (subject numbers PPD) | IA[1], IA[2],<br>IA[3], SAC<br>(GSK) |
| 25. | mITT | PFT9 | Listing of Ventilatory Parameters | Similar format to above except include a parameter column to include all ventilator parameter results at each timepoint. Non-standard modification may be required. Include footnote: Study Part 1 (subject numbers Pto PPD Study Part 2 (subject numbers PPD) | SAC |
| Biomar | kers | | | | |
| 26. | mITT | PD_L1<br>(non-standard) | Listing of RAS Peptides | See non-standard example PD_L1 Include footnote: Study Part 1 (subject numbers Pto PPD Study Part 2 (subject numbers PPD) | IA[1], SAC |
| 27. | mITT | PD_L1<br>(non-standard) | Listing of Surfactant Protein D | Non-standard example above can be followed Include footnote: Study Part 1 (subject numbers Pto PPD Study Part 2 (subject numbers PPD) | SAC |

| Non-ICI | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Immun | ogenicity | | | | |
| 28. | mITT | IMM2 | Listing of Immunogenicity Results | Note: Subjects should have data recorded at screening or period 1 pre-dose (not at both timepoints) Include footnote: Study Part 1 (subject numbers Pto PPD Study Part 2 (subject numbers PPD | SAC |
| PK | | | | | |
| 29. | PK | PKCL1X<br>(PK08) | Listing of GSK2586881 Plasma Pharmacokinetic Concentration–Time Data | Include footnote: Study Part 1 (subject numbers P to PPD Study Part 2 (subject numbers PPD | SAC |
| 30. | PK | PKPL1X<br>(PK14) | Listing of Derived GSK2586881 Plasma<br>Pharmacokinetic Parameters | See Section 8.2.3.1 for list of parameters. To include lambda_z and then additionally the first point, last point and number of points used in the determination of lambda_z for listings and R squared. Include footnote: Study Part 1 (subject numbers P to PPD Study Part 2 (subject numbers PPD) | SAC |
| 31. | mITT2 | PFT9 | Listing of Pulmonary Vascular Resistance | Follow PFT9 IDSL format, replacing the last four FEV columns on the example with one PVR column. Include footnote: Study Part 1 (subject numbers Pto PPD Study Part 2 (subject numbers PPD) | SAC (GSK) |

# 10.12. Appendix 12: Example Mock Shells for Data Displays

Data Display Specification will be made available on Request.

#### The GlaxoSmithKline group of companies

204987

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

Title : Reporting and Analysis Plan for the effects of GSK2586881 on the responses to acute hypoxia and exercise

Compound Number : GSK2586881

Effective Date : 02-MAY-2017

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 204987.
- This RAP is intended to describe the safety, pharmacodynamic and pharmacokinetic analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Interim Analysis and Statistical Analysis Complete (SAC) deliverables.

#### Author's Name and Functional Area:

| PPD | | 02 MAY 2017 |
|-------------------|-----------------------------|-------------|
| Principal Statist | ician (Clinical Statistics) | 02-MAY-2017 |
| PPD | | 02 MAN 2017 |
| Manager, Clinic | al Pharmacology (CPMS) | 02-MAY-2017 |

#### Approved by:

| PPD | 02-MAY-2017 |
|------------------------------------------------------------|--------------|
| Director, Statistics and Programming (Clinical Statistics) | 02-WA 1-2017 |

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

204987

#### **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | REPO | ORTING & ANALYSIS PLAN SYNOPSIS | 5 |
| 2. | SUMN<br>2.1.<br>2.2.<br>2.3.<br>2.4. | MARY OF KEY PROTOCOL INFORMATION Changes to the Protocol Defined Statistical Analysis Plan Study Objective(s) and Endpoint(s). Study Design Statistical Hypotheses. | 7<br>8 |
| 3. | PLANN<br>3.1.<br>3.2. | NED ANALYSESInterim AnalysesFinal Analyses | 9 |
| 4. | ANALY<br>4.1. | YSIS POPULATIONSProtocol Deviations | |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING /ENTIONS | 12 |
| 6. | STUD'<br>6.1. | Y POPULATION ANALYSES Overview of Planned Analyses | |
| 7. | PRIMA<br>7.1.<br>7.2. | ARY STATISTICAL ANALYSES Overview of Planned Analyses Planned Statistical Analyses | 14 |
| 8. | SECO<br>8.1. | NDARY ANALYSES | 16<br>16<br>17 |
| | | <ul> <li>8.2.1. Overview of Planned Pharmacokinetic Analyses</li> <li>8.2.2. Drug Concentration Measures</li> <li>8.2.3. Pharmacokinetic Parameters</li> <li>8.2.3.1. Deriving Pharmacokinetic Parameters</li> <li>8.2.4. Population Pharmacokinetic (PopPK) Analyses</li> </ul> | 18<br>19<br>19 |
| | 8.3. | Pharmacodynamic and Biomarker Analyses | 20 |
| | 8.4. | AnalysesPharmacokinetic / Pharmacodynamic Analyses | 21 |
| 9. | REFE | RENCES | 23 |
| 10. | APPEI<br>10.1. | NDICES | 25<br>25<br>26 |

| | | | 204987 |
|---|---|---|---|
| 10.2. | Appendix | c 2: Treatment States | 29 |
| | 10.2.1. | Treatment States for AE Data | 29 |
| | | 10.2.1.1. Treatment States for AE Dates | 29 |
| | 10.2.2. | Treatment States for Concomitant Medication Data | 30 |
| | | 10.2.2.1. Treatment States for Concomitant Medication Dates | 31 |
| 10.3. | Appendix | 3: Data Display Standards & Handling Conventions | |
| | 10.3.1. | | |
| | 10.3.2. | Baseline Definition & Derivations | |
| | | 10.3.2.1. Baseline Definitions | 32 |
| | | 10.3.2.2. Derivations and Handling of Missing Baseline | |
| | | Data | |
| | 10.3.3. | Reporting Process & Standards | 33 |
| 10.4. | Appendix | c 4: Derived and Transformed Data | |
| | 10.4.1. | General | |
| | 10.4.2. | Study Population | |
| | 10.4.3. | Safety | |
| | 10.4.4. | Pharmacodynamic and Biomarker | |
| 10.5. | | 5: Premature Withdrawals & Handling of Missing Data | |
| | 10.5.1. | Premature Withdrawals | |
| | 10.5.2. | Handling of Missing Data | |
| | | 10.5.2.1. Handling of Missing Dates | 39 |
| | | 10.5.2.2. Handling of Partial Dates | 39 |
| | | 10.5.2.3. Handling of Missing Data for Statistical Analysis | 40 |
| 10.6. | Appendix | c 6: Values of Potential Clinical Importance | |
| | 10.6.1. | Laboratory Values | |
| | 10.6.2. | ECG | |
| | 10.6.3. | Vital Signs | 42 |
| 10.7. | | c 7: Biomarker Details | 43 |
| 10.8. | Appendix<br>Analyses | k 8: Model Checking and Diagnostics for Statistical | 44 |
| 10.9. | | (9: Population PK and Pharmacokinetic / | |
| | | odynamic (Or Biomarker) Analyses | 45 |
| | 10.9.1. | | |
| | 10.9.2. | | |
| | 10.9.3. | Population PK/PD Dataset File Structure : ANG1-5 | 50 |
| | 10.9.4. | Population PK/PD Dataset File Structure : ANG1-7 | 52 |
| | 10.9.5. | Population PK/PD Dataset File Structure : Oxygen | |
| 10.10 | ۸ | Saturation/PASP | 55 |
| 10.10. | Appendix | x 10: Abbreviations & Trade Marks | 57 |
| | | Abbreviations | |
| 10 11 | 10.10.Z. | Trademarks | 50 |
| 10.11. | | Data Display Numbering | |
| | | Mock Example Shell Referencing | |
| | | Deliverable [Priority] | |
| | | Study Population Tables | |
| | | Safety Tables | |
| | | Safety Figures | |
| | 10.11.7 | Pharmacokinetic Tables | 67 |
| | | Pharmacokinetic Figures | |

| | 204987 |
|-----------------------------------------------------------|--------|
| 10.11.9. Pharmacodynamic and Biomarker Tables | 69 |
| 10.11.10.Pharmacodynamic and Biomarker Figures | |
| 10.11.11.Pharmacokinetic / Pharmacodynamic Figures | |
| 10.11.12.ICH Listings | 75 |
| 10.11.13.Non-ICH Listings | 78 |
| 10.12. Appendix 12: Example Mock Shells for Data Displays | |

204987

# 1. REPORTING & ANALYSIS PLAN SYNOPSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | <ul> <li>The purpose of this Reporting and Analysis Plan is to describe all planned<br/>analyses and outputs required for the Clinical Study Report (CSR) of study<br/>204987</li> </ul> |
| Protocol | <ul> <li>This RAP is based on the protocol (Dated 23/SEP/2016, GSK Document No.: 2016N283626_00) and protocol amendments 1 &amp; 2 (Dated:24/FEB/2017, GSK Document No.: 2016N283626_01 &amp; 07/MAR/2017, GSK Document No.: 2016N283626_02) of study GSK2586881/204987</li> </ul> |
| Study<br>Design | The study will be a single centre, randomised, placebo-controlled and double blind (sponsor open). Subjects will be randomised to receive a single IV dose of GSK2586881 or saline in a crossover design. Approximately 25 subjects will be enrolled to ensure that a minimum of 20 subjects complete all dosing and critical assessments (the target of 20 may be revised by the sample size reestimation) |
| Primary<br>Objective | To evaluate the effect of a single IV dose of GSK2586881 on the HPV response in healthy volunteers during exercise under hypoxic conditions |
| Primary<br>Endpoint | Change from baseline of Pulmonary Artery Systolic Pressure (PASP) measured via Echocardiography |
| Planned<br>Analyses | <ul> <li>An Interim Analysis is planned after approximately 10 patients have completed<br/>periods 1 and 2 of the study, to aid the team in decision making with regards to<br/>stopping the study for futility or a re-assessment of sample size</li> </ul> |
| | <ul> <li>All decisions regarding final analysis, as defined in this RAP document, will be<br/>made prior to Database Freeze.</li> </ul> |
| Analysis<br>Populations | All Subjects Screened Population will contain all subjects that complete at least one Visit 1 (Screening) procedure. |
| | The Modified Intent-to-Treat (mITT) Population will comprise all randomised subjects, excluding those who were randomised in error. |
| | The Pharmacokinetic (PK) Population will comprise all subjects in the mITT Population for whom a PK sample was obtained and analysed and on active treatment. |
| Hypothesis | No formal statistical hypotheses are being tested. A Bayesian statistical analysis framework with non-informative priors for model parameters (unless otherwise specified) will be used to obtain posterior distributions for effects of interest. These posterior distributions will be used to obtain a number of probability statements about the magnitude of treatment effects (e.g. probability of any treatment related reduction in PASP, or probability that the treatment related reduction in PASP ≥ 5 mmHg). A rule of thumb for "end of study success" is if the probability of any treatment related reduction in PASP (T3-T0) exceeds 0.95 (success is also conditional on the probability of (absolute) treatment related reductions in oxygen saturation exceeding 5% being small). |

204987

| Overview | Key Elements of the RAP |
|---|---|
| Primary<br>Analyses | The primary endpoint, change from baseline in PASP following exercise under hypoxic conditions (Ti-T0) will be analysed using a Bayesian repeated measures mixed effects regression model, to compare the effects of Placebo vs GSK2586881. |
| Secondary | Pharmacodynamic/Biomarker: |
| Analyses | RAS peptide responses: Ang II, Ang(1-7), Ang(1-5) will be analysed in a manner similar to the primary endpoint using Bayesian repeated measures mixed modelling to compare the effects of Placebo vs GSK2586881. |
| | Safety: |
| | Oxygen saturation will be analysed in a manner similar to the primary efficacy endpoint using Bayesian repeated measures mixed modelling to compare the effects of Placebo vs GSK2586881. Vital signs, 12-Lead ECG, AEs and Labs will be tabulated and/or listed by treatment group and timepoint as appropriate. |
| | Immunogenicity: |
| | Data will be tabulated and/or listed. |
| | Pharmacokinetic: |
| | Plasma concentrations of GSK2586881 and derived PK parameters will be summarised descriptively/graphically and listed. |
| Exploratory | Pharmacodynamic/Biomarker: |
| Analyses | The disease biomarker Surfactant Protein D will be analysed in a manner similar to the primary efficacy endpoint using Bayesian repeated measures mixed modelling to compare the effects of Placebo vs GSK2586881, if data permit. |
| | Ventilatory parameters (Oxygen consumption (VO2), Carbon dioxide production (CO2), Total Tidal Volume, Inspiratory Tidal Volume, Expiratory Tidal Volume, Total Respiratory Time, Inspiratory Time, Expiratory Time, Duty Cycle, Mean Respiratory Flow and Respiratory rate) will be summarised descriptively and listed. |
| | Pharmacogenetics |
| | Analysis of pharmacogenetic data will be carried out separately by the GSK Genetics team and a separate RAP will be produced. As this is an exploratory endpoint, the results will be available separately to the CSR (or to be included as an appendix). |

204987

#### 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no major changes or deviations to the originally planned statistical analysis specified in the protocol (Dated: 23/SEP/2016) and protocol amendments 1 and 2 (dated 24/FEB/2017 and 07/MAR/2017).

Some minor changes have been included. The variance/covariance structure to be used to account for repeated measurements has been updated to be unstructured (previously specified as compound symmetry). Statistical modelling described in this RAP will supersede any descriptions of modelling specifics provided in the protocol. In addition, the Intent-to-Treat Population has been renamed as Modified Intent-to-Treat to ensure this accurately reflects the description of the population and for suitability in any future publications.

#### 2.2. Study Objective(s) and Endpoint(s)

| Ob | jectives | En | dpoints |
|---|---|---|---|
| Pri | mary Objective | Pri | imary Endpoint |
| • | To evaluate the effect of a single IV dose of GSK2586881 on the HPV response in healthy volunteers during exercise under hypoxic conditions | • | Change from baseline of Pulmonary Artery Systolic Pressure (PASP) measured via Echocardiography |
| Se | condary Objectives | se | condary Endpoints |
| • | To evaluate the effect of a single IV dose GSK2586881 on RAS peptide responses To evaluate the safety of a single IV dose of CSK2586891 in healthy. | • | Effect of GSK2586881 on baseline levels and changes in response to hypoxia and exercise of RAS peptides (e.g. Ang II, Ang(1-7), Ang(1-5)) Vital signs (heart rate, systolic and diastolic blood |
| | IV dose of GSK2586881 in healthy volunteers | • | pressure) Oxygen saturation 12-lead ECGs Adverse Events (AEs) Immunogenicity Clinical laboratory assessments |
| • | To evaluate the pharmacokinetics of a single IV dose of GSK2586881 | • | Continuous pulse oximetry (assessed by the site) Plasma concentrations of GSK2586881 Derived pharmacokinetic parameters |
| Ex | ploratory Objectives | | ploratory Endpoints |
| • | To evaluate the effect of a single IV dose of GSK2586881 on ventilatory parameters in healthy volunteers during exercise in hypoxic conditions | Ch<br>• | ange from baseline of: Oxygen consumption (VO2) Carbon dioxide production (CO2) And other parameters as data permit |
| • | To evaluate the pharmacodynamic activity of a single IV dose of GSK2586881 in healthy volunteers during exercise in hypoxic conditions | • | Change from baseline in Surfactant Protein D and/or additional analytes to be determined |

204987

| Objectives | Endpoints |
|---|---|
| To evaluate Pharmacogenetics | Evaluate I/D polymorphisms in the Angiotensin<br>Converting Enzyme (ACE) gene and analyse the<br>impact on Ang II (and possibly other RAS peptides),<br>hypoxic pulmonary vasoconstriction and responses<br>to GSK2586881 administration |

#### 2.3. Study Design



204987

# 2.4. Statistical Hypotheses

There are no formal statistical hypotheses. This is an exploratory study and will be analysed, utilising a Bayesian framework.

# 3. PLANNED ANALYSES

# 3.1. Interim Analyses

An interim analysis is planned after approximately 10 subjects have completed the following critical assessments:

| Interim Analysis | Definition / Criteria / Purpose |
|---|---|
| PASP at T0 and<br>T3 for both stud<br>periods | from pre-dose PASP to hypoxic/exercised PASP [T3-T0]. To decide whether to continue the study or stop based on futility. To conduct an advisory sample-size re-estimation with the view to potentially reduce the number of subjects participating in the study below 20. Precision estimates will be updated based on the variability observed from the interim analyses to aid the team in decision making. PASP data will be summarised and listed. Statistical analysis will be completed as described in Section 7.2 including a graphic of treatment estimates over time. |
| Oxygen saturati<br>at T0 and T3 for<br>both study perior | change from pre-dose oxygen saturation to hypoxic/exercised oxygen |
| Adverse Events | |
| Angiotensin biomarker concentrations (Ang II, Ang(1-5 Ang(1-7)) | <ul> <li>For the first 5 subjects only to allow time for the samples to be analysed by the lab.</li> <li>Data will be listed only due to expected small sample size. Individual subject plots may be produced.</li> <li>If Angiotensin data (Ang II, Ang(1-5), Ang(1-7)) is not available at the time of the interim, analysis of the specified eCRF data will still go ahead as planned. A positive outcome in relation to PASP, Oxygen Saturation and AEs would lead to the study continuing without the need to review Angiotensin data.</li> <li>Should a negative outcome be observed with PASP or Oxygen Saturation, then confirmation of the decision to stop the study for futility would not occur until the Angiotension data from the initial transfer were available and reviewed.</li> </ul> |

204987

| Interim Analysis | Definition / Criteria / Purpose |
|---|---|
| | Any negative results with regards to AEs (as agreed by the study team), |
| | regardless of other endpoint results, would result in the study stopping. |

The interim analysis will use a data snapshot that has been cleaned to the best extent allowed by the timeframes (i.e. the interim data will not be fully cleaned or fully QC'd data and there will not be a locked database). The date of the source data cut should be indicated on each interim related output (this can be implemented in HARP via the *d\_datadate* macro input parameter in the *ts\_setup* macro call). Results will be restricted to selected members of the study team. Results or discussions will not be circulated to blinded staff involved in the conduct of the study at the sites.

The following table represents a guide to the outputs to be produced for the interim analysis. All outputs will be produced in HARP.

| Endpoint / Parameter/<br>Display Type | Absolute | | | | | | | | Change from Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | s Ana | lysis | Summary | | Individual | | Stats Analysis | | | Summary | | Individual | |
| | Τ | F | L | Τ | F | F | L | Τ | F | L | Т | F | F | L |
| PASP | | | | Υ | Υ | Υ | Υ | <b>Y</b> 3 | Υ | | Υ | | | |
| Oxygen Saturation | | | | Υ | Υ | Υ | Υ | $Y^3$ | Υ | | Υ | | | |
| All AEs | | | | Y1 | | | Y <sup>2</sup> | | | | | | | |
| RAS Peptides (AngII,<br>Ang(1-5), Ang(1-7)) | | | | | | Υ | Y | | | | | | | |

#### NOTES:

- Y = Yes display generated.
- 1. Produced if sufficient data
- 2. SAEs will be flagged within this listing
- 3. One table to include statistical analysis medians (95% Crl) and posterior probabilities. Also include within subject correlation as a footnote to support sample size re-estimation.

The sample size re-estimation will be performed once the primary analysis for the interim has been completed and assuming that no overwhelming data supporting the need to stop for futility is observed. Estimates of standard deviations and within subject correlation will be obtained from the PASP outputs produced during the interim and/or from SAS outputs from the statistical modelling. The sample size re-estimation will be performed by re-running programs (using R) used to obtain pre-study precision estimates. The sample size re-estimation program and associated excel outputs of precision estimates will be archived.

#### 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol (and subject to decisions made from the interim analyses).
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.

204987

- All criteria for unblinding the randomisation codes have been met (note that the study is being run as sponsor-unblinded, however, only a partial randomisation schedule will be made available to the GSK programming team for the interim analysis).
- 4. Randomisation codes have been distributed according to RandAll NG procedures.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Subjects<br>Screened | Comprising of all subjects who complete at least one Visit 1 (Screening) procedure. | <ul> <li>Subject disposition<br/>(including reasons for<br/>screening failures)</li> <li>Listing of any<br/>AEs/SAEs for non-<br/>randomised subjects</li> </ul> |
| Modified Intent-<br>To-Treat | Comprising of all randomised subjects, excluding those who were randomised in error. A subject who is recorded as a screen failure, run-in failure, or stabilisation failure, but is randomised and does not receive a dose of study treatment is considered to have been randomised in error. Any other subject who receives a randomisation number will be considered to have been randomised. | <ul><li>PD/Biomarkers</li><li>Safety</li></ul> |
| Pharmacokinetic | Subjects in the 'mITT' population for whom a pharmacokinetic sample was obtained and analysed and on active treatment. | • PK |

#### NOTES:

 Please refer to Appendix 11: List of Data Displays which details the population to be used for each display being generated.

#### 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, subject management or subject assessment) will be summarised and listed
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
  - o This dataset will be the basis for the summaries and listings of protocol deviations.
- A listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

204987

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 10.1 | Appendix 1: Time & Events |
| 10.2 | Appendix 2: Treatment States |
| 10.3 | Appendix 3: Data Display Standards & Handling Conventions |
| 10.4 | Appendix 4: Derived and Transformed Data |
| 10.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| 10.6 | Appendix 6: Values of Potential Clinical Importance |
| 10.7 | Appendix 7: Biomarker Details |
| 10.8 | Appendix 8: Model Checking and Diagnostics for Statistical Analyses |
| 10.9 | Appendix 9: Population PK and Pharmacokinetic / Pharmacodynamic (or Biomarker) Analyses |
| 10.10 | Appendix 10: Abbreviations & Trade Marks |
| 10.11 | Appendix 11: List of Data Displays |
| 10.12 | Appendix 12: Example Mock Shells for Data Displays |

204987

#### 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Analyses

The study population analyses will be based on the Modified Intent-To-Treat population, unless otherwise specified.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 11: List of Data Displays.

Table 2 Overview of Planned Study Population Analyses

| Data Displays Generated | | |
|---|---|---|
| Table | Figure | Listing |
| Y | | |
| Y | | Υ |
| | | Y |
| Y | | Y |
| | | Y |
| | | Y |
| | | Y |
| Y | | |
| | | Y |
| Y | | Y |
| Y | | Y |
| Y | | |
| | | Y |
| | | Υ |
| | Y Y Y Y Y Y Y Y | Table Figure Y Y Y Y Y Y Y Y Y Y Y Y Y |

#### NOTES:

- Y = Yes display generated.
- 1. Based on All Screened Population
- 2. Separate summaries for past and current conditions

204987

#### 7. PRIMARY STATISTICAL ANALYSES

#### 7.1. Overview of Planned Analyses

The primary analyses will be based on the Modified Intent-To-Treat population.

Table 3 provides an overview of the planned analyses, with full details of data displays being presented in Appendix 11: List of Data Displays.

#### Table 3 Overview of Planned Analyses

| Endpoint / | Absolute | | | | | | | | Change from Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter/ Display | Stats Analysis | | Summary | | Individual | | Stats Analysis | | Summary | | Individual | | | |
| Туре | Т | F | L | Т | F | F | L | Т | F | L | T | F | F | L |
| Primary | Primary | | | | | | | | | | | | | |
| Pulmonary Artery | | | | Υ | Y | Y | Υ | Y1 | Υ | | Y | | | |
| Systolic Pressure | | | | | | | | | | | | | | |
| (PASP) | | | | | | | | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. One table to include statistical analysis medians (95% Crl) and posterior probabilities.

#### 7.2. Planned Statistical Analyses

#### **Primary Statistical Analyses**

#### **Endpoint**

Pulmonary Artery Systolic Pressure (PASP)

#### **Model Specification**

- The description below describes the current thinking of how to analyse this endpoint. The
  proposed model will be assessed, and if not appropriate alternative models could be used.
  Reasons for and a full description of alternative modeling methods used would be fully
  documented in the CPSR.
- The data will be inspected prior to analysis to determine whether a data transformation is required. Any data transformations (e.g. natural logarithm) will be applied to observed individual data prior to any modeling or derivations (e.g. prior to deriving subject baseline)
- A Bayesian repeated measures mixed effects model (fitted using SAS PROC MCMC), will be
  used to model the change from baseline (Ti-T0) in PASP. Based on the study design there are
  4 post-dose timepoints (T1, T2, T3 and T4). The timepoint of primary interest is T3
  (immediately after exercise at altitude).
- Covariates for period, treatment and timepoint (i.e., T1 to T4) will be included as fixed effects.
   Adjusted period-specific baseline and subject-level baseline will be included as continuous
   parameters (see Section 10.3.2.1). Subject will be included as a random effect and timepoint
   will be included as a repeated effect. Treatment by timepoint and adjusted period-specific
   baseline by timepoint interactions will be included. An unstructured variance-covariance matrix
   will be fitted. Non-informative priors will be used for the model parameters, (see Section 10.8).

204987

#### **Primary Statistical Analyses**

- Examination of covariates (for example Age, Weight, Height) may take place, if data permit. In
  this case, the equivalent model may be fitted in PROC MIXED and the covariate assessed at a
  10% alpha level. The final Bayesian model would then be fit based upon the final model (after
  covariate examination) obtained using PROC MIXED. Alternatively, changes in deviance
  information criteria (DIC) may be assessed as part of the PROC MCMC modelling to examine
  covariates.
- Appropriate combinations of the model parameters would be used to obtain posterior distributions for the GSK2586881 vs placebo comparisons at each of the post dosing timepoints (T1 to T4).
- The change from baseline across the different post-dose timepoints will be represented via
  adjusted posterior medians for GSK2586881 and placebo, as well as associated 95% equitailed credible intervals. These results will be presented within tabular and graphical form after
  data has been back transformed (if applicable).
- The difference between GSK2586881 and placebo, for the change from baseline across postdose timepoints will be represented via adjusted medians, as well as their associated 95% equi-tailed credible intervals. These results will be presented within tabular form after data has been back transformed (if applicable).
- The posterior distributions will also be used to produce several posterior probability statements, presented in tabular format; the most important being the probability that the change from baseline in PASP is reduced by GSK2586881 at time T3.
- Posterior probabilities of interest include (looking for <u>high probabilities</u> to favour increases to a lesser extent in PASP on GSK2586881):
  - Probability that change from baseline in PASP is reduced by GSK2586881 (i.e., probability that a treatment difference is negative, or if a log transformation is applied then the probability that the ratio is less than 1).
  - Probability that change from baseline in PASP is reduced by >=2.5mmHg, >=5mmHg and >=7.5mmHg by GSK2586881

(i.e., probability that a treatment difference is <=-2.5 mmHg, <=-5mmHg and <=-7.5mmHg. In the case of a log-transformation, ratios of interest would be <0.95, <0.90 and <0.85, representing 5%, 10% and 15% difference between groups but may be reassessed at the time of analysis)

#### **Model Checking & Diagnostics**

• Refer to Appendix 8: Model Checking and Diagnostics for Statistical Analyses

#### **Model Results Presentation**

- Summary tables for absolute and change from baseline by treatment and timepoint (T0 to T4)
- Listing of absolute data
- Individual subject profiles by treatment group and timepoint
- Summary table of statistical analysis, adjusted change from baseline posterior medians and 95% credible intervals by treatment and timepoint, together with estimated posterior median treatment differences (GSK2586881 – Placebo) and 95% credible intervals for the change from baseline at times T1 to T4 along with posterior probabilities of interest.
- Figure of absolute PASP by timepoint
- Figure of statistical analysis adjusted change from baseline medians and 95% credible intervals by treatment group and timepoint

204987

#### 8. SECONDARY ANALYSES

# 8.1. Safety Analyses

# 8.1.1. Overview of Planned Analyses

The safety analyses will be based on the Modified Intent-To-Treat population, unless otherwise specified.

Table 4 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 11: List of Data Displays.

Table 4 Overview of Planned Safety Analyses

| Endpoint / Parameter/<br>Display Type | Absolute | | | | | | | Change from Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| - F - J - JF | Stats Analysis | | Summary | | Individual | | Stats Analysis | | | Summary | | Individual | | |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Oxygen Saturation | | • | • | • | | • | • | | | | • | | • | • |
| Oxygen Saturation, | | | | Υ | Υ | Υ | Υ | <b>Y</b> 1 | Υ | | Υ | | | |
| measured by continuous | | | | | | | | | | | | | | |
| pulse oximetry | | | | | | | | | | | | | | |
| Oxygen Saturation vs PASP <sup>2</sup> | | | | | Υ | | | | | | | | | |
| Adverse Events | | | | | | | | | | | | | | |
| All AEs for Non- | | | | | | | Υ | | | | | | | |
| randomised Subjects | | | | | | | | | | | | | | |
| All AEs by SOC and PT <sup>3</sup> | | | | Υ | | | Υ | | | | | | | |
| AEs Leading to Study | | | | | | | Υ | | | | | | | |
| Discontinuation | | | | | | | | | | | | | | |
| Drug-Related AEs by | | | | Υ | | | | | | | | | | |
| SOC and PT | | | | | | | | | | | | | | |
| All Serious AEs | | | | Υ | | | Υ | | | | | | | |
| All Laboratory <sup>4</sup> | | | | | | | | | | | | | | |
| Laboratory Values of PCI | | | | | | | Υ | | | | | | | |
| All Laboratory Data for | | | | | | | Υ | | | | | | | |
| Subjects with any Value | | | | | | | | | | | | | | |
| of PCI | | | | | | | | | | | | | | |
| ECG | | | | • | | • | | | | | • | | | |
| ECG Findings | | | | Υ | | | Υ | | | | | | | |
| ECG Values by Visit | | | | Υ | | | | | | | Υ | | | |
| ECG Values of PCI | | | | Υ | | | Υ | | | | Υ | | | |
| All ECG Values for | | | | | | | Υ | | | | | | | |
| Subjects with any Value | | | | | | | | | | | | | | |
| of PCI | | | | | | | | | | | | | | |
| Vital Signs | ı | | | | 1 | | | 1 | ı | 1 | | | | |
| Vital Signs by Visit | | | | Υ | | | | | | | Υ | | | |
| , | | | | | | | | | | | | | | |
204987

| Endpoint / Parameter/<br>Display Type | Absolute | | | Change from Baseline |
|---|---|---|---|---|
| Vital Signs of PCI | | | Υ | |
| All Vital Signs for<br>Subjects with any Value<br>of PCI | | | Y | |
| Immunogenicity | | | | |
| Immunogenicity | | Υ | Υ | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated, PCI = Potential Clinical Importance
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. One table to include statistical analysis medians (95% CrI) and posterior probabilities.
- 2. Scatter plot of x vs y by treatment group, timepoint indicated by panel
- 3. Listing will include subject's numbers for individual AE's and AE system organ classes, preferred terms and verbatim term.
- 4. Chemistry and haematology data will be assessed for PCI values.
- Chemistry collected: BUN, Creatinine, Glucose, Potassium, Sodium, Calcium, AST (SGOT), ALT (SGPT), Alkaline phosphatase, Total and direct bilirubin, Total protein, Albumin.
- Haematology collected: Platelet count, RBC count, haemoglobin, hematocrit, MCV, MCH, neutrophils, lymphocytes, monocytes, eosinophils, basophils.
- Urinalysis collected: Specific gravity, pH, glucose, protein, blood and ketones by dipstick, microscopic examination (if blood or protein is abnormal).

#### 8.1.2. Planned Safety Statistical Analyses

#### **Planned Statistical Analyses**

#### Endpoint(s)

Oxygen Saturation

#### **Model Specification**

- Refer to Section 7.2. Oxygen Saturation will be analysed in the same manner as for the primary endpoint PASP.
- Posterior probabilities of interest include (looking for <u>very low probabilities</u> to remove any concerns with regards to Oxygen Saturation reduction on GSK2586881):
  - Probability that the change from baseline on Oxygen Saturation is reduced by GSK
     (i.e., probability that a treatment difference is <0% or if a log transformation is
     applied then the probability that the ratio < 1).</li>
  - Probability that the change from baseline in Oxygen Saturation is reduced by GSK by >1%, >3% and >=5% (absolute difference) compared to placebo.
    - (i.e., probability that a treatment difference (absolute) is <-1%, <-3% and <=-5%. In the case of a log-transformation, ratios of interest would be <0.98, <0.94 and <0.92 representing 2%, 6% and 8% difference between groups but may be re-assessed at the time of analysis)

#### **Model Checking**

• Refer to Appendix 8: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

Summary tables for absolute and change from baseline by treatment and timepoint (T0 to T4)

204987

#### **Planned Statistical Analyses**

- Listing of absolute data
- Individual subject profiles by treatment group and timepoint
- Summary table of statistical analysis, adjusted change from baseline posterior medians and 95% credible intervals by treatment and timepoint, together with estimated posterior median treatment differences (GSK2586881 – Placebo) and 95% credible intervals for the change from baseline at times T1 to T4 along with posterior probabilities of interest
- Figure of absolute Oxygen Saturation by timepoint
- Figure of statistical analysis adjusted change from baseline medians and 95% credible intervals by treatment group and timepoint

# 8.2. Pharmacokinetic Analyses

## 8.2.1. Overview of Planned Pharmacokinetic Analyses

The pharmacokinetic (PK) analyses will be based on the Pharmacokinetic population, unless otherwise specified.

Table 5 provides an overview of the planned analyses, with full details being presented in Appendix 11: List of Data Displays.

Table 5 Overview of Planned Pharmacokinetic Analyses

| Endpoints | | Untrans | sformed | | Log-Transformed | | | |
|---|---|---|---|---|---|---|---|---|
| | Sum | mary | Indiv | idual | Sum | mary | Individual | |
| | F | T | F | L | F | T | F | L |
| Plasma GSK2586881 concentrations | Y1, 3 | Y | <b>Y</b> 1,2 | Y | | | | |
| Pharmacokinetic Parameters | | Y | | Υ | | Υ | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Linear and Semi-Log plots will be created on the same display.
- 2. One output for one graph per subject and a further output with all subject profiles on the same graphic
- 3. Separate Mean (± SD) and Median plots will be generated.

#### 8.2.2. Drug Concentration Measures

Refer to Appendix 3: Data Display Standards & Handling Conventions (Section 10.3.3 Reporting Process & Standards).

204987

#### 8.2.3. Pharmacokinetic Parameters

#### 8.2.3.1. Deriving Pharmacokinetic Parameters

- Refer to Appendix 3: Data Display Standards & Handling Conventions (Section 10.3.3 Reporting Process & Standards).
- The pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using Win Nonlin Pro V6.3 or greater.
- All calculations of non-compartmental parameters will be based on actual sampling times.
- Pharmacokinetic parameters described in Table 6 will be determined from the plasma concentration-time data, as data permits.

Table 6 Derived Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| AUC(0-2.5h)<br>post-dose | Area under the concentration-time curve over the study period (pre-dose to 30 mins rest post chamber exit). |
| AUC(0.5-2.0h)<br>post-dose | Area under the concentration-time curve over the time period for the hypoxia challenge (immediately prior to chamber entry to chamber exit). |
| AUC(0-∞) | Area under the concentration-time curve extrapolated to infinity. |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| t½ | Apparent terminal half-life will be calculated as: |
| | t½ = ln2 / lambda_z |
| CL | Clearance |
| V | Volume of distribution |
| Lambda_z | The first order rate constant associated with the terminal (log-linear) portion of the concentration-time curve. |
| Lambda_z_lower | First time point used in computing Lambda_z. |
| Lambda_z_upper | Last time point used in computing Lambda_z. |
| #pts | Number of points used in computing Lambda_z. |
| r-squared | R-squared of Lambda_z computation. |

#### NOTES:

- Additional parameters may be included as required.
- Lambda\_z is the terminal phase rate constant.

#### 8.2.4. Population Pharmacokinetic (PopPK) Analyses

A population PK analysis may be conducted. The plasma concentration-time data may be merged with historical data and analysed as part of a population PK meta-analysis. The timeline for these analyses will be independent of the analysis described in this RAP. To support this analysis a NONMEM-specific data file will be generated, the specifications of which are provided in Appendix 9: Population PK and Pharmacokinetic / Pharmacodynamic (or Biomarker) Analyses.

204987

# 8.3. Pharmacodynamic and Biomarker Analyses

# 8.3.1. Overview of Planned Pharmacodynamic and Biomarker Analyses

The pharmacodynamic and biomarker analyses will be based on the Modified Intent-To-Treat population, unless otherwise specified. Biomarker data will be analysed for those subjects in the Modified Intent-To-Treat population for whom a sample was obtained and analysed.

Table 7 provides an overview of the planned pharmacodynamic and Biomarker analyses, with full details of data displays being presented in Appendix 11: List of Data Displays.

Table 7 Overview of Planned Pharmacodynamic and Biomarker Analyses

| Endpoint | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | P | bsolu | ıte | | | | C | hange | from | Basel | ine | |
| | Stat | s Ana | lysis | Sum | mary | Indiv | /idual | Sta | Stats Analysis | | | Summary | | idual |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| RAS Peptide Response | s <sup>1</sup> | | | | | | | | | | | | | |
| Ang II | | | | Υ | Υ | Υ | Υ | Υ | Υ | | | | | |
| Ang(1-7) | | | | Υ | Υ | Υ | Υ | Υ | Υ | | | | | |
| Ang(1-5) | | | | Υ | Υ | Υ | Υ | Υ | Υ | | | | | |
| Other Biomarkers (Dise | ease E | Bioma | rkers | ) | | | | | | | | | | |
| Surfactant Protein D | | | | Υ | Υ | Υ | Υ | Υ | Υ | | | | | |
| <b>Ventilatory Parameters</b> | 1 | | | | | | | | | | | | | |
| Oxygen consumption (VO2) | | | | Υ | | | Υ | | | | | | | |
| Carbon Dioxide<br>Production (CO2) | | | | Υ | | | Υ | | | | | | | |
| Total Tidal Volume | | | | Υ | | | Υ | | | | | | | |
| Inspiratory Tidal<br>Volume | | | | Υ | | | Υ | | | | | | | |
| Expiratory Tidal<br>Volume | | | | Υ | | | Υ | | | | | | | |
| Total Respiratory Time | | | | Υ | | | Υ | | | | | | | |
| Inspiratory Time | | | | Υ | | | Υ | | | | | | | |
| Expiratory Time | | | | Υ | | | Υ | | | | | | | |
| Duty Cycle | | | | Υ | | | Υ | | | | | | | |
| Mean Respiratory Flow | | | | Υ | | | Υ | | | | | | | |
| Respiratory Rate | | | | Υ | | | Υ | | | | | | | |
| RAS Peptides vs PASP | & Ox | ygen | Satur | ation <sup>2</sup> | ! | | | | | | | | | |
| Ang II vs PASP | | | | | Υ | | | | | | | | | |
| Ang(1-7) vs PASP | | | | | Υ | | | | | | | | | |
| Ang(1-5) vs PASP | | | | | Υ | | | | | | | | | |
| Ang II vs Oxygen | | | | | Υ | | | | | | | | | |
| Saturation | | | | | ' | | | | | | | | | |
| Ang(1-7) vs Oxygen<br>Saturation | | | | | Υ | | | | | | | | | |
| Ang(1-5) vs Oxygen<br>Saturation | | | | | Υ | | | | | | | | | |

204987

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Parameters will be included in the same summary/figure/listing paging by RAS peptide where applicable
- 2. Scatter plots of x vs y, timepoint indicated in a legend, one plot for PASP, one plot for Oxygen Saturation (page by RAS peptide)

#### 8.3.2. Planned Pharmacodynamic and Biomarker Statistical Analyses

#### **Planned Statistical Analyses**

#### Endpoint(s)

- RAS Peptide Responses: Ang II, Ang(1-7), Ang(1-5)
- Disease Biomarker: Surfactant Protein D

#### **Model Specification**

- Refer to Section 7.2. Change from baseline in PD/Biomarker endpoints will be analysed in a manner similar to the primary endpoint PASP. Data will be assessed prior to analysis to confirm the need for any data transformations.
- Repeated measures timepoints of interest will be:
- Pre-dose (T0)
- End of Infusion
- 15 min Post-dose (T1)
- 15-45 min Post-dose
- 60 min post chamber entry (T2)
- Immediately post exercise (T3)
- Immediately post chamber exit
- 30 mins post chamber exit (T4)

#### **Model Checking**

Refer to Appendix 8: Model Checking and Diagnostics for Statistical Analyses

#### **Model Results Presentation**

- Summary tables for absolute by treatment and timepoint (as detailed above)
- · Listing of absolute data
- Individual subject profiles by treatment group and timepoint
- Summary table of statistical analysis, adjusted change from baseline posterior medians and 95% credible intervals by treatment and timepoint, together with estimated posterior median treatment differences (GSK2586881 – Placebo) and 95% credible intervals for the change from baseline at ALL timepoints (not just T1 to T4).
- Figure of absolute data by timepoint
- Figure of statistical analysis adjusted change from baseline medians and 95% credible intervals by treatment group and timepoint

204987

# 8.4. Pharmacokinetic / Pharmacodynamic Analyses

The pharmacokinetic/pharmacodynamic (PK/PD) analyses will be based on the mITT population, unless otherwise specified. For the RAS peptides, PASP and Oxygen Saturation endpoints, exploratory plots vs pharmacokinetic concentrations will initially be reviewed to identify endpoints where there is a potential trend. If there is evidence for a trend, further PK/PD analyses may be conducted. The timeline for these analyses will be independent of the analysis described in this RAP. To support this analysis a NONMEM-specific data file will be generated, the specifications of which are provided in Appendix 9: Population PK and Pharmacokinetic / Pharmacodynamic (or Biomarker) Analyses.

Table 8 provides an overview of the planned PK/PD analyses with further details of data displays being presented in Appendix 11: List of Data Displays.

Table 8 Overview of Planned PK/PD Analyses

| Absolute | | | |
|---|---|---|---|
| Sun | nmary | Individual | |
| Т | F | F | L |
| | Y1,2 | | |
| | Y1,2 | | |
| | Y1,2 | | |
| | <b>Y</b> 1 | | |
| | <b>Y</b> 1 | | |
| | Sun | Summary T F | Summary Indiv T F Y1,2 Y1,2 Y1,2 Y1,2 Y1,2 Y1 |

#### **NOTES:**

- 1. Scatter plots, timepoints indicated by panel.
- 2. RAS peptides vs PK will form one graphic, page by RAS peptide
- T = Table, F = Figure, L = Listing, Y = Yes display generated.

204987

#### 9. REFERENCES

GlaxoSmithKline Document Number.: 2016N283626\_00, The effects of GSK2586881 on the responses to acute hypoxia and exercise: Effective date: 23-Sep-2016

GlaxoSmithKline Document Number.: 2016N283626\_01, The effects of GSK2586881 on the responses to acute hypoxia and exercise: Effective date: 24-Feb-2017

GlaxoSmithKline Document Number. : 2016N283626\_02, The effects of GSK2586881 on the responses to acute hypoxia and exercise: Effective date: 07-Mar-2017

204987

# 10. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 5 | : General Considerations for Data Analyses & Data Handling Conventions |
| Section 10.1 | Appendix 1: Time and Events |
| Section 10.2 | Appendix 2: Treatment States |
| Section 10.3 | Appendix 3: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 10.4 | Appendix 4: Derived and Transformed Data |
| | General, Study Population & Safety |
| | Pharmacodynamic and or Biomarkers |
| Section 10.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Section 10.6 | Appendix 6: Values of Potential Clinical Importance |
| Section 10.7 | Appendix 7: Biomarker Details |
| Section 10.8 | Appendix 8: Model Checking and Diagnostics for Statistical Analyses |
| Section 10.9 | Appendix 9: Population PK and Pharmacokinetic / Pharmacodynamic (or |
| | Biomarker) Analyses |
| Other RAP App | endices |
| Section 10.10 | Appendix 10: Abbreviations & Trade Marks |
| Section 10.11 | Appendix 11: List of Data Displays |
| Section 10.12 | Appendix 12: Example Mock Shells for Data Displays |

204987

# 10.1. Appendix 1: Time & Events

# 10.1.1. Protocol Defined Time & Events

204987

# 10.1.1.1. Screening and Follow up

| Procedure | Screening¹<br>(up to 28 days prior to<br>Treatment Period 1, Day 1) | Follow up<br>(7-10 days post<br>last dose) | Notes |
|---|---|---|---|
| Informed consent | X | | |
| Inclusion and exclusion criteria | X | | |
| Demography | X | | |
| Full physical exam, including height and weight | Х | Χ | Height and weight to be measured at screening only. Weight at screening will be used for dosing calculation. |
| Alcohol, Drugs of Abuse, Smoking test | X | | |
| Medical history (includes substance usage [and family history of premature CV disease]) | Х | | Substances: Drugs, Alcohol, tobacco |
| Past and current medical conditions [including cardiovascular medical history] | Х | | |
| Serum OR urine pregnancy test (WCBP) | X | | |
| HIV, Hep B and Hep C screen | X | | |
| Laboratory assessments (include liver | X | Χ | Non Fasting |
| chemistries) | | | |
| Immunogenicity | | Χ | |
| 12-lead ECG | X | Χ | Triplicate ECG required at screening. |
| Vital signs | X | Χ | Triplicate vital signs required at screening. |
| Spirometry | X | | |
| Echocardiogram | X | | |
| Concomitant Medication review | X | Χ | |
| Hypoxia chamber plus exercise | X | | Tolerance to 4000m for 10 mins followed by incremental exercise testing to determine maximum oxygen uptake (VO2max) and calculate 70% of VO2max (to be used for the exercise challenge during the Treatment Periods). |
| Pharmacogenetic sample (PGx) | Х | | Can be taken any time after consent has been signed. Only required once and is optional. |
| AE/SAE review | X | Χ | As per timings detailed in protocol Section 7.2.1.1 |

<sup>1.</sup> Screening assessments are allowed to be conducted on more than one day

204987

#### 10.1.1.2. Treatment Period 1 and 2

| | | | | Tre | atmei | nt Perio | d 1 and | 2 (Washou | ıt 3-14 d | lays) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Tim<br>sta | | | | | mes rel | | e ~80 min<br>entry to | | • , | | Notes |
| Procedure | Pre-dose | 0P | 15 min | 15-45 min | 0-60 min | 60 min | 60-70 min | Immediately after<br>exercise | On exit from chamber | After 30 min rest | 60 min after exit<br>from Chamber | |
| Randomisation | Х | | | | | | | | | | | Randomisation can occur up to the day before the first treatment period |
| Brief physical exam | Χ | | | | | | | | | | | · |
| Vital signs | Χ | | | Χ | | | | Х5 | | | Х | |
| Immunogenicity | Χ | | | | | | | | | | | |
| 12-lead ECG | Χ | | | Χ | | | | | | | X | |
| Echocardiogram | Х | | Х | | | Χ | | Х | | Χ | | Echocardiogram duration approx 5 min |
| Subject enters chamber | | | | | Χ | | | | | | | Subject enters chamber approximately 30 min after study treatment |
| Study Treatment (Dosing) | | Х | | | | | | | | | | , |
| Subject leaves chamber | | | | | | | | Х | | | | Subject leaves chamber after the fourth echocardiogram, blood samples and vital signs have been taken. |
| Exercise challenge | | | | | | | Х | | | | | For approx 5-10 min |
| Ventilatory parameters | Х | | Χ | | | Х | | | | Х | | Measurements to be taken 2 min before echocardiograms. |
| Pulse Oximetry<br>(O2 saturation) | Oximetry Will be continuously monitored for s | | | | | | | Will be continuously monitored for safety. A measurement should be recorded at time of each echocardiogram and databased. | | | | |
| Telemetry | <del>(</del> = | ===== | | | ==== | | ===== | | | | :====→ | Will be continuously monitored for safety. |
| RAS Biomarkers | Χ | X <sup>1</sup> | X <sup>2</sup> | X <sup>3</sup> | | X <sup>2</sup> | | X <sup>2</sup> | X <sup>4</sup> | X <sup>2</sup> | | |
| SP-D | Χ | X <sup>1</sup> | X <sup>2</sup> | X <sup>3</sup> | | X <sup>2</sup> | | X <sup>2</sup> | X <sup>4</sup> | X <sup>2</sup> | | |

204987

| | | | | Tre | | | | l 2 (Washo | ut 3-14 d | days) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | mes rel | | | Hyp<br>(Ti | mes rel | nallenge<br>ative to<br>namber | e ~80 min<br>entry to<br>) | | | | Notes |
| Procedure | Pre-dose | Oh | 15 min | 15-45 min | 0-60 min | 60 min | 60-70 min | Immediately after<br>exercise | On exit from chamber | After 30 min rest | 60 min after exit<br>from Chamber | |
| PK sampling | Χ | Χ¹ | X <sup>2</sup> | X <sup>3</sup> | | X <sup>2</sup> | | X <sup>2</sup> | X <sup>4</sup> | X <sup>2</sup> | | |
| AE/SAE review | | <del>-==</del> | ===== | ==== | | ===== | | | | ======== | =====→ | |
| Concomitant medication review | Χ | | | | | | | | | | | |

- 1. Take at the end of the infusion

- Take at the end of the initistion
   Taken immediately after echocardiogram
   Immediately before entering the chamber
   To be taken as soon as possible after leaving chamber
   On this occasion ONLY, vital signs to be taken after the blood draw.

204987

# 10.2. Appendix 2: Treatment States

#### 10.2.1. Treatment States for AE Data

This study is a single dose two period crossover study. As such, AEs will be attributed to the treatment received within the relevant study period based on the dates and times of the AEs in relation to dosing date and time. This is as per IDSL dataset standards. This is detailed in the table below.

#### 10.2.1.1. Treatment States for AE Dates

| Treatment State | Definition |
|---|---|
| | AE Start Date / Time < Study Treatment Start Date / Time (Period 1) |
| Pre-Treatment | This will apply to all subjects enrolled into the study, including those not randomised. We may have non-randomised and randomised subjects who have pre-treatment AEs/SAEs. For non-randomised subjects these events will be captured in the 'non-randomised' listing. For randomised subjects these events will be captured in summary listings with treatment group='Pre-Treatment'. |
| On-Treatment (Period 1) | If AE Start Date / Time is on or after Study Treatment Start Date / Time (Period 1) & before Study Treatment Start Date / Time (Period 2). Study Treatment Start Date / Time (Period 1) ≤ AE Start Date / Time < Study Treatment Start Date / Time (Period 2) |
| | For randomised subjects, this derivation ensures that AEs starting on or after the Period 1 dose up until the Period 2 dose will be captured and assigned to the Period 1 treatment. |
| On-Treatment (Period 2) | If AE Start Date / Time is on or after Study Treatment Start Date / Time (Period 2) & before Follow-Up. Study Treatment Start Date / Time (Period 2) ≤ AE Start Date / Time ≤ Follow-Up Date |
| | For randomised subjects, this derivation ensures that AEs starting on or after the Period 2 dose up until the Follow-up Visit will be captured and assigned to the Period 2 treatment. |
| Post-Treatment | If AE Start Date is on or after Follow-Up. AE Start Date > Follow-Up Date |
| | There shouldn't be any instances of this. Subjects will return for a follow-up and visit and any AEs would be documented at that point (and hence included in Period 2 treatment group). No further follow-up of patients is required. |
| Onset Time Since 1st<br>Dose (Days/Hours/Mins) | If Study Treatment Start Date / Time (Period 1) ≤ AE Start Date / Time = AE Start Date / Time — Study Treatment Start Date / Time (Period 1) + 1 (min) Missing otherwise. |
| | A calculation to assess the time since the Period 1 dose up until the start time of the AE. This will be calculated for all AEs, regardless of which period/treatment |

204987

| Treatment State | Definition |
|---|---|
| | the AE was assigned to. Example: If Period 1 Dose was administered at 08:00am 01OCT2016 and Period 1 AE started at 09:10am 01OCT2016, then onset time since <b>first</b> dose would be 0d 1h 11m. If Period 2 Dose was administered at 08:30am 08OCT2016 and a Period 2 AE occurred on 08OCT2016 at 10:00am, then onset time since <b>first</b> dose would be 7d 2h 1m. |
| Onset Time Since Period<br>Dose (Days/Hours/Mins) | [PERIOD 1] If AE Start Date / Time is on or after Study Treatment Start Date / Time (Period 1) & before Study Treatment Start Date / Time (Period 2). = AE Start Date / Time – Study Treatment Start Date / Time (Period 1) +1 (min) [PERIOD 2] If AE Start Date / Time is on or after Study Treatment Start Date / Time (Period 2) & on or before Follow-Up. = AE Start Date / Time – Study Treatment Start Date / Time (Period 2) + 1 (min) Missing otherwise. A calculation to assess the time since the dose in the relevant Period/treatment to which the AE is attributable to. Example: [PERIOD 1] If Period 1 Dose was administered at 08:00am 01OCT2016 and Period 1 AE started at 09:10am 01OCT2016, then onset time since period dose would be 0d 1h 11m (i.e. identical to value in previous row example in this case) [PERIOD 2] If Period 2 Dose was administered at 08:30am 08OCT2016 and a Period 2 AE occurred on 08OCT2016 at 10:00am, then onset time since period dose would be 0d 1h 31m |
| Duration<br>(Days/Hours/Mins) | AE Resolution Date / Time – AE Start Date / Time + 1 (min) Example: AE started at 08:00am and resolved at 08:30am on the same day, then duration |
| Drug-related | would be 0d 0h 31m If relationship is marked 'YES' on eCRF OR value is missing |

#### 10.2.2. Treatment States for Concomitant Medication Data

This study is a single dose two period crossover study. As such, Concomitant Medications will be attributed to the treatment received within the relevant study period based on the dates and times of the Concomitant Medications in relation to dosing date and time. This is as per IDSL dataset standards. This is detailed in the table below.

204987

# 10.2.2.1. Treatment States for Concomitant Medication Dates

| Treatment State | Definition |
|---|---|
| Pre-Treatment | CM Start Date / Time < Study Treatment Start Date / Time (Period 1) |
| On-Treatment (Period 1) | If CM Start Date / Time is on or after Study Treatment Start Date / Time (Period 1) & before Study Treatment Start Date / Time (Period 2). Study Treatment Start Date / Time (Period 1) ≤ CM Start Date / Time < Study Treatment Start Date / Time (Period 2) |
| | For randomised subjects, this derivation ensures that CMs starting on or after the Period 1 dose up until the Period 2 dose will be captured and assigned to the Period 1 treatment group. |
| On-Treatment (Period 2) | If CM Start Date / Time is on or after Study Treatment Start Date / Time (Period 2) & before Follow-Up. Study Treatment Start Date / Time (Period 2) ≤ CM Start Date / Time ≤ Follow-Up Date |
| | For randomised subjects, this derivation ensures that CMs starting on or after the Period 2 dose up until the Follow-up Visit will be captured and assigned to the Period 2 treatment. |
| Study Day | Should relate to day since first dose i.e the day of the dose administered during Period 1 should be 'Day 1'. |
| Period Day | Day within the treatment period, for example, Period 1 Day 1 or Period 2 Day 1 |

204987

# 10.3. Appendix 3: Data Display Standards & Handling Conventions

#### 10.3.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|---|---|---|---|
| RandAll NG Data Displays for Reporting | | | ng |
| Code | Description | Description | Order [1] |
| Α | Placebo | Placebo | 1 |
| В | GSK2586881 0.8 mg/kg | GSK2586881 0.8 mg/kg | 2 |

<sup>1.</sup> Order represents treatments being presented in TFL, as appropriate.

#### 10.3.2. Baseline Definition & Derivations

#### 10.3.2.1. Baseline Definitions

For all endpoints (expect as noted in baseline definitions) the baseline value will be the latest predose assessment. Baseline definitions are applicable to each period.

| Parameter | Study Assessments Considered As Baseline | | Baseline Used in |
|---|---|---|---|
| | Screening | Day 1 (Pre-Dose) Time T0 | Data Display |
| Safety | Safety | | |
| PASP | Χ | X | T0 |
| Oxygen Saturation | | X | T0 |
| Labs | Χ | | Screening |
| ECGs | X <sup>1</sup> | X | T0 |
| Vital Signs | X <sup>1</sup> | X | T0 |
| Biomarkers/Pharmacodynamic | | | |
| RAS peptides | | X | T0 |
| Other biomarkers | | X | T0 |
| Ventilatory parameters | | X | T0 |

<sup>&</sup>lt;sup>1</sup>Unless otherwise stated, the mean of replicate assessments at any given time point will be used as the value for that time point.

For statistical analyses (for example, Bayesian mixed model for PASP):

- Baseline is defined as the measurement taken pre-dose during each treatment period (i.e., time T0). This can also be referred to as 'period-specific baseline'.
- **Subject-level baseline** is defined as the mean of the two period-specific baseline readings (the pre-dose T0 reading from each of the two treatment periods) for each subject.

204987

 Period-level baseline (or 'adjusted period-specific baseline') is defined as the difference between the baseline ('period-specific baseline') and 'subject-level baseline' for each period and each subject (i.e., the 'period-specific baseline' minus 'subject-level baseline' in each period).

The statistical modelling will include terms for 'subject-level baseline' and 'adjusted period-specific baseline'.

#### 10.3.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|----------------------|----------------------------------------------|
| Change from Baseline | = Post-Dose Visit Value – Baseline [Ti – T0] |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 10.3.2.1 Baseline Definitions will be used
  for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

#### 10.3.3. Reporting Process & Standards

# Reporting Process Software The currently supported versions of SAS software will be used to perform all data analyses. Generate tables, figures and listings. The latest version of R (or alternative supported available packages) will be used in sample size re-estimation for the interim analysis Reporting Area HARP Server : UK1SALX00175.corpnet2.com

| - I | |
|----------------|---------------------------------------------------|
| HARP Server | : UK1SALX00175.corpnet2.com |
| HARP Area | : \ARPROD\GSK2586881\204987\Internal_01 |
| | : \ARPROD\GSK2586881\204987\Final_01 |
| QC Spreadsheet | : \ARWORK\GSK2586881\204987\Internal_01\documents |
| | : \ARWORK\GSK2586881\204987\Final_01\documents |
| · | |

#### **Analysis Datasets**

- Analysis datasets will be created according to Legacy GSK A&R dataset standards (Integrated Data Standards Library)
- RAS Peptide data samples for Ang II, Ang(1-5) and Ang(1-7) will be processed by Q2 and data provided to GSK Data Management.
- Surfactant Protein D samples and Immunogenicity samples will be processed by GSK and data will be provided to GSK Data Management
- Pharmacokinetic samples will be processed by Covance and data will be provided to GSK Data Management

#### **Generation of RTF Files**

RTF files will be generated for the interim and final reporting efforts

204987

#### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - o 4.03 to 4.23: General Principles
  - o 5.01 to 5.08: Principles Related to Data Listings
  - o 6.01 to 6.11: Principles Related to Summary Tables
  - o 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses :
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

#### Unscheduled Visits

Descriptive

- Unscheduled visits will not be included in summary tables or figures, unless otherwise stated.
- All unscheduled visits will be included in listings.

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Descriptive<br>Summary Statistics<br>(Log Transformed<br>Data) | N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data and between geometric coefficient of variation (CV <sub>b/w</sub> (%)): $ \text{CV}_b \text{ (\%)} = \sqrt{\left(\text{exp}(\text{SD}^2) - 1\right) * 100} $ (NOTE: SD is the SD of log transformed data) |
| Reporting of Pharmacokinetic Concentration Data | |
| Descriptive | Refer to IDSL Statistical Principle 6.06.1 |
| Summary Statistics | Assign zero to NQ values (Refer to GUI_51487 for further details) |
| Reporting of Pharmacokinetic Parameters | |

N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD)

204987

| Reporting Standards | |
|---|---|
| Summary Statistics | of logged data and [between and or within] geometric coefficient of variation |
| (Log Transformed) | (CVb/w (%)) will be reported. |
| | [1] $CV_b$ (%) = $\sqrt{(exp(SD^2) - 1) * 100}$ |
| | (SD = SD of log transformed data) |
| | [2] $CV_w$ (%) = $\sqrt{(exp(MSE) - 1) * 100}$ |
| | (MSE = mean square error from mixed effect model of loge-transformed data). |
| Parameters Not | Tmax, first point, last point and number of points used in the determination of |
| Being Log | lambda_z for listings |
| Transformed | |
| Listings | Include the first point, last point and number of points used in the |
| | determination of lambda_z for listings and R squared |
| Graphical Displays | |
| Refer to IDSL Statistical Principles 7.01 to 7.13. | |

204987

# 10.4. Appendix 4: Derived and Transformed Data

#### 10.4.1. General

#### **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target then the mean will be taken.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Study Day**

- Calculated as the number of days from randomisation date :
  - Ref Date = Missing
- → Study Day = Missing
- Ref Date < Randomisation Date → Study Day = Ref Date Randomisation Date
- Ref Data ≥ Randomisation Date → Study Day = Ref Date (Randomisation Date) + 1

#### 10.4.2. Study Population

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed
  as follows:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)]<sup>2</sup>

#### **Extent of Exposure**

- Number of days of exposure to study drug will be calculated based on the formula:
   Duration of Exposure in Days = Treatment Stop Date (Treatment Start Date) + 1
- Subjects who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.

204987

#### 10.4.3. Safety

#### **ECG Parameters**

#### **RR Interval**

• IF RR interval (msec) is not provided directly, then RR can be derived as :

[1] If QTcB is machine read & QTcF is not provided, then :

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^{3} \right] * 1000$$

 If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.

#### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fridericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as :

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1

# 10.4.4. Pharmacodynamic and Biomarker

# **Biomarkers**

#### **RAS Peptides**

• Ang II, Ang(1-5), Ang(1-7)

#### **Disease Biomarker**

Surfactant Protein D

Variance stabilising transformations (e.g. taking natural logarithms of the observed responses) may be implemented on a per endpoint basis, if deemed necessary by the study statistician. If transformations are used the results will be reported on the back-transformed response scales.

204987

# 10.5. Appendix 5: Premature Withdrawals & Handling of Missing Data

# 10.5.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as any subject who completes all phases in the study including the follow-up visit.</li> <li>Withdrawn subjects will not be replaced in the study.</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 10.5.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument : |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to</li> </ul> |
| | be missing data and should be displayed as such. |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |
| PK | If dosing and/or sampling times are missing, the relevant concentrations will be deleted from the population PK and PK/PD analysis dataset and summarized in a deletion record listing. Samples listed as having no sample (NS), no result (NR) or insufficient sample (IS) will be excluded from the PK data set and also included in the deletion record listing. GSK2586881 concentrations below the lower limit of quantification (LLQ) for the assay will be reported as NQ (Below Quantification Limit). All NQ values will be set to "." (missing) in the population PK and PK/PD dataset. Individuals with all plasma concentrations reported as NQ will be included in the data set. |
| Biomarkers | Any values below the Lower Limit of Quantification (LLQ) will be assigned a value of ½ LLQ for display purposes in Figures and for computation of summary statistics. Any values above the Upper Limit of Quantification (ULQ) will be assigned to the ULQ for display purposes in Figures and for computation of summary statistics. If multiple LLQ and /or ULQ values are available per assay (for example if multiple runs with different standard curves are utilised) then the LLQ and/or ULQ value used for the above imputation shall be the minimum of the available LLQs and/or the maximum of the ULQs. If the number of LLQ (and/or ULQ) values is large for an individual biomarker then alternative applying strategies may be required. "I arrae" in head to define |
| | If the number of LLQ (and/or ULQ) values is large for an individual biomarker then alternative analysis strategies may be required. "Large" is hard to define |

204987

| Element | Reporting Detail |
|---|---|
| | prospectively and may depend upon the dataset in question but a general rule of thumb is if >30% of values are LLQ and/or ULQ. If "large" numbers of LLQ and/or ULQ values are observed methodologies to summarise and analyse the responses similar to those detailed in "Standards for the Handling of NQ impacted PK Parameters" (Respiratory DB and CPMS - 14 <sup>th</sup> December 2009) may be employed. Any such methodology will be documented in the statistical contributions to the clinical study report. |

# 10.5.2.1. Handling of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Treatment States and Phases.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> <li>Start or end dates which are completely missing (i.e. no year specified) will remain missing, with no imputation applied.</li> </ul> |

# 10.5.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant Medications | Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: |
| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will<br/>be used for the month</li> </ul> |
| | If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month. The partial date is a stop date, a '28/29/30/31' will be used for the month. |
| | The recorded partial date will be displayed in listings. |
| Adverse<br>Events | Any partial dates for adverse events will be raised to data management. If the full date cannot be ascertained, the following assumptions will be made: |
| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will<br/>be used for the month.</li> </ul> |
| | <ul> <li>However, if these results in a date prior to Week 1 Day 1 and the event<br/>could possibly have occurred during treatment from the partial information,</li> </ul> |

204987

| Element | Reporting Detail |
|---|---|
| | then the Week 1 Day 1 date will be assumed to be the start date. |
| | <ul> <li>The AE will then be considered to start on-treatment (worst case).</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day</li> </ul> |
| | (dependent on the month and year) and 'Dec' will be used for the month. |
| | The recorded partial date will be displayed in listings. |

# 10.5.2.3. Handling of Missing Data for Statistical Analysis

No missing data imputation methods will be used.

204987

# 10.6. Appendix 6: Values of Potential Clinical Importance

# 10.6.1. Laboratory Values

Laboratory parameters have been reviewed against those specified in the protocol and any parameters not specified here have been assigned as not essential for assessment.

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| I la manta anit | Datia at 1 | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| Homoglobin | g/L | Male | | 180 |
| Hemoglobin | | Female | | 180 |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.8 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | mmol/L | | 30 | |
| BUN | mmol/L | | | ≥ 2x ULN |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | mmol/L | | | ≥ 1.3x ULN |
| Glucose | mmol/L | | 3 | 9 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

204987

# 10.6.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | ≥ 500 | |
| Absolute PR Interval | msec | < 110 | > 220 |
| Absolute QRS Interval | msec | < 75 | > 110 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | > 60 | |

# 10.6.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

| Vital Sign Parameter | Units | Clinical Concern Range | | | |
|---|---|---|---|---|---|
| (Change from Baseline) | | Decrease Increase | | | ease |
| | | Lower | Upper | Lower | Upper |
| Systolic Blood Pressure | mmHg | ≥ 20 | ≥ 40 | ≥ 20 | ≥ 40 |
| Diastolic Blood Pressure | mmHg | ≥ 10 | ≥ 20 | ≥ 10 | ≥ 20 |
| Heart Rate | bpm | ≥ 15 | ≥ 30 | ≥ 15 | ≥ 30 |

204987

# 10.7. Appendix 7: Biomarker Details

| Biomarker<br>Category | Analyte | Method | Lab | Matrix | Total samples expected per subject |
|---|---|---|---|---|---|
| RAS Peptides <sup>1</sup> | Ang II | LCMS | Q2 | Blood | 8 |
| (key | Ang (1-5) | LCMS | Q2 | Blood | 8 |
| endpoints) | Ang (1-7) | LCMS | Q2 | Blood | 8 |
| Disease<br>Biomarkers | Surfactant Protein D | Elisa | GSK | Serum | 8 |

#### NOTES:

- 1. These peptides will be included in the interim analysis.
- Sampling times for each period: Pre-dose (T0), End of Infusion, 15 min Post-dose (T1), 15-45 min Post-dose, 60 min post chamber entry (T2), immediately post exercise (T3), immediately post chamber exit, 30 mins post chamber exit (T4).

204987

# 10.8. Appendix 8: Model Checking and Diagnostics for Statistical Analyses

| Endpoint(s) | • PASP |
|-------------|--------------------------------------------------------------|
| | Oxygen Saturation |
| | <ul> <li>RAS Peptides (AngII, Ang(1-5), Ang(1-7))</li> </ul> |
| | Surfactant Protein D |
| Analysis | SAS PROC MCMC: Bayesian repeated measures mixed model |

- Fixed effects will be assigned a non-informative prior of N(0, Var=1E6) and may be entered as separate univariate priors or as part of a multivariate distribution (variance covariance structure with zeros for off diagonals) in model hyperpriors.
- The non-informative UN priors should be an inverse Wishart distribution. If the equivalent of an unstructured variance covariance matrix does not fit then an AR(1) w/Random Effect structure may be considered, with non-informative priors of U[-1,1] for the off diagonal elements and  $\sigma^2 \sim \text{invGamma}(0.0001, \text{coale}=0.0001)$ .

$$AR(1) = \begin{pmatrix} 1 & \phi & \phi^2 \\ \phi & 1 & \phi \\ \phi^2 & \phi & 1 \end{pmatrix} * \sigma^2$$

- Appropriate SAS helper procedures (e.g. PROC TRANSREG) may be used to convert typical "long and thin" PROC MIXED input datasets into a format appropriate for repeated measures modelling in PROC MCMC (e.g. constructing sets of factors for each class level and fixing the final level to zero)
- Centring of continuous covariates will take place at the input dataset stage: (valuei average) for each subject i.
- Examination of trace plots of samples versus the simulation number and Geweke diagnostics
  to assess convergence. Autocorrelation plots and lag summary table to assess the degree of
  autocorrelation. Monte Carlo standard errors compared to posterior standard deviations (a rule
  of thumb but not binding target would be <0.05). If further diagnostics required a scatterplot
  matrix plot of the posterior samples of each parameter.</li>
- Number of burn ins, thinning, starting points, number of posterior draws to take (10,000 as a starting default) will be customised to each model and may not be possible to specify in advance but will be modified to ensure satisfactory diagnostics are produced.
- For robustness, where non-informative priors are used the equivalent PROC MIXED model
  may be fitted (no output from this would be reported) and LS Means and estimates of
  treatment differences compared to the results obtained from the PROC MCMC analysis. SAS
  code for the random and repeated statements would be:

random int / subject=subjid s vcorr;

repeated visit / subject=subjid\*ptrtgrp type=un r rcorr;

 Model assumptions will be applied, but appropriate adjustments may be made based on the data.

204987

# 10.9. Appendix 9: Population PK and Pharmacokinetic / Pharmacodynamic (Or Biomarker) Analyses

# 10.9.1. Population PK Dataset File Structure

The PME compliant file structure is a space-delimited file with each row containing the following columns of information. Data from all active treatments will be included (i.e. exclude placebo).

Decision as to whether this will be required will be made following the planned interim analysis.

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| С | Data Identifier | Integer | - | 0 |
| STUD | Protocol Number | Integer | - | 204987 |
| DRUG | Name of Drug | Integer | - | Maximum 10 characters (numeric or text). 2586881 |
| SUBJ | Subject identifier in study | Integer | - | Maximum 10 characters (numeric or text). Different identifier for each subject |
| CENT | Study centre identifier | Integer | - | |
| LABL | Indicator field describing the type of assessment in that record | Integer | See<br>footnot<br>es | See footnotes |
| AMT | Dose of<br>GSK2586881 | Decimal | Mg | Amount of drug given = Total GSK2586881 dose (mg/kg)* WT For dosing events: total dose of GSK2586881 taken For concentration events: 0 |
| INF | Infusion Time | Decimal | h | Time during which total dose infused. (Time at end of infusion – Time of start infusion) |
| RATE | Rate of Infusion | Decimal | Mg/h | Rate of infusion (AMT/INF) |
| DGRP | Treatment Identifier | Decimal | - | DGRP=0.8 for 0.8 mg/kg treatment<br>Dose of GSK2586881 (for all events) |
| PART | Study Part | Integer | - | 1=Period 1 or 2=Period 2 |
| DAY | Study day | Integer | - | Maximum 10 characters (numeric or text) N= Day N, Actual Study Day |
| CTIM | Clock Time of Event | HH:MM:SS | - | Clock Time of Event |
| DATE | Date of Record | (DD/MM/YY<br>YY) | - | Date of Record |
| TRFD | Actual time relative to FIRST dose | Decimal | Hours | When LABL = 4, TIME = 0 Hours since start of <u>first</u> active infusion (on Day 1). For pre-dose sample, TRFD is relative to FIRST dose/infusion |

204987

| Variable<br>short<br>name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| TRLD | Actual time relative to LAST dose | Decimal | Hours | When LABL = 4, TIME = 0 Hours since start of LAST infusion. For pre-dose sample, TRLD is relative to previous dose prior to sample For single dose studies TRFD and TRLD are the same |
| TFLAG | Time Flag | Integer | - | At T0 and LABL=6, TFLAG=0<br>At T1 and LABL=6, TFLAG=1<br>At T2 and LABL=6, TFLAG=2<br>At T3 and LABL=6, TFLAG=3<br>At T4 and LABL=6, TFLAG=4<br>Otherwise if LABL=6, TFLAG=5<br>If LABL="0" or "4", TFLAG=6 |
| DV | Dependent Variable | Decimal | pg/mL | When LABL=6, observed GSK2586881 concentration at time specified by TRLD. When LABL=4 (dosing record), DV=0 |
| MDV | Missing Data<br>Variable | Integer | - | Either '0' if DV value present or 1 if DV value is non-quantifiable (NQ) or LABL=4 |
| MDV1 | Missing data variable | Integer | - | Either '0' if LABL=6 or '1' if LABL=4 |
| TYPE | F-Flag | Integer | - | If MDV1='1' then TYPE ='0', If DV value present (but not NQ) TYPE= '1' If DV value NQTYPE = '2' |
| LLQ | Lower Limit of quantification | Integer | pg/mL | Lower limit of quantification for specific analyte SMS dataset (PCLLQ) |
| CMT | Compartment data item | Integer | - | DOSE event: CMT=1, specifies the compartment into which DOSE is introduced. OBSERVATION event: CMT =1, specifies compartment from which observation is obtained. |
| AGE | Age | Decimal | Yrs | Integer. Age in years at time of screening rounded down to give age at last birthday. |
| WT | Weight | Decimal | Kg | Weight in kilograms at time of screening. |
| HT | Height | Decimal | Cm | Height in centimetres at time of screening. |
| SEX | Subject gender | Integer | - | Integer. One of the following -<br>1 = male<br>2 = female |
| ETHN | Subject ethnicity | Integer | - | Integer. Code as CRF |
| RACE | Subject race | Integer | - | Integer. Code as CRF |
| BMI | Body mass index | Decimal | kg/m^2 | body mass index calculated as weight divided by height squared |

204987

| Variable<br>short<br>name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| EVID | Event<br>Indentification data<br>item | Integer | - | Flag indicating whether LABL contains dosing admin info or drug concentration data. Valid values are - 1 – each dosing record for subject 0 - for all other records |

# Assessments captured in the LABL variable

| Label | Description | Units |
|---|---|---|
| 4 | Dosing records for 0.8 mg/Kg GSK2586881 | |
| 6 | Observed concentration record for GSK2586881 at time specified by TRLD; excludes NA, IS and NR, includes non-quantifiable (NQ) data | pg/mL |

204987

# 10.9.2. Population PK/PD Dataset File Structure : ANGII

The PME compliant file structure is a space-delimited file with each row containing the following columns of information. Data from all treatments will be included.

Decision as to whether this will be required will be made following the planned interim analysis.

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| С | Data Identifier | Integer | - | 0 |
| STUD | Protocol Number | Integer | - | 204987 |
| DRUG | Name of Drug | Integer | - | Maximum 10 characters (numeric or text). 2586881 |
| SUBJ | Subject identifier in study | Integer | - | Maximum 10 characters (numeric or text). Different identifier for each subject |
| CENT | Study centre identifier | Integer | - | |
| LABL | Indicator field describing the type of assessment in that record | Integer | See<br>footnotes | See footnotes |
| AMT | Dose of<br>GSK2586881 | Decimal | Mg | Amount of drug given = Total<br>GSK2586881 dose (mg/kg) * WT.<br>AMT=0 when LABL=0<br>For dosing events: total dose of<br>GSK2586881 taken<br>For concentration events: 0 |
| INF | Infusion Time | Decimal | h | Time during which total dose infused. (Time at end of infusion – Time of start infusion) |
| RATE | Rate of Infusion | Decimal | Mg/h | Rate of infusion (AMT/INF) |
| DGRP | Treatment Identifier | Decimal | - | DGRP=0 for placebo treatment DGRP=0.8 for 0.8 mg/kg treatment Dose of GSK2586881 (for all events) |
| PART | Study Part | Varchar | - | 1=Period 1 or 2=Period 2 |
| DAY | Study day | Integer | - | Maximum 10 characters (numeric or text) N= Day N, Actual Study Day |
| CTIM | Clock time of Dose or measurement | HH:MM:SS | - | |
| DATE | Date of record | DD/MM/YYY | | |
| TRFD | Actual time relative to FIRST dose | Decimal | Hours | When LABL=0 or 4, TIME =0<br>Hours since start of FIRST<br>infusion (on Day 1). For pre-dose<br>sample, TRFD is relative to FIRST<br>dose |

204987

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| TRLD | Actual time relative to LAST dose | Decimal | Hours | When LABL=0 or 4, TIME=0 Hours since start of LAST dose/infusion. For pre-dose sample,TRLD is relative to previous dose For single dose studies TRLD = TRFD |
| TFLAG | Time Flag | Integer | - | At T0 and LABL=6, TFLAG=0 At T1 and LABL=6, TFLAG=1 At T2 and LABL=6, TFLAG=2 At T3 and LABL=6, TFLAG=3 At T4 and LABL=6, TFLAG=4 Otherwise if LABL=6, TFLAG=5 If LABL="0" or "4", TFLAG=6 |
| BLII | AngII concentration record | Decimal | | Baseline value (pre-dose value) |
| DV | Angll concentration record | Decimal | | When LABL=6, observed AngII concentration at time specified by TRLD. When LABL=0 or 4, AngII=0 |
| MDV | Missing data variable | Integer | - | Either '0' if DV value present or 1 if DV is non-quantifiable (NQ) value or LABL=0 or 4 |
| MDV1 | Missing data variable | Integer | - | '1' if LABL=0 or 4 "0" when LABL=6 |
| TYPE | F-Flag | Integer | - | If MDV1='1' then TYPE ='0', If DV value present (but not NQ) TYPE= '1' If DV value NQTYPE = '2' |
| CMT | Compartment data item | Integer | - | DOSE event: CMT=1, specifies the compartment into which DOSE is introduced. OBSERVATION event: CMT=3 for DV (ANGII) observation event. |
| AGE | Age | Decimal | Yrs | Integer. Age in years at time of screening rounded down to give age at last birthday. |
| WT | Weight | Decimal | Kg | Weight in kilograms at time of screening. |
| HT | Height | Decimal | Cm | Height in centimetres at time of screening. |
| SEX | Subject gender | Integer | - | Integer. One of the following -<br>1 = male<br>2 = female |
| ETHN | Subject ethnicity | Integer | - | Integer. Code as CRF |
| RACE | Subject race | Integer | - | Integer. Code as CRF |
| BMI | Body mass index | Decimal | kg/m^2 | body mass index calculated as weight divided by height squared |

204987

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| EVID | Event Indentification | Integer | | Flag indicating whether LABL |
| LVID | data item | integer | | contains dosing admin info or drug concentration data. Valid values are - 1 – each dosing record for subject 0 - for all other records |

# Assessments captured in the LABL variable

| Label | Description | Units |
|---|---|---|
| 0 | Dosing record for placebo | |
| 4 | Dosing records for 0.8 mg/Kg GSK2586881 | |
| 6 | Observed record (concentration or ratio) at time specified by TRLD; excludes NA, IS and NR, includes non-quantifiable (NQ) data | |

# 10.9.3. Population PK/PD Dataset File Structure : ANG1-5

The PME compliant file structure is a space-delimited file with each row containing the following columns of information. Data from all treatments will be included.

Decision as to whether this will be required will be made following the planned interim analysis.

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| С | Data Identifier | Integer | - | 0 |
| STUD | Protocol Number | Integer | - | 204987 |
| DRUG | Name of Drug | Integer | - | Maximum 10 characters (numeric or text). 2586881 |
| SUBJ | Subject identifier in study | Integer | - | Maximum 10 characters (numeric or text). Different identifier for each subject |
| CENT | Study centre identifier | Integer | - | |
| LABL | Indicator field<br>describing the type<br>of assessment in<br>that record | Integer | See<br>footnotes | See footnotes |
| AMT | Dose of<br>GSK2586881 | Decimal | Mg | Amount of drug given = Total<br>GSK2586881 dose (mg/kg) * WT.<br>AMT=0 when LABL=0<br>For dosing events: total dose of<br>GSK2586881 taken<br>For concentration events: 0 |
| INF | Infusion Time | Decimal | h | Time during which total dose infused. (Time at end of infusion – |

204987

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| | | | | Time of start infusion) |
| RATE | Rate of Infusion | Decimal | Mg/h | Rate of infusion (AMT/INF) |
| DGRP | Treatment Identifier | Decimal | - | DGRP=0 for placebo treatment<br>treatment<br>DGRP=0.8 for 0.8 mg/kg<br>treatment<br>Dose of GSK2586881 (for all events) |
| PART | Study Part | Varchar | - | 1=Period 1 or 2=Period 2 |
| DAY | Study day | Integer | - | Maximum 10 characters (numeric or text) N= Day N, Actual Study Day |
| CTIM | Clock time of Dose or measurement | HH:MM:SS | - | |
| DATE | Date of record | DD/MM/YYY | | |
| TRFD | Actual time relative to FIRST dose | Decimal | Hours | When LABL=0 or 4, TIME =0 Hours since start of FIRST infusion (on Day 1). For pre-dose sample, TRFD is relative to FIRST dose |
| TRLD | Actual time relative to LAST dose | Decimal | Hours | When LABL=0 or 4, TIME=0 Hours since start of LAST dose/infusion. For pre-dose sample,TRLD is relative to previous dose For single dose studies TRLD = TRFD |
| TFLAG | Time Flag | Integer | - | At T0 and LABL=6, TFLAG=0 At T1 and LABL=6, TFLAG=1 At T2 and LABL=6, TFLAG=2 At T3 and LABL=6, TFLAG=3 At T4 and LABL=6, TFLAG=4 Otherwise if LABL=6, TFLAG=5 If LABL="0" or "4", TFLAG=6 |
| BL15 | Ang1-5<br>concentration<br>record | Decimal | | Baseline value |
| DV | Angl1-5<br>concentration<br>record | Decimal | | When LABL=6, observed Ang1-5 concentration at time specified by TRLD. When LABL=0or 4, Ang1-5=0 |
| MDV | Missing data variable | Integer | - | Either '0' if DV value present or 1 if DV is non-quantifiable (NQ) value or LABL=0 or,4 |
| MDV1 | Missing data variable | Integer | - | '1' if LABL=0 or 4 "0" when LABL=6 |
| TYPE | F-Flag | Integer | - | If MDV1='1' then TYPE ='0', If DV value present (but not NQ) TYPE= '1' If DV value NQTYPE = '2' |

204987

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| CMT | Compartment data item | Integer | - | DOSE event: CMT=1, specifies the compartment into which DOSE is introduced. OBSERVATION event CMT=5 for ANG1-5 observation event. |
| AGE | Age | Decimal | Yrs | Integer. Age in years at time of screening rounded down to give age at last birthday. |
| WT | Weight | Decimal | Kg | Weight in kilograms at time of screening. |
| HT | Height | Decimal | Cm | Height in centimetres at time of screening. |
| SEX | Subject gender | Integer | - | Integer. One of the following -<br>1 = male<br>2 = female |
| ETHN | Subject ethnicity | Integer | - | Integer. Code as CRF |
| RACE | Subject race | Integer | - | Integer. Code as CRF |
| BMI | Body mass index | Decimal | kg/m^2 | body mass index calculated as weight divided by height squared |
| EVID | Event Indentification data item | Integer | - | Flag indicating whether LABL contains dosing admin info or drug concentration data. Valid values are - 1 – each dosing record for subject 0 - for all other records |

#### Assessments captured in the LABL variable

| Label | Description | Units |
|---|---|---|
| 0 | Dosing record for placebo | |
| 4 | Dosing records for 0.8 mg/Kg GSK2586881 | |
| 6 | Observed record (concentration or ratio) at time specified by TRLD; excludes NA, IS and NR, includes non-quantifiable (NQ) data | |

# 10.9.4. Population PK/PD Dataset File Structure : ANG1-7

The PME compliant file structure is a space-delimited file with each row containing the following columns of information. Data from all treatments will be included.

Decision as to whether this will be required will be made following the planned interim analysis.
| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| С | Data Identifier | Integer | - | 0 |
| STUD | Protocol Number | Integer | - | 204987 |
| DRUG | Name of Drug | Integer | - | Maximum 10 characters (numeric or text). 2586881 |
| SUBJ | Subject identifier in study | Integer | - | Maximum 10 characters (numeric or text). Different identifier for each subject |
| CENT | Study centre identifier | Integer | - | |
| LABL | Indicator field<br>describing the type<br>of assessment in<br>that record | Integer | See<br>footnotes | See footnotes |
| AMT | Dose of<br>GSK2586881 | Decimal | Mg | Amount of drug given = Total<br>GSK2586881 dose (mg/kg) * WT.<br>AMT=0 when LABL=0<br>For dosing events: total dose of<br>GSK2586881 taken<br>For concentration events: 0 |
| INF | Infusion Time | Decimal | h | Time during which total dose infused. (Time at end of infusion – Time of start infusion) |
| RATE | Rate of Infusion | Decimal | Mg/h | Rate of infusion (AMT/INF) |
| DGRP | Treatment Identifier | Decimal | - | DGRP=0 for placebo treatment<br>treatment<br>DGRP=0.8 for 0.8 mg/kg<br>treatment<br>Dose of GSK2586881 (for all events) |
| PART | Study Part | Varchar | - | 1=Period 1 or 2=Period 2 |
| DAY | Study day | Integer | - | Maximum 10 characters (numeric or text) N= Day N, Actual Study Day |
| CTIM | Clock time of Dose or measurement | HH:MM:SS | - | |
| DATE | Date of record | DD/MM/YYY | | |
| TRFD | Actual time relative to FIRST dose | Decimal | Hours | When LABL=0 or 4, TIME =0<br>Hours since start of FIRST<br>infusion (on Day 1). For pre-dose<br>sample, TRFD is relative to FIRST<br>dose |
| TRLD | Actual time relative to LAST dose | Decimal | Hours | When LABL=0 or 4, TIME=0 Hours since start of LAST dose/infusion. For pre-dose sample,TRLD is relative to previous dose For single dose studies TRLD = TRFD |
| TFLAG | Time Flag | Integer | - | At T0 and LABL=6, TFLAG=0<br>At T1 and LABL=6, TFLAG=1 |

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| | | | | At T2 and LABL=6, TFLAG=2<br>At T3 and LABL=6, TFLAG=3<br>At T4 and LABL=6, TFLAG=4<br>Otherwise if LABL=6, TFLAG=5<br>If LABL="0" or "4", TFLAG=6 |
| BL17 | Ang1-7<br>concentration<br>record | Decimal | | Baseline value |
| ANG1-7 | Ang1-7<br>concentration<br>record | Decimal | | When LABL=6, observed Ang1-7 concentration at time specified by TRLD. When LABL=0or ,4, DV=0 |
| MDV | Missing data variable | Integer | - | Either '0' if DV value present or 1 if DV is non-quantifiable (NQ) value or LABL=0 or 4 |
| MDV1 | Missing data variable | Integer | - | '1' if LABL=0 or 4<br>"0" when LABL=6 |
| TYPE | F-Flag | Integer | - | If MDV1='1' then TYPE ='0', If ANG1-7 value present (but not NQ) TYPE= '1' If ANG1-7 value NQTYPE = '2' |
| СМТ | Compartment data item | Integer | - | DOSE event: CMT=1, specifies the compartment into which DOSE is introduced. OBSERVATION event: CMT=4 for ANG1-7 observation event. |
| AGE | Age | Decimal | Yrs | Integer. Age in years at time of screening rounded down to give age at last birthday. |
| WT | Weight | Decimal | Kg | Weight in kilograms at time of screening. |
| HT | Height | Decimal | Cm | Height in centimetres at time of screening. |
| SEX | Subject gender | Integer | - | Integer. One of the following -<br>1 = male<br>2 = female |
| ETHN | Subject ethnicity | Integer | - | Integer. Code as CRF |
| RACE | Subject race | Integer | - | Integer. Code as CRF |
| BMI | Body mass index | Decimal | kg/m^2 | body mass index calculated as weight divided by height squared |
| EVID | Event Indentification data item | Integer | - | Flag indicating whether LABL contains dosing admin info or drug concentration data. Valid values are - 1 – each dosing record for subject 0 - for all other records |

204987

### Assessments captured in the LABL variable

| Label | Description | Units |
|---|---|---|
| 0 | Dosing record for placebo | |
| 4 | Dosing records for 0.8 mg/Kg GSK2586881 | |
| 6 | Observed record (concentration or ratio) at time specified by TRLD; excludes NA, IS and NR, includes non-quantifiable (NQ) data | |

# 10.9.5. Population PK/PD Dataset File Structure : Oxygen Saturation/PASP

The PME compliant file structure is a space-delimited file with each row containing the following columns of information. Data from all treatments will be included.

Decision as to whether this will be required will be made following the planned interim analysis.

| Variable | Assessment | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| short name | description | | | |
| С | Data Identifier | Integer | - | 0 |
| STUD | Protocol Number | Integer | - | 204987 |
| DRUG | Name of Drug | Integer | - | Maximum 10 characters (numeric or text). 2586881 |
| SUBJ | Subject identifier in study | Integer | - | Maximum 10 characters (numeric or text). Different identifier for each subject |
| CENT | Study centre identifier | Integer | - | |
| LABL | Indicator field<br>describing the type<br>of assessment in<br>that record | Integer | See<br>footnotes | See footnotes |
| AMT | Dose of<br>GSK2586881 | Decimal | Mg | Amount of drug given = Total GSK2586881 dose (mg/kg) * WT. AMT=0 when LABL=0 For dosing events: total dose of GSK2586881 taken For concentration events: 0 |
| INF | Infusion Time | Decimal | h | Time during which total dose infused. (Time at end of infusion – Time of start infusion) |
| RATE | Rate of Infusion | Decimal | Mg/h | Rate of infusion (AMT/INF) |
| DGRP | Treatment Identifier | Decimal | - | DGRP=0 for placebo treatment<br>treatment<br>DGRP=0.8 for 0.8 mg/kg<br>treatment<br>Dose of GSK2586881 (for all events) |
| PART | Study Part | Varchar | - | 1=Period 1 or 2=Period 2 |
| DAY | Study day | Integer | - | Maximum 10 characters (numeric or text) N= Day N, Actual Study |

204987

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| | | | | Day |
| CTIM | Clock time of Dose or measurement | HH:MM:SS | - | |
| DATE | Date of record | DD/MM/YYY | | |
| TRFD | Actual time relative to FIRST dose | Decimal | Hours | When LABL=1 or 4 , TIME =0 Hours since start of FIRST infusion (on Day 1). For pre-dose sample, TRFD is relative to FIRST dose |
| TRLD | Actual time relative to LAST dose | Decimal | Hours | When LABL=0 or 4, TIME=0 Hours since start of LAST dose/infusion. For pre-dose sample,TRLD is relative to previous dose For single dose studies TRLD = TRFD |
| TFLAG | Time Flag | Integer | - | At T0 and LABL=6, TFLAG=0 At T1 and LABL=6, TFLAG=1 At T2 and LABL=6, TFLAG=2 At T3 and LABL=6, TFLAG=3 At T4 and LABL=6, TFLAG=4 Otherwise if LABL=6, TFLAG=5 If LABL="0" or "4", TFLAG=6 |
| BLPASP | PASP | Decimal | mmHg | Baseline Value |
| PASP | PASP | Decimal | mmHg | When LABL=6, PASP at time specified by TRLD. When LABL=1, or4, PASP=0 |
| BLOS | Oxygen Saturation | Decimal | % | Baseline Value |
| OS | Oxygen Saturation | Decimal | % | When LABL=6, Oxygen Saturation at time specified by TRLD. When LABL=1 or 4, Oxygen Saturation=0 |
| EVID | Event Identification data item | Integer | - | Flag indicating whether LABL contains dosing admin info or drug concentration data. Valid values are - 1 – each dosing record for subject 0 - for all other records |

# Assessments captured in the LABL variable

| Label | Description | Units |
|---|---|---|
| 0 | Dosing record for placebo | |
| 4 | Dosing records for 0.8 mg/Kg GSK2586881 | |
| 6 | Observed record (concentration or ratio) at time specified by TRLD; | |
| | excludes NA, IS and NR | |

204987

# 10.10. Appendix 10: Abbreviations & Trade Marks

### 10.10.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ACE2 | Angiotensin converting enzyme type 2 |
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| ALT | Alanine aminotranferase (SGPT) |
| Ang II | Angiotensin II |
| AST | Aspartate aminotransferase (SGOT) |
| AUC(0-2.5h) | Area under the concentration-time curve over the study period |
| AUC(0.5-2.0h) | Area under the concentration-time curve over the hypoxia challenge |
| A&R | Analysis and Reporting |
| BUN | Blood urea nitrogen |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CL | Clearance |
| Cmax | Maximum observed plasma concentration |
| CO2 | Carbon Dioxide |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DOB | Date of Birth |
| DP | Decimal Places |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Record Form |
| GSK | GlaxoSmithKline |
| GUI | Guidance |
| HPV | Hypoxic Pulmonary Vasoconstriction |
| IA | Interim Analysis |
| ICH | International Conference on Harmonisation |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| mITT | Modified Intent-To-Treat |
| IV | Intravenous |
| LOC | Last Observation Carries Forward |
| MMRM | Mixed Model Repeated Measures |
| O2 | Oxygen |
| PASP | Pulmonary Artery Systolic Pressure |

204987

| Abbreviation | Description |
|--------------|---------------------------------------------------|
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| QC | Quality Control |
| QTcF | Fridericia's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| RAS | Renin-Angiotensin System |
| SAC | Statistical Analysis Complete |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| Tmax | Time to maximum observed concentration |
| T1/2 | Apparent terminal phase half-life |
| V | Volume of Distribution |
| VO2 | Oxygen Consumption |

### 10.10.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| HARP |
| RANDALL NG |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| R (Statistical programming |
| package/language) |
| SAS |
| WinNonLin |

204987

### 10.11. Appendix 11: List of Data Displays

### 10.11.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------------------|------------|------------|
| Study Population | 1.1 to 1.n | 1.1 to 1.n |
| Efficacy | 2.1 to 2.n | 2.1 to 2.n |
| Safety | 3.1 to 3.n | 3.1 to 3.n |
| Pharmacokinetic | 4.1 to 4.n | 4.1 to 4.n |
| Pharmacodynamic and / or Biomarker | 5.1 to 5.n | 5.1 to 5.n |
| Pharmacokinetic / Pharmacodynamic | 6.1 to 6.n | 6.1 to 6.n |
| Section | List | ings |
| ICH Listings | 1 to x | |
| Other Listings | y to z | |

### 10.11.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix 12: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------------------------|---------|---------|----------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Pharmacodynamic and / or Biomarker | PD_Fn | PD_Tn | PD_Ln |
| Pharmacokinetic / Pharmacodynamic | PKPD_Fn | PKPD_Tn | PK/PD_Ln |

#### NOTES:

### 10.11.3. Deliverable [Priority]

| Delivery | Description |
|---|---|
| IA | Interim Analysis (Planned to be completed by GSK) |
| SAC* Final Statistical Analysis Complete (Planned to be completed) | |

<sup>\*</sup>Please note that where IA and SAC are noted together next to an output, GSK internal stats and programming team will take responsibility for this output, unless otherwise stated.

Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

204987

# 10.11.4. Study Population Tables

| Study | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Subjec | t Disposition | | | | |
| 1.1. | mITT | ES1A | Summary of Subject Disposition for the Subject Conclusion Record | | SAC |
| 1.2. | All Subjects<br>Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | | SAC |
| Protoc | ol Deviation | | | | |
| 1.3. | mITT | DV1 | Summary of Important Protocol Deviations | | SAC |
| Popula | tions Analysed | | | | • |
| 1.4. | mITT | SP1A | Summary of Study Populations | Total column only. Include All Screened, mITT and PK. Footnote that percentages based on those in the mITT population, so only PK pop will have a percentage. | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 1.5. | mITT | DM3 | Summary of Demographic Characteristics | | SAC |
| 1.6. | mITT | DM5 | Summary of Race and Racial Combinations | Only total column needs to be included for a crossover study | SAC |
| Medica | I Conditions | | | | • |
| 1.7. | mITT | MH1 | Summary of Past Medical Conditions | | SAC |
| 1.8. | mITT | MH1 | Summary of Current Medical Conditions | | SAC |

204987

### 10.11.5. Safety Tables

| Safety : | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PASP | | | | | |
| 3.1. | mITT | PFT1 | Summary of PASP | IDSL example PFT1 can be followed ('Day' won't be needed). If a log-transformation is required for analysis please include log-transformed summary as a second page using PFT2 example. | IA, SAC<br>(GSK) |
| 3.2. | mITT | PFT3 | Summary of PASP Change from Baseline | IDSL example PFT3 can be followed ('Day' won't be needed). If a log-transformation is required for analysis please include log-transformed summary as a second page using PFT2 example. | IA, SAC<br>(GSK) |
| 3.3. | mITT | SAFE_T1<br>(non-standard) | Summary of Repeated Measures Bayesian<br>Statistical Analysis of Change from Baseline in<br>PASP | As per non-standard example SAFE_T1 but parameter column could be removed. Note that adjusted treatment differences and posterior probabilities (<0, <-2.5, <-5, <-7.5) are included on page 2 of mock example. Please note details regarding treatment differences in Section 7.2 and update output accordingly if a log-transformation is required (SAFE_T2 applies in this case with addition of posterior probabilities to be added). | IA, SAC<br>(GSK) |

| Safety : | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Oxygen | Saturation | | | | |
| 3.4. | mITT | PFT1 | Summary of Oxygen Saturation | IDSL example PFT1 can be followed ('Day' won't be needed). If a log-transformation is required for analysis please include log-transformed summary as a second page using PFT2 example. | IA, SAC<br>(GSK) |
| 3.5. | mITT | PFT3 | Summary of Oxygen Saturation Change from Baseline | IDSL example PFT1 can be followed ('Day' won't be needed). If a log-transformation is required for analysis please include log-transformed summary as a second page using PFT2 example. | IA, SAC<br>(GSK) |
| 3.6. | mITT | SAFE_T1<br>(non-standard) | Summary of Repeated Measures Bayesian<br>Statistical Analysis of Change from Baseline in<br>Oxygen Saturation | As per SAFE_T1 but parameter column could be removed. Note that adjusted treatment differences are included on page 2 of mock example. For OS expecting that we'll need to update the Posterior Probability labels, to <0%, <-1%, <-3%, <-5%, where 5% is the clinical concern level for a treatment difference where GSK reduces OS to a greater extent. Please see Section 8.1.2 with regards to changes required should a log transformation be needed (SAFE_T2 applies in this case with addition of posterior probabilities to be added). | IA, SAC<br>(GSK) |

| Safety : | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Adverse | Adverse Events (AEs) | | | | |
| 3.7. | mITT | AE1CP (same<br>as CP_AE1x) | Summary of All Adverse Events by System Organ<br>Class and Preferred Term | Summarise by treatment group. Any pretreatment AEs to be included in the listing only. Will only be created for interim if sufficient number of AEs are observed. | IA (GSK),<br>SAC (FSP) |
| 3.8. | mITT | AE1CP (same<br>as CP_AE1x) | Summary All Drug-Related Adverse Events by<br>System Organ Class and Preferred Term/by Overall<br>Frequency | Summarise by treatment group. | SAC |
| 3.9. | mITT | AE1CP (same as CP_AE1x) | Summary of All Serious Adverse Events by System<br>Organ Class and Preferred Term | Production of this will be dependent on the number of SAEs, listing may suffice (based on clin pharm IDSL standards advice, this is a conditional summary). Summarise by treatment group. Any pre-treatment SAEs to be included only in listing. | SAC |
| ECG | | | | | |
| 3.10. | mITT | EG1 | Summary of ECG Findings | | SAC |
| 3.11. | mITT | EG2 | Summary of ECG Values | | SAC |
| 3.12. | mITT | CP_EG11 | Frequency of ECG Values by Pre-Specified PCI Categories | Categories as per PCI details in Section 10.6.2. | SAC |
| 3.13. | mITT | EG2 | Summary of Change from Baseline in ECG Values | | SAC |
| 3.14. | mITT | CP_EG12 | Frequency of Change from Baseline ECG Values by Pre-Specified PCI Categories | Categories as per PCI details in Section 10.6.2. | SAC |
| Vital Sig | gns | | | | |
| 3.15. | mITT | VS1 | Summary of Vital Signs | | SAC |
| 3.16. | mITT | VS1 | Summary of Change from Baseline in Vital Signs | | SAC |
| Immuno | ogenicity | | | | |

204987

| Safety : | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.17. | mITT | IMM1 | Summary of Positive Immunogenicity Results | | SAC |

### 10.11.6. Safety Figures

| Safety : | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PASP | | | | | |
| 3.1. | mITT | (non-standard) | Summary of PASP (Absolute) | x-axis will be timepoints T0 to T4, see other mock examples, y-axis will be mean PASP including 95% CI, by treatment groups (add to legend). If data is log-transformed for the analysis then this graphic will need to show geometric means and 95% CIs. | IA, SAC (GSK) |

| Safety : | Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.2. | mITT | SAFE_F1<br>(non-standard) | Adjusted Median Responses and 95% Credible Interval vs Time Profiles of Change from Baseline in PASP | If possible please also add a horizontal line within the graph to indicate the 'hypoxia' in chamber period (approx 30 mins post dose to 120 mins post-dose). Add major tick marks for labels indicated in example graphic. Major tick marks to be PTM labels (or shortened version of). If data is log-transformed for analysis then this graphic will be presenting median ratios. | IA, SAC (GSK) |
| 3.3. | mITT | SAFE_F2<br>(non-standard) | Individual Subject Profiles of PASP | Adjust as space permits, with fewer subjects per page if needed. X-axis and footnote for illustration, can be amended/improved. Vertical reference lines represent start and stop of hypoxia/chamber period. | IA, SAC (GSK) |
| Oxygen | Saturation | | | | |
| 3.4. | mITT | (non-standard) | Summary of Oxygen Saturation (Absolute) | x-axis will be timepoints T0 to T4, see other mock examples, y-axis will be mean Oxygen Saturation including 95% CI, by treatment groups (add to legend) If data is log-transformed for the analysis then this graphic will need to show geometric means and 95% CIs. | IA, SAC (GSK) |

| Safety : Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.5. | mITT | SAFE_F1<br>(non-standard) | Adjusted Median Responses and 95% Credible Interval vs Time Profiles of Change from Baseline in Oxygen Saturation | As above | IA, SAC (GSK) |
| 3.6. | mITT | SAFE_F2<br>(non-standard) | Individual Subject Profiles of Oxygen Saturation | As above | IA, SAC (GSK) |
| 3.7. | mITT | PD_F1<br>(non-standard) | Scatter Plot of Oxygen Saturation vs PASP | Scatter plot: PASP on y axis, treatment groups side by side, timepoint (T0 to T4) split into panels. | SAC |

204987

### 10.11.7. Pharmacokinetic Tables

| Pharmacokinetic : Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Con | centration Data | a | | | |
| 4.1. | PK | PKCT1 (PK01) | Summary of GSK2586881 Pharmacokinetic Concentration-Time Data (ng/mL) | | SAC |
| PK Para | ameter Data | | | | |
| 4.2. | PK | PKPT1 (PK03) | Summary Statistics of Derived Plasma GSK2586881<br>Pharmacokinetic Parameters | See Section 8.2.3.1 for list of parameters to be expected | SAC |
| 4.3. | PK | PKPT3 (PK05) | Summary Statistics of Log-Transformed Derived Plasma<br>GSK2586881 Pharmacokinetic Parameters | See Section 8.2.3.1 for list of parameters to be expected and Section 10.3.3 for details of those NOT to be log transformed | SAC |

204987

# 10.11.8. Pharmacokinetic Figures

| Pharma | Pharmacokinetic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Con | centration Dat | a | | | |
| 4.1. | PK | PKCF1X<br>(PK16b) | Individual GSK2586881 Plasma Concentration–Time Plots (Linear and Semi-log) | By Subject plots | SAC |
| 4.2. | PK | PKCF6 (PK24) | Individual GSK2586881 Plasma Concentration–Time Plot (Linear and Semi-log) | All individual subject profiles on the same graphic. If N>15 then split over two pages e.g. 8 or more subjects per page | SAC |
| 4.3. | PK | PKCF2 (PK17) | Mean Plasma GSK2586881 Concentration-Time Plot (Linear and Semi-Log) | | SAC |
| 4.4. | PK | PKCF3 (PK18) | Median Plasma GSK2586881 Concentration-Time Plot (Linear and Semi-Log) | | SAC |

204987

### 10.11.9. Pharmacodynamic and Biomarker Tables

| Pharma | Pharmacodynamic and Biomarker : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| RAS Pe | ptides – Key | | | | |
| 5.1. | mITT | PD_T1 (or<br>modify PFT1 &<br>PFT2 | Summary of Key RAS Peptides (Absolute Data) | Log-transformed summary to be included as a second page for each parameter if data is log-transformed for analysis. Ang II, Ang(1-5), Ang(1-7) | SAC |
| 5.2. | mITT | SAFE_T2<br>(non-standard) | Summary of Repeated Measures Bayesian<br>Statistical Analysis of Change from Baseline in<br>Key RAS Peptides | Log transformation likely to be required so output as per SAFE_T2. RAS Peptides are collected at timepoints other than T1 to T4 so these will need to be included. Note that adjusted treatment differences are included on page 2 of mock example. Posterior probabilities not required. Ang II, Ang(1-5), Ang(1-7) | SAC |
| Disease | Biomarkers | | | | |
| 5.3. | mITT | PD_T1 (or<br>modify PFT1 &<br>PFT2 | Summary of Surfactant Protein D (Absolute Data) | Log-transformed summary to be included as a second page if data is log-transformed for analysis. Surfactant Protein D | SAC |
| 5.4. | mITT | SAFE_T2<br>(non-standard) | Summary of Repeated Measures Bayesian<br>Statistical Analysis of Change from Baseline in<br>Surfactant Protein D | Log transformation likely to be required so output as per SAFE_T2, otherwise SAFE_T1 (no posterior probabilities). SPD is collected at timepoints other than T1 to T4 so these will need to be included. Note that adjusted treatment differences are included on page 2 of mock example. Posterior probability not required. | SAC |

204987

| Pharmacodynamic and Biomarker : Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Deliverable<br>[Priority] | |
| Ventilat | tory Parameter | S | | | |
| 5.5. | mITT | PFT1 | Summary of Ventilatory Parameters (Absolute Data) | Ventilatory parameters are collected at the same timepoints as PASP, with the exception of the post exercise timepoint. Order parameters as follows: Oxygen consumption (VO2), Carbon dioxide production (CO2), Total Tidal Volume, Inspiratory Tidal Volume, Expiratory Tidal Volume, Total Respiratory Time, Inspiratory Time, Expiratory Time, Duty Cycle, Mean Respiratory Flow,Respiratory rate | SAC |

# 10.11.10. Pharmacodynamic and Biomarker Figures

| Pharma | Pharmacodynamic and Biomarker : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| RAS Peptides – Key | | | | | |
| 5.1. | mITT | (non-standard) | Summary of Key RAS Peptides (Absolute) | x-axis will be timepoints T0 to T4 (plus additional timepoints - see other mock examples), y-axis will be mean RAS including 95% CI, by treatment groups (add to legend). One page per endpoint (3 x RAS endpoints) If a log-transformation is required for analysis please present geometric means and 95% CIs on a second page. | SAC |

| Pharma | Pharmacodynamic and Biomarker : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.2. | mITT | SAFE_F1<br>(non-standard) | Adjusted Median Responses and 95%<br>Credible Interval vs Time Profiles of<br>Change from Baseline in Key RAS<br>Peptides | See example mock SAFE_F1 but page by endpoint (3 RAS endpoints). If log-transformed then median ratios will be plotted. If possible please also add a horizontal line within the graphic to indicate the 'hypoxia' in chamber period (approx 30 mins post dose to 120 mins post-dose). Add major tick marks for labels indicated in example graphic. Major tick marks to be PTM labels (or shortened version of). Note more timepoints for biomarkers other than T1 to T4. | SAC |
| 5.3. | mITT | SAFE_F2<br>(non-standard) | Individual Subject Profiles of Key RAS<br>Peptides | All subjects on one page, one page per RAS endpoint. X-axis and footnote for illustration and can be amended/improved. Vertical reference lines represent start and stop of hypoxia/chamber period. Note more timepoints for biomarkers other than T1 to T4. Please note, mock shows raw data scales, but data may need to be log-transformed so in this case please provide a second page per RAS endpoint with y-axis to accommodate log-transformed data. | IA, SAC (GSK) |
| Disease | Biomarkers | | | | |
| 5.4. | mITT | (non-standard) | Summary of Surfactant Protein D (Absolute) | x-axis will be timepoints T0 to T4 (plus additional timepoints - see other mock examples), y-axis will be mean SPD including 95% CI, by treatment groups (add to legend). If a log-transformation is required for analysis please present geometric means and 95% CIs on a second page. | SAC |

| Pharma | codynamic and | d Biomarker : Fig | ures | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | itle Programming Notes | |
| 5.5. | mITT | SAFE_F1<br>(non-standard) | Adjusted Median Responses and 95%<br>Credible Interval vs Time Profiles of<br>Change from Baseline in Surfactant<br>Protein D | If log-transformed then median ratios will be plotted. If possible please also add a horizontal line within the graphic to indicate the 'hypoxia' in chamber period (approx 30 mins post dose to 120 mins post-dose). Add major tick marks for labels indicated in example graphic. Major tick marks to be PTM labels (or shortened version of). Note more timepoints for biomarkers other than T1 to T4. | SAC |
| 5.6. | mITT | SAFE_F2<br>(non-standard) | Individual Subject Profiles of Surfactant<br>Protein D by Treatment Group and<br>Timepoint | Adjust as space permits, with fewer subjects per page if needed. X-axis and footnote for illustration and can be amended/improved. Vertical reference lines represent start and stop of hypoxia/chamber period. Note more timepoints for biomarkers other than T1 to T4. Please note, mock shows raw data scales, but data may need to be log-transformed so in this case please provide a second page with y-axis to accommodate log-transformed data. | SAC |
| Key RA | S Peptides vs | PASP & Oxygen S | Saturation | | |
| 5.7. | mITT | PD_F1<br>(non-standard) | Scatter Plot of RAS Peptides (Ang II,<br>Ang(1-7) and Ang(1-5)) vs PASP | Scatter plot: PASP on y axis. Page by RAS endpoint, treatment groups side by side, timepoints T0 to T4 within panels (2 columns, 5 rows per page, 3 pages). Plot T0 to T4 timepoints (timepoints that match for the two endpoints of interest) If RAS data is log-transformed, please include a second page y-axis to accommodate log-transformed data. | SAC |

| Pharmacodynamic and Biomarker : Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | |
| 5.8. | mITT | PD_F1<br>(non-standard) | Scatter Plot of RAS Peptides (Ang II,<br>Ang(1-7) and Ang(1-5)) vs Oxygen<br>Saturation | Scatter plot: Oxygen Saturation on y axis. Page by RAS endpoint, treatment groups side by side, timepoints T0 to T4 within panels (2 columns, 5 rows per page, 3 pages). Plot T0 to T4 timepoints (timepoints that match for the two endpoints of interest) If RAS data is log-transformed, please include a second page y-axis to accommodate log-transformed data. | SAC |

204987

### 10.11.11. Pharmacokinetic / Pharmacodynamic Figures

| Pharma | Pharmacokinetic / Pharmacodynamic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.1. | mITT | PK_F1 | Scatter Plot of Plasma GSK2586881 Concentration vs PASP | Timepoint split into panels (matching timepoints are T0 to T4) Placebo PASP data included at concentration of zero for comparison, see mock example. | SAC |
| 6.2. | mITT | PK_F1 | Scatter Plot of Plasma GSK2586881 Concentration vs RAS Peptides (Ang II, Ang(1-5) and Ang(1-7)) | Timepoint split into panels (matching timepoints are T0 to T4) One page per RAS endpoint. Placebo RAS data included at concentration of zero for comparison, see mock example. Please note, if RAS data is log-transformed then also include a second page per RAS endpoint displaying log-transformed RAS vs concentrations. | SAC |
| 6.3. | mITT | PK_F1 | Scatter Plot of AUC(0.5-2h) vs PASP | Timepoint T2 and T3 only, to be included as two separate panels Please include log-transformed AUC graphic on a second page. | SAC |

204987

### 10.11.12. ICH Listings

| ICH : Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | tle Programming Notes | |
| Subject | Disposition | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure | | SAC |
| 2. | mITT | ES2 | Listing of Reasons for Study Withdrawal | | SAC |
| 3. | mITT | BL2 | Listing of Subjects for Whom the Treatment Blind was Broken | | SAC |
| 4. | mITT | CP_TA2 | Listing of Randomised and Actual Treatments | | SAC |
| Protoco | l Deviations | | | | |
| 5. | mITT | DV2 | Listing of Important Protocol Deviations | | SAC |
| 6. | mITT | IE4 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC |
| Populat | tions Analysed | | | | |
| 7. | All Screened<br>Subjects | SP3a | Listing of Subjects Excluded from Any Population | | SAC |
| Demog | raphic and Bas | eline Characterist | tics | | |
| 8. | mITT | DM4 | Listing of Demographic Characteristics | | SAC |
| 9. | mITT | DM10 | Listing of Race | | SAC |
| Prior ar | nd Concomitan | t Medications | | | |
| 10. | mITT | CP_CM4 | Listing of Concomitant Medications | For small studies / limited conmed data, a listing can be used in place of summary table, hence no summary table requested for this study. | SAC |
| Exposu | re and Treatme | ent Compliance | | | |
| 11. | mITT | EX4 | Listing of Exposure Data | | SAC |

| ICH : L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | | | | |
| 12. | All Screened | AE9CP | Listing of All Adverse Events for Non-randomised subjects | Only output AEs that occurred for non-<br>randomised subjects only. These<br>should be assigned as pre-treatment. If<br>no AEs then list 'No data to report'.<br>Any SAEs will be noted on this listing | SAC |
| 13. | mITT | AE9CP | Listing of All Adverse Events | Will include AEs for mITT patients, including those that occurred pretreatment. | IA (GSK),<br>SAC (FSP) |
| Serious | and Other Sig | nificant Adverse | Events | | |
| 14. | mITT | AE9CPA (same as CP_AE9a) | Listing of Serious Adverse Events | As above | SAC |
| 15. | mITT | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | | SAC |
| All Lab | oratory | | | | |
| 16. | mITT | LB6 | Listing of All Laboratory Data for Subjects with Any Value of Potential Clinical Concern/Potential Clinical Importance | Group by chemistry and haematology | SAC |
| 17. | mITT | LB6 | Listing of Laboratory Values of Potential Clinical Importance | Group by chemistry and haematology | SAC |
| ECG | | | | | |
| 18. | mITT | CP_EG4 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | | SAC |
| 19. | mITT | CP_EG4 | Listing of ECG Values of Potential Clinical Importance | | SAC |
| 20. | mITT | CP_EG6 | Listing of Abnormal ECG Findings | | SAC |

| ICH : Li | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Vital Sig | gns | | | | |
| 21. | mITT | CP_VS5 | Listing of All Vital Signs Data for Subjects with Any Value of Potential Clinical Importance | | SAC |
| 22. | mITT | CP_VS5 | Listing of All Vital Signs Data of Potential Clinical Importance | | SAC |

204987

# 10.11.13. Non-ICH Listings

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Safety | | | | | |
| 23. | mITT | PFT9 | Listing of PASP | Follow PFT9 IDSL format, replacing the last four FEV columns on the example with one PASP column. | IA, SAC (GSK) |
| 24. | mITT | PFT9 | Listing of Oxygen Saturation | As above | IA, SAC (GSK) |
| 25. | mITT | PFT9 | Listing of Ventilatory Parameters | Similar format to above except include a parameter column to include all ventilator parameter results at each timepoint. Non-standard modification may be required. | SAC |
| Biomar | kers | | | | |
| 26. | mITT | PD_L1 (non-standard) | Listing of RAS Peptides | See non-standard example PD_L1 | IA, SAC (GSK) |
| 27. | mITT | PD_L1<br>(non-standard) | Listing of Surfactant Protein D | Non-standard example above can be followed | SAC |
| Immun | ogenicity | | | • | |
| 28. | mITT | IMM2 | Listing of Immunogenicity Results | Note: Subjects should have data recorded at screening or period 1 pre-dose (not at both timepoints) | SAC |
| PK | | | | • | |
| 29. | PK | PKCL1X<br>(PK08) | Listing of GSK2586881 Plasma<br>Pharmacokinetic Concentration–Time<br>Data | | SAC |
| 30. | PK | PKPL1X<br>(PK14) | Listing of Derived GSK2586881 Plasma<br>Pharmacokinetic Parameters | See Section 8.2.3.1 for list of parameters. To include lambda_z and the additionally the first point, last point and number of points used in the determination of lambda_z for listings and R squared. | SAC |

204987

#### 10.12. Appendix 12: Example Mock Shells for Data Displays

: SAFE\_T1 : 204987  Example

Protocol

Population : Modified Intent-To-Treat

> Table x.x Summary of Repeated Measures Bayesian Statistical Analysis of Change from Baseline in XXXX

| Parameter | Treatment | Timepoint | N | n | Posterior<br>Median (Std Dev) | 95% Credible<br>Interval |
|---|---|---|---|---|---|---|
| XXXX | Placebo | T1: 15 M Post Infusion | XX | XX | xx.x (xx.xx) | (xx.x, xx.x) |
| | | T2: 60 M Post Chamber Entry | XX | XX | xx.x (xx.xx) | (xx.x, xx.x) |
| | | T3: Immediately Post Exercise | XX | XX | xx.x (xx.xx) | (xx.x, xx.x) |
| | | T4: 30 M Post Chamber Exit | XX | XX | xx.x (xx.xx) | (xx.x, xx.x) |
| | GSK2586881 0.8 mg/kg | T1: 15 M Post Infusion | XX | XX | xx.x (xx.xx) | (xx.x, xx.x) |
| | | T2: 60 M Post Chamber Entry | XX | XX | xx.x (xx.xx) | (xx.x, xx.x) |
| | | T3: Immediately Post Exercise | XX | XX | xx.x (xx.xx) | (xx.x, xx.x) |
| | | T4: 30 M Post Chamber Exit | XX | XX | xx.x (xx.xx) | (xx.x, xx.x) |

No transformation has been applied to the data Non-informative prior used for all modelling parameters Unstructured covariance matrix fitted

Cont.....

204987

Example : SAFE\_T1 Protocol : 204987

Population : Modified Intent-To-Treat

Table x.x
Summary of Repeated Measures Bayesian Statistical Analysis of Change from Baseline in XXXX

| Parameter | Comparison | Timepoint | Posterior Median | 95% Credible | Posterio | r Prob. o | f True D | Oiff > X(units) |
|---|---|---|---|---|---|---|---|---|
| | | • | Difference (Std Dev) | Interval | <0 | <-2.5 | <-5 | <-7.5 |
| XXXX | GSK2586881 0.8 mg/kg | T1: 15 M Post Infusion | xx.x (xx.xx) | (xx.x, xx.x) | 0.xx | 0.xx | 0.xx | 0.xx |
| | Vs Placebo | T2: 60 M Post Chamber Entry | xx.x (xx.xx) | (xx.x, xx.x) | 0.xx | 0.xx | 0.xx | 0.xx |
| | | T3: Immediately Post Exercise | xx.x (xx.xx) | (xx.x, xx.x) | 0.xx | 0.xx | 0.xx | 0.xx |
| | | T4: 30 M Post Chamber Exit | xx.x (xx.xx) | (xx.x, xx.x) | 0.xx | 0.xx | 0.xx | 0.xx |

No transformation has been applied to the data Non-informative prior used for all modelling parameters Unstructured covariance matrix fitted

Programming Note: Mock assumes no transformation. If transformation is required please update table appropriately (see SAFE\_T2) to present backtransformed data e.g. present Adjusted Median Ratios, Posterior Probability Ratio <1, see Section 7.2 and Section 8.1.2. Add any additional footnotes required to clarify analyses performed. Timepoint explanation could be added as footnote if there are column space limitations, example given only. Parameter column could be removed for only one parameter in a summary.

204987


Example Protocol : SAFE\_T2 : 204987

: Modified Intent-To-Treat Population

> Table x.x Summary of Repeated Measures Bayesian Statistical Analysis of Change from Baseline in XXXX

| Parameter | Treatment | Timepoint | N | n | Posterior<br>Median Ratio<br>(SD(Log)) | 95% Credible<br>Interval |
|---|---|---|---|---|---|---|
| XXXX | Placebo | T1: 15 M Post Infusion | XX | XX | x.xx (x.xxx) | (x.xx, x.xx) |
| | | T2: 60 M Post Chamber Entry | XX | XX | x.xx (x.xxx) | (x.xx, x.xx) |
| | | T3: Immediately Post Exercise | XX | XX | x.xx (x.xxx) | (x.xx, x.xx) |
| | | T4: 30 M Post Chamber Exit | XX | XX | x.xx (x.xxx) | (x.xx, x.xx) |
| | GSK2586881 0.8 mg/kg | T1: 15 M Post Infusion | XX | XX | x.xx (x.xxx) | (x.xx, x.xx) |
| | | T2: 60 M Post Chamber Entry | XX | XX | x.xx (x.xxx) | (x.xx, x.xx) |
| | | T3: Immediately Post Exercise | XX | XX | x.xx (x.xxx) | (x.xx, x.xx) |
| | | T4: 30 M Post Chamber Exit | XX | XX | x.xx (x.xxx) | (x.xx, x.xx) |

A log-transformation was applied to the raw data prior to analysis. Non-informative prior used for all modelling parameters Unstructured covariance matrix fitted.

Cont.....

204987

Example : SAFE\_T2 

Protocol: 204987

Population : Modified Intent-To-Treat

Table x.x
Summary of Repeated Measures Bayesian Statistical Analysis of Change from Baseline in XXXX

| Parameter | Comparison | Timepoint | Posterior Median<br>Ratio (SD(Log)) | 95% Credible<br>Interval |
|---|---|---|---|---|
| XXXX | GSK2586881 0.8 mg/kg | T1: 15 M Post Infusion | xx.x (xx.xx) | (xx.x, xx.x) |
| | Vs Placebo | T2: 60 M Post Chamber Entry | xx.x (xx.xx) | (xx.x, xx.x) |
| | | T3: Immediately Post Exercise | xx.x (xx.xx) | (xx.x, xx.x) |
| | | T4: 30 M Post Chamber Exit | xx.x (xx.xx) | (xx.x, xx.x) |

A log-transformation was applied to the raw data prior to analysis. Non-informative prior used for all modelling parameters Unstructured covariance matrix fitted.

Programming Note: Mock assumes log transformation. Add any additional footnotes required to clarify analyses performed. Timepoint explanation could be added as footnote if there are column space limitations, example given only. Parameter column could be removed for only one parameter in a summary.

204987

Example : SAFE\_F1 Page 1 of n
Protocol : 204987

Population : Modified Intent-To-Treat

Figure x.x
Adjusted Median Responses and 95% Credible Interval vs Time Profiles of Change from Baseline in XXXX



Programming notes: Major tick marks to be PTM labels (or shortened version of). Adjusted median ratios to be presented if data is log-transformed.

204987

Example : SAFE\_F2 Protocol : 204987 Page 1 of n

Population : Modified Intent-To-Treat

Figure x.x Individual Subject Profiles of XXXX



204987


Example : PD\_T1 Protocol : 204987

. 204907

Population : Modified Intent-To-Treat

Table x.x Summary of RAS Peptide Parameters

**Actual Treatment** Analyte Group Ν Time n [1] Mean SD Median Min Max n AngII (pg/mL) Placebo Pre-Dose  $\chi\chi$ XX Χ XX.XX XX.XXX XX.XX XX.X XX.X Infusion XX Χ XX.XX XX.XXX XX.XX XX.X XX.X 15 m Post Infusion XX Χ XX.XX XX.XXX XX.XX XX.X XX.X 15-45 m Post Infusion XX Χ XX.XX XX.XXX XX.XX XX.X XX.X 60 m Post Infusion XX Χ XX.XX XX.XXX XX.XX XX.X XX.X Immediately Post Ex. Χ XX XX.XX XX.XXX XX.XX XX.X XX.X Post Chamber Exit XX Χ XX.XX XX.XXX XX.XX XX.X XX.X 30 m Post Chm. Exit XX Χ XX.XX XX.XXX XX.XX XX.X XX.X GSK2586881 0.8 mg/kg xx Pre-Dose XX Х XX.XX XX.XXX XX.XX XX.X XX.X Infusion XX Χ XX.XX XX.XXX XX.XX XX.X XX.X 15 m Post Infusion Χ XX XX.XX XX.XXX XX.XX XX.X XX.X 15-45 m Post Infusion Χ XX XX.XX XX.XXX XX.XX XX.X XX.X 60 m Post Infusion Χ XX.XX XX.XXX XX.XX XX.X XX.X Immediately Post Ex. Χ XX XX.XX XX.XXX XX.XX XX.X XX.X Post Chamber Exit Χ XX XX.XX XX.XXX XX.XX XX.X XX.X 30 m Post Chm. Exit XX Х XX.XX XX.XXX XX.XX XX.X XX.X

Ang(1-5) and Ang(1-7).....

NC – value below LLQ, NA – number of imputed values exceeds 75% of total number of evaluable values, CV – Between subject coefficient of variation **Cont....** 

<sup>[1]</sup> Number of imputed observations (imputed using ½ of the LLQ).

204987

Page x of n

Example : PD\_T1 Protocol : 204987

204907

Population : Modified Intent-To-Treat

### Table x.x Summary of RAS Peptide Parameters

| | Actual Treatment | | | | | Geo. | 95% CI of Geo | | |
|---|---|---|---|---|---|---|---|---|---|
| Analyte | Group | N | Planned Relative Time | n | n [1] | Mean | Mean | SD Logs | CV (%) |
| Angll (pg/mL) | Placebo | XX | Pre-Dose | XX | Х | XX.XX | (xx.xx, xx.xx) | X.XXX | XX.X |
| | | | Infusion | XX | Χ | XX.XX | (xx.xx, xx.xx) | X.XXX | XX.X |
| | | | 15 m Post Infusion | XX | Χ | XX.XX | (xx.xx, xx.xx) | X.XXX | XX.X |
| | | | 15-45 m Post Infusion | XX | Χ | XX.XX | (xx.xx, xx.xx) | X.XXX | XX.X |
| | | | 60 m Post Infusion | XX | Χ | XX.XX | (xx.xx, xx.xx) | X.XXX | XX.X |
| | | | Immediately Post Ex. | XX | Χ | XX.XX | (xx.xx, xx.xx) | X.XXX | XX.X |
| | | | Post Chamber Exit | XX | Χ | XX.XX | (xx.xx, xx.xx) | X.XXX | XX.X |
| | | | 30 m Post Chm. Exit | XX | X | XX.XX | (xx.xx, xx.xx) | X.XXX | XX.X |
| | GSK2586881 0.8 mg/kg | g xx | Pre-Dose | XX | Х | XX.XX | (xx.xx, xx.xx) | X.XXX | XX.X |
| | | - | Infusion | XX | X | XX.XX | (xx.xx, xx.xx) | X.XXX | XX.X |

Ang(1-5) and Ang(1-7).....

Programming notes: Summarise Angll, Ang(1-5) and Ang(1-7) within the summary table, for untransformed and log transformed summary statistics as shown in mock shell.

<sup>[1]</sup> Number of imputed observations (imputed using ½ of the LLQ).

NC – value below LLQ, NA – number of imputed values exceeds 75% of total number of evaluable values, CV – Between subject coefficient of variation.

204987


Example : PD\_F1 Protocol : 204987

Population : Modified Intent-To-Treat

Figure x.x
Scatter Plot of PASP vs RAS Peptides by Timepoint and Treatment



204987


Example : PK\_F1 Protocol : 204987

Population : Modified Intent-To-Treat

Figure x.x Scatter Plot of Plasma GSK2586881 Concentration vs PASP



204987


Example Protocol : PD\_L1 : 204987

Population : Modified Intent-To-Treat

### Listing x Listing of RAS Peptide Parameters

| Invid/<br>Subject | Treatment/<br>Period | Analyte<br>(units) | Date | Actual<br>Time | Planned<br>Time | Time<br>dev. | Rel. Time<br>To Ref. | Result | Imputed<br>Result |
|---|---|---|---|---|---|---|---|---|---|
| xxxx/<br>PPD | Placebo/<br>1 | AngII<br>(pg/mL) | XX <mark>PPD</mark> XXXX | XX:XX | Pre-Dose | | -0.xx | XX.X | |
| | | • / | | XX:XX | Infusion | -0.xx | -0.xx | XX.X | |
| | | | | XX:XX | 15 m Post Infusion | -0.xx | -0.xx | XX.X | |
| | | | | XX:XX | 15-45 m Post Infusion | -0.xx | -0.xx | XX.X | |
| | | | | XX:XX | Imm. Post Exercise | -0.xx | -0.xx | XX.X | |
| | | | | XX:XX | Post Chamber Exit | -0.xx | -0.xx | XX.X | |
| | | | | XX:XX | 30 m Post Chamber Ex | it-0.xx | -0.xx | XX.X | |
| | | Ang(1-5)<br>(pg/mL) | xPPD xx | xx:xx | Pre-Dose | -0.xx | -0.xx | NQ | XX.X |
| | | (F3,) | | XX:XX | Infusion | -0.xx | -0.xx | XX.X | |
| | | | | XX:XX | 15 m Post Infusion | -0.xx | -0.xx | XX.X | |

.....

Note: NQ = Not Quantifiable (Lower Limit of Quantification shown in parentheses), NA=Not Applicable Note: "Infusion" sample is drawn at the end of the infusion